Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – Probenecid vs Allopurinol

NCT04746989

September 12, 2021

### 1. Comparison Details

### a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>probenecid versus allopurinol</u> for gout.

### b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

### 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

### 3. Data Source(s)

Medicare, 2007-2017

### 4. Study Design Diagrams





### 5. Cohort Identification

### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing probenecid to allopurinol. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of probenecid or allopurinol (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

### b. Key details regarding cohort creation

#### Index date:

Day of initiation of new probenecid or allopurinol use

### Inclusion criteria for analyses 1, 3, 4:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of probenecid or allopurinol or any other urate lowering agents (febuxostat, pegloticase, lesinurad) any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- · No history of nursing home admission recorded in any time prior to and including index date
- At least one inpatient or one outpatient claim with gout diagnosis recorded in 365 days prior to and including index date

### Inclusion criteria for analysis 2:

- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of probenecid or allopurinol or any other urate lowering agents (febuxostat, pegloticase, lesinurad) any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least one inpatient or one outpatient claim gout diagnosis recorded in 365 days prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- 180-day continuous use of probenecid or allopurinol starting on the index date

# c. Flowchart of the study cohort assembly

| | Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 7,964,044 |
| Did not meet cohort entry criteria | -6,153,654 | 1,810,390 |
| Excluded due to insufficient enrollment | -637,012 | 1,173,378 |
| Excluded due to prior use of referent | -800,273 | 373,105 |
| Excluded due to prior use of exposure | -20,221 | 352,884 |
| Excluded because patient qualified in >1 exposure category | -194 | 352,690 |
| Excluded based on Dementia Exclusion | -11,861 | 340,829 |
| Excluded based on Gout | -24,396 | 316,433 |
| Excluded based on Nursing Home Admission | -9,840 | 306,593 |
| Excluded based on Urate-lowering drugs | -10,841 | 295,752 |
| Excluded because patient did not begin follow-up | -874 | 294,878 |
| Patients in allopurinol group | | 286,763 |
| Patients in probenecid group | | 8,115 |
| Final cohort | | 294,878 |

## 6. Variables

## a. Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of probenecid

## Comparator:

Initiators of probenecid will be compared to initiators of allopurinol

### b. <u>Covariates:</u>

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes Depression | |
| Obesity | Anxiety |
| Hypertension | Bipolar disorder |
| Coronary artery disease | Schizophrenia |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of hospitalizations |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of rheumatologist visits |
| Pneumococcal vaccination | Number of C-reactive protein tests ordered |
| Herpes zoster vaccination | Osteoporosis |
| Bone mineral density test | Fractures |

| Number of distinct generic agents | Falls |
|-----------------------------------|----------------------------|
| Number of emergency room visits | Use of supplemental oxygen |
| Number of outpatient visits | Combined comorbidity score |

| Comedication use | |
|---|---|
| Lithium | Angiotensin II receptor blockers |
| Anti-epileptic mood stabilizers | Angiotensin converting enzyme inhibitors |
| Anti-epileptics (other than mood stabilizers) | Beta blockers |
| Atypical antipsychotics | Calcium channel blockers |
| Benzodiazepines | Diuretics |
| Serotonin-norepinephrine reuptake Inhibitors | Nitrates |
| Selective serotonin reuptake inhibitors | Lipid lowering drugs |
| Tricyclic antidepressants (TCAs) | Non-insulin diabetes medications |
| Typical antipsychotics | Insulin |
| Anticoagulants | Antidepressants |
| Antiplatelet agents | |

| Gout related factors | |
|----------------------|---------------------------------------------|
| Colchicine use | Nonsteroidal anti-inflammatory drugs/COXIBs |
| Opioids | Glucocorticoid use |
| Uric acid testing | |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Renal dysfunction |
| Coronary artery disease | Chronic liver disease |
| Heart failure | Asthma |
| Stroke or transient ischemic attack | Ischemic heart disease |
| Peripheral vascular disease | Chronic obstructive pulmonary disease |
| Hypertension | Malignancy |
| Diabetes | Drug or alcohol abuse or dependence |
| Hyperlipidemia | Venous thromboembolism |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:

Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of probenecid or allopurinol and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- · End of the study period,
- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (probenecid and allopurinol) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses) or switch between exposure groups

For analysis 2, the follow-up will start 180 days after initiation of probenecid or allopurinol and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

# 7. Feasibility counts

| Analysis scheme | Total<br>allopurinol/probenecid<br>initiators | N outcome | Dementia Rate per 1,000 person-years (95% CI) | Follow-up time in days;<br>Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 286,763 (97.2%)<br>8,115 (2.8%) | 8,633 | 18.13 (17.74, 18.51) | 243 [81, 843] |
| 2: 6 mo induction period, 'as started' | 163,743 (98.2)<br>3,012 (1.8%) | 7,824 | 20.95 (20.48, 21.41) | 1,095 [548, 1,095] |
| 3: exclude 6 mo follow-up (symptoms to claims period) | 162,550 (98.2%)<br>2,992 (1.8%) | 7,206 | 19.49 (19.05, 19.95) | 561 [181, 1,233] |
| 4: Outcome Dx + Rx | 286,763 (97.2%)<br>8,115 (2.8%) | 2,802 | 5.81 (5.59, 6.02) | 246 [82, 857] |

### 8. Propensity score analysis

We will use a propensity-score (PS)¹-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.² Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,³ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁴

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>5</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>6</sup>

# a. PS distributions stratified by treatment group

# Pre-matching propensity score overlap:



## Post-matching propensity score overlap:



# b. Table for covariate balance

| | Unmatched | | | PS-Matched | | |
|---|---|---|---|---|---|---|
| Variable | Probenecid<br>(N = 8,115) | Allopurinol<br>(N = 286,763) | St. Diff | Probenecid<br>(N = 8,115) | Allopurinol<br>(N = 8,115) | St. Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 75.05 (7.20) | 75.04 (7.11) | 0.00 | 75.05 (7.20) | 75.16 (7.23) | -0.02 |
| Gender, n (%) | | | | | | |
| Male | 4,380 (54.0%) | 156,832 (54.7%) | -0.01 | 4,380 (54.0%) | 4,310 (53.1%) | 0.02 |
| Female | 3,735 (46.0%) | 129,931 (45.3%) | 0.01 | 3,735 (46.0%) | 3,805 (46.9%) | -0.02 |
| Race, n (%) | | | | | | |
| White | 6,404 (78.9%) | 225,761 (78.7%) | 0.00 | 6,404 (78.9%) | 6,407 (79.0%) | 0.00 |
| Black | 1,145 (14.1%) | 37,669 (13.1%) | 0.03 | 1,145 (14.1%) | 1,180 (14.5%) | -0.01 |
| Asian | 288 (3.5%) | 11,350 (4.0%) | -0.03 | 288 (3.5%) | 256 (3.2%) | 0.02 |
| Hispanic | 97 (1.2%) | 4,372 (1.5%) | -0.03 | 97 (1.2%) | 97 (1.2%) | 0.00 |
| Native American | 20 (0.2%) | 876 (0.3%) | -0.02 | 20 (0.2%) | 25 (0.3%) | -0.02 |
| Other | 142 (1.7%) | 5,386 (1.9%) | -0.02 | 142 (1.7%) | 137 (1.7%) | 0.00 |
| Unknown | 19 (0.2%) | 1,349 (0.5%) | -0.05 | 19 (0.2%) | 13 (0.2%) | 0.00 |
| Region, n (%) | | | | | | |
| Northeast | 901 (11.1%) | 48,575 (16.9%) | -0.17 | 901 (11.1%) | 924 (11.4%) | -0.01 |
| South | 3,978 (49.0%) | 121,284 (42.3%) | 0.13 | 3,978 (49.0%) | 4,059 (50.0%) | -0.02 |
| North Central | 1,881 (23.2%) | 66,726 (23.3%) | 0.00 | 1,881 (23.2%) | 1,830 (22.6%) | 0.01 |
| West | 1,348 (16.6%) | 49,713 (17.3%) | -0.02 | 1,348 (16.6%) | 1,298 (16.0%) | 0.02 |
| Unknown | 7 (0.1%) | 465 (0.2%) | -0.03 | 7 (0.1%) | 4 (0.0%) | 0.04 |
| Calendar year of index date, n (%) | | | | | | |
| 2007 | 1,618 (19.9%) | 36,567 (12.8%) | 0.19 | 1,618 (19.9%) | 1,662 (20.5%) | -0.01 |
| 2008 | 443 (5.5%) | 11,558 (4.0%) | 0.07 | 443 (5.5%) | 494 (6.1%) | -0.03 |

| 2009 | 961 (11.8%) | 33,085 (11.5%) | 0.01 | 961 (11.8%) | 946 (11.7%) | 0.00 |
|---|---|---|---|---|---|---|
| 2010 | 825 (10.2%) | 32,364 (11.3%) | -0.04 | 825 (10.2%) | 896 (11.0%) | -0.03 |
| 2011 | 1,101 (13.6%) | 33,726 (11.8%) | 0.05 | 1,101 (13.6%) | 1,055 (13.0%) | 0.02 |
| 2012 | 836 (10.3%) | 31,189 (10.9%) | -0.02 | 836 (10.3%) | 795 (9.8%) | 0.02 |
| 2013 | 649 (8.0%) | 28,194 (9.8%) | -0.06 | 649 (8.0%) | 647 (8.0%) | 0.00 |
| 2014 | 367 (4.5%) | 16,497 (5.8%) | -0.06 | 367 (4.5%) | 346 (4.3%) | 0.01 |
| 2015 | 666 (8.2%) | 31,883 (11.1%) | -0.10 | 666 (8.2%) | 647 (8.0%) | 0.01 |
| 2016 | 322 (4.0%) | 15,398 (5.4%) | -0.07 | 322 (4.0%) | 307 (3.8%) | 0.01 |
| 2017 | 327 (4.0%) | 16,302 (5.7%) | -0.08 | 327 (4.0%) | 320 (3.9%) | 0.01 |
| Low income subsidy, n (%) | 2,012 (24.8%) | 70,235 (24.5%) | 0.01 | 2,012 (24.8%) | 1,965 (24.2%) | 0.01 |
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 3,473 (42.8%) | 131,007 (45.7%) | -0.06 | 3,473 (42.8%) | 3,379 (41.6%) | 0.02 |
| Obesity | 1,038 (12.8%) | 46,660 (16.3%) | -0.10 | 1,038 (12.8%) | 1,002 (12.3%) | 0.02 |
| Hypertension | 7,346 (90.5%) | 264,969 (92.4%) | -0.07 | 7,346 (90.5%) | 7,324 (90.3%) | 0.01 |
| Coronary artery disease | 3,217 (39.6%) | 116,906 (40.8%) | -0.02 | 3,217 (39.6%) | 3,201 (39.4%) | 0.00 |
| Depression | 692 (8.5%) | 26,580 (9.3%) | -0.03 | 692 (8.5%) | 668 (8.2%) | 0.01 |
| Anxiety | 670 (8.3%) | 22,410 (7.8%) | 0.02 | 670 (8.3%) | 662 (8.2%) | 0.00 |
| Bipolar disorder | 43 (0.5%) | 1,787 (0.6%) | -0.01 | 43 (0.5%) | 41 (0.5%) | 0.00 |
| Schizophrenia | 21 (0.3%) | 703 (0.2%) | 0.02 | 21 (0.3%) | 24 (0.3%) | 0.00 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 1,121 (13.8%) | 42,703 (14.9%) | -0.03 | 1,121 (13.8%) | 1,093 (13.5%) | 0.01 |
| Mammography, n (%) | 996 (12.3%) | 38,292 (13.4%) | -0.03 | 996 (12.3%) | 986 (12.2%) | 0.00 |
| Colonoscopy, n (%) | 850 (10.5%) | 30,716 (10.7%) | -0.01 | 850 (10.5%) | 856 (10.5%) | 0.00 |
| Fecal occult blood test, n (%) | 679 (8.4%) | 24,114 (8.4%) | 0.00 | 679 (8.4%) | 681 (8.4%) | 0.00 |
| Influenza vaccination, n (%) | 4,763 (58.7%) | 173,930 (60.7%) | -0.04 | 4,763 (58.7%) | 4,779 (58.9%) | 0.00 |
| Pneumococcal vaccination, n (%) | 1,059 (13.0%) | 46,623 (16.3%) | -0.09 | 1,059 (13.0%) | 1,041 (12.8%) | 0.01 |
| Herpes zoster vaccination, n (%) | 51 (0.6%) | 1,593 (0.6%) | 0.00 | 51 (0.6%) | 50 (0.6%) | 0.00 |

| Bone mineral density test, n (%) | 549 (6.8%) | 21,394 (7.5%) | -0.03 | 549 (6.8%) | 611 (7.5%) | -0.03 |
|---|---|---|---|---|---|---|
| Number of distinct generic agents, | | | | | | |
| mean (SD) | 12.90 (6.27) | 13.11 (6.26) | -0.03 | 12.90 (6.27) | 12.73 (5.83) | 0.03 |
| Number of emergency room visits, | | | | | | |
| mean (SD) | 0.78 (1.52) | 0.76 (1.42) | 0.01 | 0.78 (1.52) | 0.75 (1.40) | 0.02 |
| Number of outpatient visits, mean | | | | | | |
| (SD) | 14.79 (18.58) | 14.97 (18.33) | -0.01 | 14.79 (18.58) | 14.93 (21.18) | -0.01 |
| Number of hospitalizations, mean | / 1 | | | | | |
| (SD) | 0.38 (0.86) | 0.42 (0.92) | -0.04 | 0.38 (0.86) | 0.36 (0.85) | 0.02 |
| Number of physician office visits, | 0.00 (0.00) | 0.40.40.00 | | 0.00 (0.00) | 0.05 (0.05) | |
| mean (SD) | 0.38 (0.86) | 0.42 (0.92) | -0.04 | 0.38 (0.86) | 0.36 (0.85) | 0.02 |
| Number of rheumatologist visits, | 0.20 /4.47\ | 0.24 (4.40) | 0.00 | 0.20 (4.47) | 0.20 (4.40) | 0.00 |
| mean (SD) | 0.28 (1.17) | 0.31 (1.19) | -0.03 | 0.28 (1.17) | 0.30 (1.19) | -0.02 |
| Number of C-reactive protein tests | 0.24 (0.76) | 0.20 (0.04) | 0.05 | 0.24 (0.76) | 0.26 (0.80) | 0.03 |
| ordered, mean (SD) Number of serum creatinine tests | 0.24 (0.76) | 0.28 (0.84) | -0.05 | 0.24 (0.76) | 0.26 (0.80) | -0.03 |
| ordered, mean (SD) | 3.54 (3.38) | 4.05 (3.66) | -0.14 | 3.54 (3.38) | 3.51 (3.17) | 0.01 |
| Composite frailty score, mean (SD) | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.16 (0.05) | 0.16 (0.05) | 0.00 |
| Osteoporosis, n (%) | 738 (9.1%) | 27,517 (9.6%) | -0.02 | 738 (9.1%) | 805 (9.9%) | -0.03 |
| Fractures, n (%) | 515 (6.3%) | 17,379 (6.1%) | 0.01 | 515 (6.3%) | 544 (6.7%) | -0.02 |
| Falls, n (%) | 288 (3.5%) | 9,836 (3.4%) | 0.01 | 288 (3.5%) | 295 (3.6%) | -0.01 |
| Use of supplemental oxygen, n (%) | 101 (1.2%) | 4,295 (1.5%) | -0.03 | 101 (1.2%) | 93 (1.1%) | 0.01 |
| Combined comorbidity score, mean | 101 (1.270) | 1,233 (1.370) | 0.03 | 101 (1.270) | 33 (1.170) | 0.01 |
| (SD) | 1.91 (2.67) | 2.32 (2.87) | -0.15 | 1.91 (2.67) | 1.86 (2.61) | 0.02 |
| Comedication use, n (%) | | - ( - , | | | | |
| Lithium | 11 (0.1%) | 290 (0.1%) | 0.00 | 11 (0.1%) | 13 (0.2%) | -0.03 |
| Anti-epileptic mood stabilizers | 68 (0.8%) | 2,528 (0.9%) | -0.01 | 68 (0.8%) | 61 (0.8%) | 0.00 |
| Anti-epileptics (other than mood | · · | , , | | , , | , , | |
| stabilizers) | 1,061 (13.1%) | 37,625 (13.1%) | 0.00 | 1,061 (13.1%) | 1,020 (12.6%) | 0.01 |
| Atypical antipsychotics | 85 (1.0%) | 3,337 (1.2%) | -0.02 | 85 (1.0%) | 77 (0.9%) | 0.01 |
| Benzodiazepines | 419 (5.2%) | 17,154 (6.0%) | -0.03 | 419 (5.2%) | 415 (5.1%) | 0.00 |

| Serotonin-norepinephrine reuptake | 4 | | | | | |
|---|---|---|---|---|---|---|
| inhibitors | 232 (2.9%) | 8,490 (3.0%) | -0.01 | 232 (2.9%) | 224 (2.8%) | 0.01 |
| Selective serotonin reuptake | 0.43 /4.0 40/) | 20 002 (40 00/) | 0.04 | 0.42 (4.0.40() | 024 (40 20() | 0.04 |
| inhibitors Tricyclic antidepressants (TCAs) | 843 (10.4%) | 30,983 (10.8%) | -0.01 | 843 (10.4%) | 831 (10.2%) | 0.01 |
| , | 344 (4.2%) | 11,088 (3.9%) | 0.02 | 344 (4.2%) | 362 (4.5%) | -0.01 |
| Typical antipsychotics | 32 (0.4%) | 745 (0.3%) | 0.02 | 32 (0.4%) | 29 (0.4%) | 0.00 |
| Anticoagulants | 1,473 (18.2%) | 50,451 (17.6%) | 0.02 | 1,473 (18.2%) | 1,443 (17.8%) | 0.01 |
| Antiplatelet agents | 1,143 (14.1%) | 39,983 (13.9%) | 0.01 | 1,143 (14.1%) | 1,133 (14.0%) | 0.00 |
| Angiotensin II receptor blockers | 2,080 (25.6%) | 80,839 (28.2%) | -0.06 | 2,080 (25.6%) | 2,083 (25.7%) | 0.00 |
| Angiotensin converting enzyme | | | | | | |
| inhibitors | 3,514 (43.3%) | 127,490 (44.5%) | -0.02 | 3,514 (43.3%) | 3,483 (42.9%) | 0.01 |
| Beta blockers | 4,326 (53.3%) | 164,799 (57.5%) | -0.08 | 4,326 (53.3%) | 4,295 (52.9%) | 0.01 |
| Calcium channel blockers | 2,919 (36.0%) | 107,797 (37.6%) | -0.03 | 2,919 (36.0%) | 2,902 (35.8%) | 0.00 |
| Diuretics | 4,035 (49.7%) | 153,289 (53.5%) | -0.08 | 4,035 (49.7%) | 4,017 (49.5%) | 0.00 |
| Nitrates | 1,083 (13.3%) | 38,031 (13.3%) | 0.00 | 1,083 (13.3%) | 1,070 (13.2%) | 0.00 |
| Lipid lowering drugs | 4,693 (57.8%) | 179,495 (62.6%) | -0.10 | 4,693 (57.8%) | 4,574 (56.4%) | 0.03 |
| Non-insulin diabetes medications | 2,077 (25.6%) | 77,555 (27.0%) | -0.03 | 2,077 (25.6%) | 1,990 (24.5%) | 0.03 |
| Insulin | 691 (8.5%) | 28,499 (9.9%) | -0.05 | 691 (8.5%) | 646 (8.0%) | 0.02 |
| Antidepressants | 1,509 (18.6%) | 54,092 (18.9%) | -0.01 | 1,509 (18.6%) | 1,523 (18.8%) | -0.01 |
| Goud related factors | | | | | | |
| Colchicine, n (%) | 5,996 (73.9%) | 112,474 (39.2%) | 0.75 | 5,996 (73.9%) | 5,937 (73.2%) | 0.02 |
| Nonsteroidal anti-inflammatory | | | | | | |
| drugs/Coxibs, n (%) | 3,490 (43.0%) | 119,656 (41.7%) | 0.03 | 3,490 (43.0%) | 3,521 (43.4%) | -0.01 |
| Opioids, n (%) | 4,690 (57.8%) | 158,624 (55.3%) | 0.05 | 4,690 (57.8%) | 4,754 (58.6%) | -0.02 |
| Glucocorticoids use, n (%) | 3,060 (37.7%) | 117,638 (41.0%) | -0.07 | 3,060 (37.7%) | 3,025 (37.3%) | 0.01 |
| Number of uric acid tests, mean (SD) | 1.08 (1.10) | 1.32 (1.20) | -0.21 | 1.08 (1.10) | 1.10 (0.96) | -0.02 |
| Comorbid conditions, n (%) | 1 | \ -/ | | · - / | (/ | |
| Atrial fibrillation | 1,647 (20.3%) | 59,789 (20.8%) | -0.01 | 1,647 (20.3%) | 1,593 (19.6%) | 0.02 |
| Heart failure | 1,907 (23.5%) | 72,788 (25.4%) | -0.04 | 1,907 (23.5%) | 1,857 (22.9%) | 0.01 |

| Stroke or transient ischemic attack | 808 (10.0%) | 29,978 (10.5%) | -0.02 | 808 (10.0%) | 787 (9.7%) | 0.01 |
|---|---|---|---|---|---|---|
| Peripheral vascular disease | 1,309 (16.1%) | 48,179 (16.8%) | -0.02 | 1,309 (16.1%) | 1,320 (16.3%) | -0.01 |
| Hyperlipidemia | 6,157 (75.9%) | 230,086 (80.2%) | -0.10 | 6,157 (75.9%) | 6,058 (74.7%) | 0.03 |
| Renal dysfunction | 2,106 (26.0%) | 104,266 (36.4%) | -0.23 | 2,106 (26.0%) | 2,021 (24.9%) | 0.03 |
| Chronic liver disease | 431 (5.3%) | 16,903 (5.9%) | -0.03 | 431 (5.3%) | 386 (4.8%) | 0.02 |
| Asthma | 890 (11.0%) | 32,849 (11.5%) | -0.02 | 890 (11.0%) | 850 (10.5%) | 0.02 |
| Ischemic heart disease | 3,157 (38.9%) | 114,685 (40.0%) | -0.02 | 3,157 (38.9%) | 3,153 (38.9%) | 0.00 |
| Chronic obstructive pulmonary disease | 1,904 (23.5%) | 64,444 (22.5%) | 0.02 | 1,904 (23.5%) | 1,894 (23.3%) | 0.00 |
| Malignancy | 1,994 (24.6%) | 77,101 (26.9%) | -0.05 | 1,994 (24.6%) | 1,983 (24.4%) | 0.00 |
| Drug or alcohol abuse or | F12 (6 20/) | 16 660 (5 99/) | 0.03 | F12 (C 20/) | F00 (6.3%) | 0.00 |
| dependence Venous thromboembolism | 513 (6.3%)<br>499 (6.1%) | 16,660 (5.8%)<br>16,171 (5.6%) | 0.02 | 513 (6.3%)<br>499 (6.1%) | 500 (6.2%)<br>499 (6.1%) | 0.00 |

### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

### 10. References

- 1. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf*. May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 5. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. Comp Effect Res 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- 7. Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.

| # | Implementation in routine care | |
|---|---|---|
| | EXPOSURE vs. COMPARISON | |
| | Probenecid vs Allopurinol | |
| | INCLUSION CRITERIA | |
| 1 | No prior use of urate-lowering agents | Depending on the comparison group, we will require new-use (defined as no use anytime prior to index date) of urate-lowering agents, including probenecid and allopurinol |
| 2 | Sufficient enrollment | Medicare Part A, B, and D enrollment with no HMO coverage for 365 days prior to and on the cohort entry date |
| | | EXCLUSION CRITERIA |
| | Prior history of dementia | Measured any time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| 1 | | ICD9 diagnosis – 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 ICD10 diagnosis – F01.xx-F03.xx, G30.xx-G31.85, R41.xx |
| | | NDC brand name – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or "REMINYL" |
| | No prior history of gout | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| 2 | | ICD9 diagnosis – 274.xx<br>ICD10 diagnosis – M10.00, M10.30, M10.40, M10.4, M1A.00X1, M1A.20X1, M1A.30X1, M1A.40X1, M1A.9XX0, M1A.9XX1, N20.0 |
| | Nursing home admission | Measured 365 days prior to drug initiation – |
| 3 | | MEDPAR - Short Stay/Long Stay/SNF Indicator Code – N = SNF Stay (Prvdr3 = 5, 6, U, W, Y, or Z) |

| Covariate list | |
|---|---|
| Catagony | Potential confounders |
| Category | ICD-9 |
| | Age |
| | Gender |
| Demographics | Race |
| Demographics | Region |
| | Calendar year of index date |
| | Low income subsidy |
| | Diabetes |
| | Obesity |
| | Hypertension |
| Dementia risk factors | Coronary artery disease |
| | Depression |
| | Anxiety |
| | Bipolar disorder |
| | Schizophrenia |
| | Smoking |
| | Mammography |
| | Colonoscopy |
| Lifestyle factors and markers for healthy behavior | Fecal occult blood test |
| · | Influenza vaccination |
| | Pneumococcal vaccination |
| | Herpes zoster vaccination |
| | BMD test |
| | Number of distinct generic agents |
| | Number of emergency room visits |
| | Number of outpatient visits |
| Healthcare utilization measures | Number of hospitalizations |
| | Number of physician office visits |
| | Number of rheumatologist visits Number of CRP tests ordered |
| | Number of CRP tests ordered Number of serum creatinine tests ordered |
| | Number of serum creatinine tests of dered |
| | Composite frailty score |
| | Osteoporosis |
| | Fractures |
| Frailty markers | Falls |
| | Use of supplemental oxygen |
| | A combined comorbidity score |
| | A combined comorbidity score |
| Goutsnacif | ic comorbidities |
| Odd:-specifi | Lithium |
| | Anti-epileptic mood stabilizers |
| | Anti-epiteptic mood stabilizers |

| | Anti anilantics (athor than mood stabilizars) |
|----------------------|-----------------------------------------------|
| | Anti-epileptics (other than mood stabilizers) |
| | Atypical antipsychotics |
| | Benzodiazepines |
| | SNRIs |
| | SSRIs |
| | TCAs |
| | Typical antipsychotics |
| | Anticoagulants |
| Comedications | Antiplatelet agents |
| | Angiotensin II receptor blockers |
| | Angiotensin converting enzyme inhibitors |
| | Beta blockers |
| | Calcium channel blockers |
| | Diuretics |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | Colchicine |
| | NSAID/COXIB |
| Gout related factors | Opioids |
| | Glucocorticoids |
| | Uric acid test |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Hypertension |
| | Diabetes |
| | Hyperlipidemia |
| Comorbid conditions | Renal dysfunction |
| | Chronic liver disease |
| | Asthma |
| | Ischemic heart disease |
| | COPD |
| | Malignancy |
| | Drug or alcohol abuse or dependence |
| | VTE |
| | VIE |

# Appendix A Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2007 |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |

### Low income subsidy

 $\frac{https://www.cms.gov/Medicare/Fligibility-and-}{Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pd}$ 

### Diabetes


## Obesity


Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

Orlistat Sibutramine

Hypertension

| Hypertension | | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
| I10 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| I10 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| I160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| I161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| I110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| I110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, malignant, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| l129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| l120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |

| 11311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
|---|---|---|---|
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | stage renal disease | or end stage renal disease |
| 11310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| 1130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| I1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| 1150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| 1158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| 1150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| 1151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| 1152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| 1158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| 1158 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |
| 1133 | 40333 | pecondary hypertension, unspecified | Totaler anapeditied secondary hypertension |

onary artery disease


| Infarction Inf | 1252 | 412 | Old myocardial | Old myocardial |
|---|---|---|---|---|
| Dilation of Coronary Artery, One Artery, Percutaneous transluminal Device, Percutaneous Approach Dilation of Coronary Artery, One Artery with Percutaneous Percutaneous Approach Percutaneou | | | infarction | infarction |
| Bifurcation, with Drug-eluting Intraluminal coronary angioplasty PTCA | ICD10 Px | ICD9 Px | LongDeslCD10 | LongDeslCD9 |
| Device, Percutaneous Approach Device, Percutaneous Approach Device, Percutaneous Approach Device, Percutaneous Approach Drug-eluting Intraluminal Device, Percutaneous Approach Device, Percutaneous Approach Device, Percutaneous Approach Drug-eluting Intraluminal Device, Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dev | 0270346 | 0066 | Dilation of Coronary Artery, One Artery, | Percutaneous |
| Dilation of Coronary Artery, One Artery with Proceedings Proceedin | | | Bifurcation, with Drug-eluting Intraluminal | transluminal |
| Dilation of Coronary Artery, One Artery with Percutaneous Pe | | | Device, Percutaneous Approach | coronary |
| 0270342 0066 Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, Percutaneous Approach Perc | | | | angioplasty |
| Drug-eluting Intraluminal Device, Percutaneous Approach O270356 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270352 O066 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270352 O066 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270366 O066 Dilation of Coronary Artery, One Artery, Percutaneous Intraluminal Devices, Percutaneous Approach O270367 O270368 O066 Dilation of Coronary Artery, One Artery, Percutaneous Approach Intraluminal Devices, Percutaneous Approach Percutaneous Approach O270367 O066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270376 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Approach A | | | | [PTCA] |
| Percutaneous Approach O270356 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270352 O066 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270352 O066 Dilation of Coronary Artery, One Artery with Percutaneous Two Drug-eluting Intraluminal Devices, Percutaneous Approach O270366 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270362 O066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270376 O060 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Transluminal Coronary Angioplasty PITCA] O270376 O060 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Devices, Perc | 027034Z | 0066 | Dilation of Coronary Artery, One Artery with | Percutaneous |
| angioplasty PTCA | | | Drug-eluting Intraluminal Device, | transluminal |
| Dilation of Coronary Artery, One Artery, Percutaneous transluminal Intraluminal Devices, Percutaneous Approach Percutane | | | Percutaneous Approach | coronary |
| 0270356 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Percutaneous Approach Percutaneous Approach O270352 O066 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Perc | | | | angioplasty |
| Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous transluminal Coronary angioplasty (PTCA) Description of Coronary Artery, One Artery with Percutaneous transluminal Coronary angioplasty (PTCA) Description of Coronary Artery, One Artery, Percutaneous transluminal Intraluminal Devices, Percutaneous Coronary angioplasty (PTCA) Description of Coronary Artery, One Artery, Percutaneous Coronary Approach Intraluminal Devices, Percutaneous Coronary Angioplasty (PTCA) Description of Coronary Artery, One Artery with Percutaneous Tansluminal Coronary Angioplasty (PTCA) Description of Coronary Artery, One Artery, Percutaneous Transluminal Coronary Angioplasty (PTCA) Description of Coronary Artery, One Artery, Percutaneous Transluminal Coronary Approach Intraluminal Devices, Percutaneous Approach Intraluminal Coronary Approach Intraluminal Coronary Approach Intraluminal Coronary Artery, One Artery with Pour or More Drug-eluting Intraluminal Coronary Approach Intraluminal Coronary Artery, One Artery with Percutaneous Transluminal Coronary Approach Intraluminal Coronary Artery, One Artery with Percutaneous Transluminal Coronary Approach Intraluminal Corona | | | | [PTCA] |
| Intraluminal Devices, Percutaneous Approach Approach Approach Approach Approach Approach Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Devices, Percutaneous Approach Devices, Percutaneous Approach Devices, Percutaneous Approach Coronary Angioplasty | 0270356 | 0066 | Dilation of Coronary Artery, One Artery, | Percutaneous |
| Intraluminal Devices, Percutaneous Approach Approach Approach Approach Approach Approach Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Devices, Percutaneous Approach Devices, Percutaneous Approach Devices, Percutaneous Approach Coronary Angioplasty | | | | transluminal |
| Derivative of the process of the p | | | Intraluminal Devices, Percutaneous | coronary |
| Derivative of the process of the p | | | Approach | angioplasty |
| Two Drug-eluting Intraluminal Devices, Percutaneous Approach 0270366 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 0270376 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach 0270372 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty Percutaneous Transluminal T | | | | [PTCA] |
| Two Drug-eluting Intraluminal Devices, Percutaneous Approach 0270366 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach 0270376 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach 0270372 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty Percutaneous Transluminal T | 027035Z | 0066 | Dilation of Coronary Artery, One Artery with | Percutaneous |
| Percutaneous Approach O270366 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270362 O066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270376 O066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270376 O066 Dilation of Coronary Artery, One Artery, Percutaneous Approach Dilation of Coronary Artery, One Artery, Percutaneous Intraluminal Devices, Percutaneous Approach O270372 O066 Dilation of Coronary Artery, One Artery, Percutaneous Approach O270372 O066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O270372 O066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O270372 O067 O068 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O270372 O068 O069 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O270372 | | | | transluminal |
| angioplasty [PTCA] 0270366 | | | | coronary |
| [PTCA] | | | | angioplasty |
| Bifurcation, with Three Drug-eluting transluminal coronary Approach (PTCA) 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous transluminal coronary angioplasty (PTCA) 0270376 0066 Dilation of Coronary Artery, One Artery, One Artery, Percutaneous transluminal coronary angioplasty (PTCA) 0270376 0066 Dilation of Coronary Artery, One Artery, Percutaneous transluminal Intraluminal Devices, Percutaneous coronary angioplasty (PTCA) 027037Z 0066 Dilation of Coronary Artery, One Artery with Percutaneous transluminal Devices, Percutaneous Approach coronary angioplasty (PTCA) | | | | |
| Bifurcation, with Three Drug-eluting transluminal coronary Approach (PTCA) 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous transluminal coronary angioplasty (PTCA) 0270376 Dilation of Coronary Artery, One Artery, One Artery, angioplasty (PTCA) 0270376 Dilation of Coronary Artery, One Artery, Percutaneous transluminal Intraluminal Devices, Percutaneous angioplasty (PTCA) 0270377 Dilation of Coronary Artery, One Artery with Approach angioplasty (PTCA) 0270372 Dilation of Coronary Artery, One Artery with Percutaneous transluminal Devices, Percutaneous Approach angioplasty (PTCA) 0270372 Dilation of Coronary Artery, One Artery with Percutaneous transluminal Devices, Percutaneous Approach coronary angioplasty | 0270366 | 0066 | Dilation of Coronary Artery, One Artery, | |
| Intraluminal Devices, Percutaneous Approach O27036Z O066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach O270376 O066 Dilation of Coronary Artery, One Artery, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O27037Z O066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Transluminal Coronary Angioplasty Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty Angioplasty | | | | |
| Approach Approach Approach Approach Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty [PTCA] Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery Approach Dilation of Coronary Artery, One Artery Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Devices, Percutaneous Approach Coronary Angioplasty | | | | |
| Dilation of Coronary Artery, One Artery with Percutaneous Three Drug-eluting Intraluminal Devices, Percutaneous Approach Percutaneous Approach Percutaneous Approach Percutaneous Approach Percutaneous Approach Percutaneous Perc | | | · | • |
| 027036Z 0066 Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach coronary angioplasty [PTCA] 0270376 0066 Dilation of Coronary Artery, One Artery, Percutaneous transluminal Intraluminal Devices, Percutaneous coronary angioplasty [PTCA] 0270372 0066 Dilation of Coronary Artery, One Artery with Pour or More Drug-eluting angioplasty [PTCA] 027037Z 0066 Dilation of Coronary Artery, One Artery with Percutaneous Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach coronary angioplasty | | | The same | _ · · · · |
| Three Drug-eluting Intraluminal Devices, Percutaneous Approach 0270376 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach 027037Z 0066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty | 0270367 | 0066 | Dilation of Coronary Artery, One Artery with | |
| Percutaneous Approach O270376 O066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach O27037Z O066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Approach Percutaneous Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Angioplasty | 0270002 | 0000 | | |
| angioplasty [PTCA] 0270376 0066 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach 027037Z 0066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach coronary angioplasty [PTCA] Percutaneous transluminal transluminal coronary angioplasty | | | | |
| [PTCA] | | | , er satanesas / ipp/ satan | • |
| 0270376 Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Approach Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary Artery one Artery with Coronary Artery one Artery one Artery with Coronary Artery one Artery one Artery with Coronary Artery one Artery one Artery with Coronary Artery one Artery one Artery with Coronary Artery one Artery one Artery one Artery with Coronary Artery one Artery one Artery one Artery with Coronary Artery one Artery one Artery one Artery with Coronary Artery one Arte | | | | |
| Bifurcation, with Four or More Drug-eluting transluminal coronary Approach angioplasty [PTCA] 027037Z 0066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal transluminal Devices, Percutaneous Approach coronary angioplasty | 0270376 | 0066 | Dilation of Coronary Artery, One Artery | |
| Intraluminal Devices, Percutaneous Approach O27037Z O066 Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Coronary angioplasty | 0270370 | 0000 | | |
| Approach angioplasty [PTCA] 027037Z 0066 Dilation of Coronary Artery, One Artery with Percutaneous Four or More Drug-eluting Intraluminal transluminal Devices, Percutaneous Approach coronary angioplasty | | | | |
| 027037Z 0066 Dilation of Coronary Artery, One Artery with Percutaneous Four or More Drug-eluting Intraluminal transluminal Devices, Percutaneous Approach coronary angioplasty | | | • | · |
| 027037Z 0066 Dilation of Coronary Artery, One Artery with Percutaneous Four or More Drug-eluting Intraluminal transluminal Devices, Percutaneous Approach coronary angioplasty | | | , tpproduct | |
| Four or More Drug-eluting Intraluminal transluminal coronary angioplasty | 0270377 | 0066 | Dilation of Coronary Artery, One Artery with | |
| Devices, Percutaneous Approach coronary angioplasty | 0270372 | 0000 | | |
| angioplasty | | | | |
| | | | Devices, Fercutarieous Approach | • |
| [FTCA] | | | | _ · · · · |
| 02703D6 0066 Dilation of Coronary Artery, One Artery, Percutaneous | 0270206 | 0066 | Dilation of Coronary Artory One Artory | |
| Bifurcation, with Intraluminal Device, transluminal | 02/0300 | 0000 | | |
| | | | ref cutaffeous Apploach | |
| angioplasty | | | | |
| [PTCA] | 0270207 | 0000 | Dilation of Coronary Artary Con Antary with | |
| 02703DZ 0066 Dilation of Coronary Artery, One Artery with Percutaneous | 02/03DZ | UUbb | | |
| Intraluminal Device, Percutaneous Approach transluminal | | | intratuminal Device, Percutaneous Approach | |
| coronary | | | | • |
| angioplasty | | | | |
| [PTCA] | | | | |
| 02703E6 0066 Dilation of Coronary Artery, One Artery, Percutaneous | 02703E6 | 0066 | | |
| Bifurcation, with Two Intraluminal Devices, transluminal | | | | |
| Percutaneous Approach coronary | | | Percutaneous Approach | • · |
| angioplasty | | | | |
| [PTCA] | | | | [PTCA] |


| 33519 |
|----------|
| 33520 |
| 33521 |
| 33522 |
| 33523 |
| 33524 |
| 33525 |
| 33526 |
| 33527 |
| 33528 |
| 33529 |
| 33530 |
| 33531 |
| 33532 |
| 33533 |
| 33534 |
| 33535 |
| 33536 |
| 33545 |
| 33572 |
| CPT |
| 92973 |
| 92982 |
| 92984 |
| 92995 |
| 92996 |
| 92920 |
| 92921 |
| 92924 |
| 92925 |
| 92937 |
| 92938 |
| 92941 |
| 92943 |
| 92944 |
| ICD10 Dx |

ICD9 Dx LongDesICD9 LongDesICD10 1208 4130 Other forms of angina pectoris Angina decubitus Prinzmetal 1201 4131 Angina pectoris with documented spasm angina Other and unspecified 1208 4139 Other forms of angina pectoris angina pectoris Other and unspecified 1209 4139 Angina pectoris, unspecified angina pectoris Atherosclerotic heart disease of native Other and coronary artery with angina pectoris with unspecified 125111 4139 documented spasm angina pectoris Atherosclerotic heart disease of native Other and coronary artery with other forms of angina unspecified 4139 125118 angina pectoris Atherosclerotic heart disease of native Other and coronary artery with unspecified angina unspecified 125119 4139 angina pectoris Atherosclerosis of coronary artery bypass Other and graft(s), unspecified, with angina pectoris unspecified 125701 4139 with documented spasm angina pectoris Atherosclerosis of coronary artery bypass Other and graft(s), unspecified, with other forms of unspecified 125708 4139 angina pectoris angina pectoris


| Dilation of Coronary Artery, Two Arteries with cronary artery stent(s) Dilation of Coronary Artery, Two Arteries, coronary artery stent(s) Dilation of Coronary Artery, Two Arteries, direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of direction of direction of direction of direction of direction of direction of Dilation of Coronary Artery, Three Arteries, direction of Dilation of Coronary Artery, Three Arteries, direction of direction of direction of Dilation of Coronary Artery, Three Arteries direction of | luccution of | | 1 | |
|---|---|---|---|---|
| Three Drug-eluting Intraluminal Devices, coronary artery | Insertion of | Dilation of Caranagu Artagu Two Artarias with | | |
| Dilation of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries with a forum of Grown of Grown of Coronary Artery, Two Arteries with forum of Grown of More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal or Grown or Approach stent(s) Dilation of Coronary Artery, Three Arteries, and Grown or G | = = | · | | |
| Dilation of Coronary Artery, Two Arteries, dinsertion of Bifurcation, with Four or More Drug-eluting drug-eluting drug-eluting coronary artery stent(s) 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with Insertion of Grug-eluting Devices, Percutaneous Endoscopic coronary artery stent(s) 0271472 3607 Approach Significant of Coronary Artery, Two Arteries with Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) 0272046 3607 Device, Open Approach stent(s) 0272047 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272048 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery stent(s) 0272049 Significant of Coronary Artery, Three Arteries, drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272050 Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272051 Significant of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach Stent(s) 0272052 3607 Open Approach Significant of Coronary Artery, Three Arteries Sifurcation, with Twee Drug-eluting Coronary artery Stent(s) 0272066 Significant of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) 0272067 Significant Signific | | , | 2607 | 0274467 |
| Bifurcation, with Four or More Drug-eluting coronary artery stent(s) 10271476 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Two Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, and for Special Stent(s) Dilation of Coronary Artery, Three Arteries with four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries selfurcation, with Two Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Thre | ` ' | | 3607 | 02/1462 |
| Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) | | · | | |
| Dilation of Coronary Artery, Three Arteries with Insertion of Grug-eluting Intraluminal Devices, Open Approach | 0 0 | , | | |
| Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary arte | | - | 2607 | 0274476 |
| Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting mornary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) | | | 3607 | 02/14/6 |
| Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | · | | |
| 027147Z 3607 Approach Stent(s) Insertion of drug-eluting coronary artery stent(s) O272046 3607 Device, Open Approach O272046 O272047 O272047 O272047 O272048 O | ŭ ŭ | | | |
| Dilation of Coronary Artery, Three Arteries, setults and setulting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, with Drug-eluting Intraluminal pevice, Open Approach Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, site of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, site of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sith Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sith four or More Drug-eluting Intraluminal coronary artery stent(s) | | - | 2607 | 0274 477 |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Device, Open Approach Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, T | ` ' | Approacn | 3607 | 02/14/2 |
| Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting lintraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | Dilation of Common Adam Thomas Adams | | |
| 0272046 3607 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting sention of Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting linsertion of linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting linsertion of drug-eluting linsertion of drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) | = = | · | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting gradient stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | ` ' | Device, Open Approach | 3607 | 0272046 |
| with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272052 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) | | | | |
| 0272042 3607 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, with Two Drug-eluting Intraluminal Devices, oronary artery 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 027206B 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, with Three Drug-eluting Coronary artery 027206C 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Coronary artery stent(s) Insertion of drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery Open | = = | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 10272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027207G 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 1 Insertion of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 2 Stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery 2 Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | ' ' | | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Insertion of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Stent(s) | | Approach | 3607 | 027204Z |
| Bifurcation, with Two Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery coronary artery stent(s) | | | | |
| 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) O27205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Three Drug-eluting coronary artery stent(s) O272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) | | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) 3607 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | | | |
| Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, stent(s) Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Oz72066 3607 Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Sifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion Of Gronary Artery Stent Stent(s) Insertion Of Gronary Artery Stent Stent(s) Insertion Of Gronary Artery Stent St | ` ' | Intraluminal Devices, Open Approach | 3607 | 0272056 |
| with Two Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, With Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Sifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | | | | |
| 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery with Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Insertion of drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery | | · | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z O27 | , coronary artery | with Two Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting O272076 3607 Dilation of Coronary Artery, Three Arteries Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting O272072 3607 Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O272072 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O272072 3607 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O272072 O272072 O272072 O272072 O272072 O272072 O272073 O272074 O272075 O272075 O272075 O272076 O272076 O272076 O272076 O272077 O272077 O272077 O272077 O272077 O272078 O272078 O272078 O272079 O27 | stent(s) | Open Approach | 3607 | 027205Z |
| Bifurcation, with Three Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 0272072 3607 Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 0272072 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting drug-eluting coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting coronary artery 027207Z Grid drug-eluting drug-eluting coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Four or More Drug-eluting coronary artery stent(s) O272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) O27207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Three Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery Bifurcation, with Four or More Drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, green of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Dilation of Coronary Artery, Three Arteries, green artery drug-eluting Insertion of drug-eluting Elifurcation, with Drug-eluting Intraluminal coronary artery | | Intraluminal Devices, Open Approach | 3607 | 0272066 |
| with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting | Insertion of | | | |
| 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting insertion of drug-eluting coronary artery coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z Graph Grap | es, coronary artery | with Three Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal 027207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery drug-eluting drug-eluting coronary artery | stent(s) | Open Approach | 3607 | 027206Z |
| Bifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Insertion of drug-eluting coronary artery | Insertion of | | | |
| 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Four or More Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | stent(s) | Intraluminal Devices, Open Approach | 3607 | 0272076 |
| with Four or More Drug-eluting Intraluminal coronary artery 3607 Devices, Open Approach stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | 0 0 | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | l coronary artery | with Four or More Drug-eluting Intraluminal | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | Devices, Open Approach | 3607 | 027207Z |
| Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| | drug-eluting | | | |
| 0272346 3607 Device, Percutaneous Approach | coronary artery | Bifurcation, with Drug-eluting Intraluminal | | |
| Jeney | stent(s) | Device, Percutaneous Approach | 3607 | 0272346 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Drug-eluting Intraluminal Device, coronary artery | coronary artery | with Drug-eluting Intraluminal Device, | | |
| 027234Z 3607 Percutaneous Approach stent(s) | stent(s) | Percutaneous Approach | 3607 | 027234Z |
| Dilation of Coronary Artery, Three Arteries, Insertion of | Insertion of | Dilation of Coronary Artery, Three Arteries, | | |
| Bifurcation, with Two Drug-eluting drug-eluting | drug-eluting | Bifurcation, with Two Drug-eluting | | |
| Intraluminal Devices, Percutaneous coronary artery | coronary artery | Intraluminal Devices, Percutaneous | | |
| 0272356 3607 Approach stent(s) | stent(s) | Approach | 3607 | 0272356 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Two Drug-eluting Intraluminal Devices, coronary artery | | | | |
| 027235Z 3607 Percutaneous Approach stent(s) | | | 3607 | 027235Z |


| | | Dilation of Coronary Artory Four or Moro | Insertion of |
|---|---|---|---|
| | | Dilation of Coronary Artery, Four or More | |
| | | Arteries, Bifurcation, with Two Drug-eluting | drug-eluting |
| 0273456 | 3607 | Intraluminal Devices, Percutaneous | coronary artery |
| 0273450 | 3607 | Endoscopic Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Two Drug-eluting Intraluminal | drug-eluting |
| 027345Z | 3607 | Devices, Percutaneous Endoscopic | coronary artery |
| 0273432 | 3007 | Approach Dilation of Coronary Artery, Four or More | stent(s) Insertion of |
| | | Arteries, Bifurcation, with Three Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 0273466 | 3607 | Endoscopic Approach | stent(s) |
| 0273400 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Three Drug-eluting Intraluminal | drug-eluting |
| | | Devices, Percutaneous Endoscopic | coronary artery |
| 027346Z | 3607 | Approach | stent(s) |
| 0275402 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries, Bifurcation, with Four or More | drug-eluting |
| | | Drug-eluting Intraluminal Devices, | coronary artery |
| 0273476 | 3607 | Percutaneous Endoscopic Approach | stent(s) |
| 0270770 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Four or More Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 027347Z | 3607 | Endoscopic Approach | stent(s) |
| 0270172 | 3007 | 211doscopie i ippi oddi. | Insertion of |
| | | | drug-eluting |
| | | | coronary artery |
| NoPCS | 3607 | | stent(s) |
| СРТ | | | 100 |
| | - | | |
| 92980 | | | |
| 92981 | | | |
| 92981<br>92928 | 1 | | |
| 92928 | - | | |
| 92928<br>92929 | - | | |
| 92928<br>92929<br>92933 | <br> -<br> -<br> - | | |
| 92928<br>92929 | - | | |
| 92928<br>92929<br>92933 | ICD9 Dx | Long DeslCD10 | LongDesICD9 |
| 92928<br>92929<br>92933<br>92934 | ICD9 Dx | Long DesiCD10 | Postmyocardial |
| 92928<br>92929<br>92933<br>92934 | ICD9 Dx<br>4110 | LongDesICD10 Dressler's syndrome | _ |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Dressler's syndrome | Postmyocardial |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx | | Dressler's syndrome Unstable angina | Postmyocardial infarction syndrome |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx<br>1241 | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx<br>1241 | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92928<br>92929<br>92933<br>92934<br>ICD10 Dx<br>1241 | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 I25720 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 I25720 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of native coronary | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 I25720 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |


Depression


Anxiety


Bipolar disorder


Schizophrenia


# Appendix A Dementia risk factors


### Smoking


OR dispensing of: At least one nicotine or varenicline prescription

### Mammography


Colonoscopy


**CPT**45378
45379

110

Appendix A Lifestyle factors and markers for healthy behavior

| 45380 |
|-------|
| 45381 |
| 45382 |
| 45383 |
| 45384 |
| 45385 |
| 45386 |
| 45387 |
| 45388 |
| 45389 |
| 45390 |
| 45391 |
| 45392 |
| HCPCS |
| G0105 |
| G0121 |

## Fecal occult blood test


### Influenza vaccination


| 90655 |
|-------|
| 90656 |
| 90657 |
| 90658 |
| 90659 |
| 90660 |
| 90724 |
| HCPCS |
| G0008 |

### Pneumococcal vaccination


Appendix A Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

## Herpes zoster vaccination


### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

### Healthcare utilization measures

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

### Number of rheumatologist visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

66 = Rheumatology (eff 5/92) Note: during 93/94 DMERC also used this to mean medical supply company with respiratory therapist

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99000 | 99141 | 99249 | 99347 | 99450 | 99603 |
| 99001 | 99142 | 99250 | 99348 | 99454 | 99604 |
| 99002 | 99143 | 99251 | 99349 | 99455 | 99605 |
| 99003 | 99144 | 99252 | 99345 | 99456 | 99606 |
| 99004 | 99145 | 99253 | 99350 | 99460 | 99607 |
| 99005 | 99148 | 99254 | 99351 | 99461 | 99615 |
| 99006 | 99149 | 99255 | 99352 | 99462 | 99649 |
| 99010 | 09915 | 99256 | 99353 | 99463 | 99675 |
| 99011 | 99150 | 9925S | 99354 | 99464 | 99684 |
| 99012 | 99160 | 99261 | 99355 | 99465 | 99700 |
| 99014 | 99163 | 99262 | 99356 | 99466 | 99703 |
| 99015 | 99166 | 99263 | 99357 | 99467 | 99707 |
| 99020 | 99170 | 99270 | 99358 | 99468 | 99713 |
| 99023 | 99171 | 99271 | 99359 | 99469 | 99714 |

| 99024 99172 99272 99350 99471 99737 99025 99173 99274 99360 99471 99732 99026 99174 99274 99361 99475 99762 99027 99175 99275 99362 99475 99762 99028 99178 99280 99363 99476 99770 99032 99183 99280 99363 99477 99770 99032 99183 99281 99364 99477 99772 99038 99184 99282 99365 99478 99776 99038 99185 99284 99367 99479 99780 99039 99186 99284 99367 99480 99799 99040 99188 99284 99367 99480 99799 99041 99180 99286 99371 99482 99381 99041 99190 99286 99371 99485 99801 99042 99191 99288 99373 99485 99802 99047 99195 99288 99373 99486 99803 99048 99199 99200 99375 99487 99806 99049 99049 99191 99289 99376 99489 99810 99049 99049 99200 99375 99489 99810 99051 99200 99292 99377 99489 99810 99051 99200 99292 99377 99489 99811 99051 99200 99292 99377 99489 99811 99052 99203 99378 99495 99383 99384 99810 99054 99200 99292 99377 99489 99811 99059 99009 99200 99399 99399 99399 99381 99309 99009 99200 99399 993999 99399 993999 99399 9939 | | | | | | |
|---|---|---|---|---|---|---|
| 99026 99174 99274 99361 99475 9976 99776 99027 99178 99280 99362 99475 99770 99028 99178 99280 99383 99476 99770 99032 99183 99281 99384 99282 99385 99478 99776 99038 99188 99282 99385 99478 99776 99038 99188 99282 99385 99478 99776 99038 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99779 99039 99186 99284 99367 99480 99779 99039 99180 99286 99271 99480 99780 99780 99286 99271 99485 99801 99002 99180 99286 99277 99485 99801 99002 99190 99286 99277 99485 99801 99002 99190 99286 99277 99485 99801 99002 9919190 99286 99277 99485 99801 99004 99190 99286 99277 99485 99801 99004 99190 99286 99277 99485 99801 99004 99286 99290 99277 99485 99802 99277 99485 99802 99279 99289 99289 99277 99485 99802 99279 99289 99279 99289 99289 99279 99289 99289 99279 99289 | 99024 | 99172 | 99272 | 9935D | 99470 | 99717 |
| 99027 99175 99275 99362 99475 99762 997028 99178 992028 99178 99203 99318 99281 99365 99476 99777 99772 99035 99183 99281 99365 99476 99776 99772 99035 99184 99283 99366 99479 99780 99036 99185 99283 99366 99479 99780 99039 99185 99283 99366 99479 99780 99039 99186 99284 99367 99480 99799 99780 99040 99188 99285 99286 99377 99480 99799 99790 992040 99188 99286 99371 99482 99372 99486 99801 99204 99190 99286 99377 99480 99399 99304 99190 99286 99377 99486 99800 99999 99047 99195 99286 99377 99486 99800 99049 99049 99199 99290 99375 99488 99801 99049 99049 99199 99290 99375 99488 99811 99060 99291 99376 99489 99814 99050 9920 99378 99496 99881 99801 99051 99202 99378 99496 99881 99060 99201 99202 99377 99490 99814 99050 99200 99200 99378 99496 99881 99060 99200 99200 99200 99378 99496 99881 99060 99200 99200 99200 99200 99200 99200 99200 99300 9930 | 99025 | 99173 | 99273 | 99360 | 99471 | 99732 |
| 99027 99175 99275 99362 99475 99762 997028 99178 992028 99178 99203 99318 99281 99365 99476 99777 99772 99035 99183 99281 99365 99476 99776 99772 99035 99184 99283 99366 99479 99780 99036 99185 99283 99366 99479 99780 99039 99185 99283 99366 99479 99780 99039 99186 99284 99367 99480 99799 99780 99040 99188 99285 99286 99377 99480 99799 99790 992040 99188 99286 99371 99482 99372 99486 99801 99204 99190 99286 99377 99480 99399 99304 99190 99286 99377 99486 99800 99999 99047 99195 99286 99377 99486 99800 99049 99049 99199 99290 99375 99488 99801 99049 99049 99199 99290 99375 99488 99811 99060 99291 99376 99489 99814 99050 9920 99378 99496 99881 99801 99051 99202 99378 99496 99881 99060 99201 99202 99377 99490 99814 99050 99200 99200 99378 99496 99881 99060 99200 99200 99200 99378 99496 99881 99060 99200 99200 99200 99200 99200 99200 99200 99300 9930 | 99026 | 99174 | 99274 | 99361 | 99472 | 99736 |
| 99028 99178 99280 99364 99477 99770 99032 99184 99281 99364 99477 99770 99035 99184 99282 99365 99478 99776 99038 99186 99282 99365 99478 99776 99038 99186 99284 93667 99480 99776 99038 99186 99284 93667 99480 99779 99041 99180 99286 99371 99482 99780 99041 99191 99287 99286 99371 99482 993602 99045 99191 99287 99288 99373 99485 99302 99045 99195 99289 99373 99485 99302 99045 99195 99289 99374 99487 99806 99049 99049 99195 99290 99375 99488 99374 99488 99311 99049 99200 9921 99376 99488 99371 99480 993811 99059 99202 99203 99377 99490 99381 99381 99059 99202 99203 99377 99490 99381 99381 99059 99202 99203 99379 99496 99381 99059 99205 | | | | | | |
| 99032 99183 99281 99364 99477 99772 99035 99184 99282 99365 9478 99776 99038 99185 99284 99367 99480 99780 99039 99186 99284 99367 99480 99799 99039 99186 99285 99368 99481 9979A 99041 99190 99286 99271 99482 99381 99041 99190 99286 99271 99482 99382 99042 99111 99286 99271 99485 99801 99043 99191 99286 99271 99485 99802 99047 99195 99288 99374 99485 99803 99047 99195 99288 99374 99487 99803 99048 99199 99290 99375 99488 99810 99049 99200 99291 99376 99489 99811 99050 99201 99292 99377 99490 99381 99051 99202 99293 99378 99496 99833 99054 99205 99296 99381 99494 99399 99054 99206 99296 99381 99498 99841 99056 99206 99296 99381 99499 99841 99056 99207 99298 99382 99499 99849 99058 99207 99298 99383 99500 99804 99069 99208 9930 99384 99501 99881 99060 99208 99209 9930 99385 99502 99899 99060 99208 9930 99385 99502 99899 99061 99208 9930 99385 99502 99899 99063 99208 9930 99385 99502 99899 99064 99208 9930 99385 99502 99899 99065 99208 9930 99385 99502 99899 99066 99208 9930 99385 99502 99899 99071 99208 9930 99385 99502 99899 99071 99208 9930 99387 99505 99309 99307 99208 9930 9938 9930 99385 99502 99899 99071 99208 9930 99387 99505 99300 99891 99070 99208 9930 99387 99505 99309 99007 99208 99309 9930 99385 99502 99899 99071 99210 99303 99337 99505 99907 99072 99210 99303 99337 99505 99907 99073 99210 99303 99305 99505 99907 99074 99210 99303 99305 99505 99907 99075 99211 99303 99305 99505 99907 99076 99217 99310 99303 99397 99501 99907 99077 99210 99303 99305 99505 99909 9910 99006 | | | | | | |
| 99035 99184 99282 99365 99478 99776 99038 99186 99284 99366 9477 99780 99039 99186 99284 99367 99480 99799 99030 99186 99284 99367 99480 99799 99040 99188 99285 99368 9481 99793 99041 99190 99286 9271 99482 99801 99042 99191 99287 99372 39485 99802 99043 99195 99288 99373 99486 99802 99044 99195 99289 99374 99487 99806 99048 99199 99290 99375 99488 99811 99049 99200 99201 99376 99488 99811 99050 99201 99376 99489 99811 99050 99201 99377 99490 99381 99051 99202 9923 99377 99490 99814 99051 99202 9923 99377 99490 99814 99052 99204 99295 99380 99495 99821 99053 99204 99295 99380 99497 99880 99881 99054 99206 99296 99381 99498 99841 99056 99206 99297 99382 99499 99881 99840 99058 99206 99297 99382 99499 99881 99841 99058 99206 99297 99382 99499 99881 99806 99060 99201 99200 99201 99379 99496 99881 99058 99206 99207 99382 99379 99498 99841 99058 99206 99207 99382 99498 99841 99058 99206 99207 99382 99499 99881 99058 99207 99382 99389 | | | | | | |
| 99038 99186 99284 99367 99480 99799 9040 99188 99285 92368 99480 99799 9041 99180 99286 92371 99482 99301 9042 99191 99286 99371 99482 99801 9042 99191 99288 99373 99485 99803 9044 99192 99288 99373 99486 99803 9047 99195 99288 99374 99487 99803 9048 99199 99290 99375 99488 99810 9008 99199 99290 99375 99488 99810 9008 99199 99290 99375 99488 99810 9008 99201 99292 99377 99480 99814 9009 99201 99292 99377 99480 99814 9001 99202 99293 99378 99495 99821 9002 99203 99294 99377 99490 99814 9005 99206 99206 99380 99497 99848 9008 99199 99206 99389 99496 99881 9009 99200 99209 99378 99496 99883 9001 99200 99209 99378 99496 99881 9002 99208 99209 99378 99496 99881 9003 99206 99206 99389 99389 99497 99849 9005 99206 99206 99381 99499 99881 99841 90056 99206 99206 99381 99497 99881 90056 99206 99206 99383 99500 99884 99881 90050 99207 99228 99383 99500 99884 99881 99806 90208 99209 99309 99384 99500 99884 99806 99206 99 | | | | | | |
| 99033 99186 99285 99386 99481 99799 99001 99188 99285 99386 99481 99799 99001 99188 99286 99371 99482 99801 99042 99191 99286 99371 99485 99803 99043 99191 99288 99373 99485 99806 99047 99195 99288 99373 99486 99803 99047 99195 99288 99373 99486 99806 99048 99199 99290 99376 99488 99377 99488 99381 99048 99199 99200 99291 99376 99489 99811 99050 99200 99291 99376 99489 99811 99050 99202 99293 99378 99495 99495 99495 99495 99496 99505 99204 99292 99378 99496 99497 99406 99295 99296 99383 99497 99406 99295 99296 99383 99497 99406 99295 99296 99383 99497 99406 99296 99296 99383 99498 99498 99406 99296 99299 99383 99500 99296 99384 99500 99296 99385 99500 99296 99385 99500 99296 99385 99500 99296 99296 99385 99500 99596 99296 99385 99500 99596 99386 99500 99200 99299 99385 99500 99596 99386 99500 99296 99386 99500 99596 99386 99500 99596 | 99035 | 99184 | 99282 | 99365 | 99478 | 99776 |
| 99040 99188 99285 99388 99481 9979A 99001 99041 99191 99286 99771 99485 99802 99191 99287 99288 99273 99486 99802 99047 99191 99288 99273 99486 99802 99047 99195 99288 99274 99487 99806 99806 99003 99047 99195 99289 99374 99487 99886 99806 99008 99009 99290 99290 99375 99488 99810 99009 99009 99290 99290 99376 99489 99811 99000 99291 99376 99489 99811 99000 99291 99376 99490 99814 99000 99291 99377 99490 99814 99000 99290 99290 99378 99496 99833 990052 99203 99294 99379 99389 99496 99833 99055 99206 99206 99206 99206 99206 99207 99295 99380 99497 99884 99006 99206 99206 99296 99381 99498 99881 99006 99206 99206 99296 99381 99498 99881 99006 99206 99206 99296 99381 99499 99881 99006 99206 99206 99206 99296 99381 99499 99881 99006 99206 99206 99299 99384 99500 99894 99006 99206 | 99038 | 99185 | 99283 | 99366 | 99479 | 99780 |
| 99040 99188 99285 99388 99481 9979A 99001 99041 99191 99286 99771 99485 99802 99191 99287 99288 99273 99486 99802 99047 99191 99288 99273 99486 99802 99047 99195 99288 99274 99487 99806 99806 99003 99047 99195 99289 99374 99487 99886 99806 99008 99009 99290 99290 99375 99488 99810 99009 99009 99290 99290 99376 99489 99811 99000 99291 99376 99489 99811 99000 99291 99376 99490 99814 99000 99291 99377 99490 99814 99000 99290 99290 99378 99496 99833 990052 99203 99294 99379 99389 99496 99833 99055 99206 99206 99206 99206 99206 99207 99295 99380 99497 99884 99006 99206 99206 99296 99381 99498 99881 99006 99206 99206 99296 99381 99498 99881 99006 99206 99206 99296 99381 99499 99881 99006 99206 99206 99206 99296 99381 99499 99881 99006 99206 99206 99299 99384 99500 99894 99006 99206 | 99039 | 99186 | 99284 | 99367 | 99480 | 99799 |
| 99041 99190 99287 99371 99482 99801 99042 99191 99287 99372 99486 99803 99047 99192 99288 99373 99486 99803 99047 99195 99288 99374 99486 99803 99048 99199 99290 99375 99488 99810 99048 99199 99290 99375 99488 99810 99049 99000 99291 99376 99489 99811 99050 99200 99291 99376 99489 99811 99050 99200 99292 99377 99490 99381 99050 99202 99293 99378 99495 99821 99052 99293 99378 99495 99821 99052 99293 99378 99495 99821 99052 99293 99378 99496 99821 99056 99206 99293 99380 99497 99494 99381 99056 99206 99297 99382 99380 99497 99494 99381 99056 99206 99297 99383 99499 99881 99058 99206 99297 99383 99499 99881 99058 99206 99297 99383 99499 99881 99058 99206 99299 99380 99399 99300 | | | | | | |
| 99042 99191 99288 99372 99485 99802 99045 99192 99288 99374 99486 99802 99047 99195 99288 99374 99487 99806 99049 99199 99290 99375 99488 99811 99049 99200 99291 99375 99488 99811 99059 99291 99376 99489 99811 99051 99292 99377 99490 98814 99051 99202 99292 99377 99490 98814 99051 99203 99203 99293 99378 99496 99881 99052 99203 99204 99292 99378 99496 99833 99053 99204 99295 99380 99496 99833 99205 99205 99206 99295 99380 99497 99496 99831 99205 99206 99297 99380 99498 99498 99491 99056 99206 99206 99297 99382 99499 99881 99056 99206 99297 99383 99500 99206 99299 99384 99501 99897 99003 99208 99299 99384 99501 99897 99003 99208 99299 99384 99501 99897 99003 99208 99209 99390 99386 99500 99209 9930 9930 9930 9930 9930 9930 9 | | | | | | |
| 99045 99192 99288 99373 99486 99803 99047 99195 99296 99274 99487 99806 99047 99195 99290 99375 99488 99810 99009 99200 99291 99376 99489 99811 99050 99376 99489 99811 99050 99202 99293 99378 99495 99812 99051 99062 99293 99378 99495 99812 99052 99203 99293 99378 99495 99812 99052 99204 99295 99378 99496 99833 99064 99295 99296 99381 99496 99833 99065 99206 99296 99381 99496 99383 99496 99206 99296 99383 99497 99840 99056 99296 99383 99496 99881 99056 99296 99383 99500 99296 99383 99500 99894 99060 99299 9930 9930 99385 99500 99894 99060 99299 9930 99385 99500 99899 99000 99200 99300 99385 99502 99899 99006 99200 99300 99385 99502 99899 99001 99070 99200 99300 99385 99502 99899 99070 99200 99300 99385 99502 99899 99070 99200 99300 99385 99506 99506 99070 99200 99300 99385 99506 99506 99070 99200 99300 99385 99506 99506 99070 99200 99300 99385 99506 99506 99070 99200 99300 99385 99506 99907 99070 99200 99300 99300 99385 99506 99907 99070 99200 99300 99300 99386 99500 99910 99070 99200 99300 99300 99386 99500 99910 99070 99200 99300 99300 99386 99500 99910 99070 99200 99300 99300 99385 99506 99907 99071 99210 99303 99305 99506 99911 99307 99211 99303 99305 99506 99911 99075 99211 99306 99339 99506 99911 99076 99213 99306 99339 99506 99914 99079 99215 99306 99339 99512 99913 99076 99215 99306 99339 99512 99921 99078 99215 99306 99339 99512 99921 99079 99215 99310 99306 99339 99512 99921 99079 99215 99310 99400 99513 99940 99216 99300 99319 99400 99551 99319 99000 99215 99311 99400 99551 99910 99000 99215 99311 99400 99551 99910 99000 99215 99311 99400 99551 99911 99000 99215 99311 99400 99551 99919 99000 99215 99311 99400 99551 99919 99000 99215 99311 99400 99551 99919 99000 99215 99311 99400 99551 99919 99000 99215 99311 99400 99550 99990 99000 99215 99311 99400 99550 99990 99000 99215 99311 99400 99550 99990 99000 99215 99311 99400 99550 99990 99000 99215 99311 99400 99550 99990 99000 99215 99311 99322 99400 99550 99990 99900 99215 99311 99323 99331 99400 99550 99990 99900 99215 99331 99332 99400 99550 99990 999 | | | | | | |
| 99047 99195 99289 99374 99487 99806 99048 99191 99290 99275 99488 99810 99048 9919 99200 99291 99375 99489 99811 99049 99200 99291 99376 99489 99811 99050 99201 99201 99376 99489 99811 99051 99201 99202 99377 99490 99814 99051 99202 9923 99377 99490 99814 99051 99203 99378 99496 99833 99052 99203 99204 99295 99380 99496 99833 99053 99205 99205 99205 99380 99496 99833 990554 99205 99206 99296 99381 99498 99488 99841 99056 99207 99382 99498 99881 99056 99207 99382 99498 99881 99056 99207 99382 99499 99881 99056 99208 99209 99384 99500 99894 99063 99208 99209 99384 99501 99887 99065 99208 99209 99386 99500 99889 99065 9920A 99300 99386 99503 99901 99065 9920A 99300 99386 99503 99901 99070 9920X 99301 99387 99505 99907 9920X 99301 99387 99505 99907 99071 09921 99302 99339 99364 99505 99907 99071 09921 99302 99339 99367 99505 99907 99071 09921 99302 99339 99360 99389 99505 99907 99071 09921 99304 99304 99339 99505 99907 99074 99211 99303 99339 99505 99907 99074 99211 99304 99339 99309 99505 99907 99075 99212 99305 99339 99505 99907 99075 99212 99306 99309 9 | | | | | | |
| 99048 99199 99200 99291 99375 99488 99810 99049 99200 99291 99376 99489 99811 99050 99201 99201 99376 99480 99814 99051 99202 99203 99293 99378 99495 99814 99052 99203 99204 99204 99379 99496 99833 99053 99204 99205 99380 99497 99840 99881 99053 99204 99205 99380 99497 99840 99881 99056 99206 99381 99499 99881 99056 99206 99206 99381 99499 99881 99056 99206 99206 99381 99499 99881 99056 99206 99207 99382 99499 99881 99056 99206 99207 99382 99499 99881 99050 99207 99299 99384 99500 99899 99060 99200 99200 99200 99300 99385 99500 99897 99065 99200 99200 99300 99385 99500 99897 99065 99200 99300 99386 99500 99899 99000 99000 99200 99300 99386 99500 99900 99000 99000 99200 99300 99386 99500 99900 99000 99000 99200 99300 99386 99500 99900 99000 99000 99200 99300 99386 99500 99910 99000 | | 99192 | | | 99486 | |
| 99049 99200 99201 99376 99483 99811 99050 99201 99292 99377 99490 99814 99051 99202 99377 99496 99814 99051 99202 99203 99378 99496 99831 99052 99203 99203 99204 99379 99496 99833 99503 99204 99295 99380 99497 99840 99840 99205 99205 99206 99381 99498 99841 99056 99205 99206 99381 99498 99881 99056 99207 99382 9449 99881 99058 99207 99382 9449 99881 99058 99207 99383 99500 99894 99500 99208 99209 99384 99501 99897 99060 99208 99209 99384 99501 99897 99060 99208 99209 99386 99500 99899 99399 99386 99503 99901 99070 99200 99300 99385 99503 99901 99070 99200 99300 99386 99503 99901 99070 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99387 99506 99200 99301 99301 99387 99506 99200 99301 99 | 99047 | 99195 | 99289 | 99374 | 99487 | 99806 |
| 99050 99201 99202 99377 99490 99814 99051 99202 99293 99378 99495 99813 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99058 99206 99297 99382 99499 99881 99058 99206 99297 99383 99500 99884 99059 99206 99297 99383 99500 99884 99050 99206 99299 99384 99501 99897 99060 99208 99299 99384 99501 99897 99060 99208 99299 99384 99501 99897 99060 99208 99300 99330 99335 99502 99889 99060 99208 99299 99384 99501 99897 99070 9920X 99301 9930 99386 99503 99901 99070 9920X 99301 9930 99386 99503 99901 99071 99210 99303 99302 99391 99506 99910 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99394 99508 99913 99076 99214 99307 99396 99396 99914 99077 99216 99306 99399 99396 99919 99079 99215 99306 99396 99396 99919 99079 99215 99308 99397 99511 99907 99078 99216 99308 99397 99511 99907 99079 99215 99308 99397 99511 99907 99078 99217 99310 99400 99399 99519 99919 99079 99215 99308 99397 99511 99907 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99929 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99078 99217 99310 99400 99513 99920 99079 99215 99308 99399 99551 99990 99089 99217 99311 99400 99551 99991 99078 99217 99313 99401 99551 99991 99079 99215 99318 99400 99551 99990 99089 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99319 99317 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99215 99318 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99319 99319 99400 99551 99990 99099 99214 99331 99401 99556 99990 99099 99214 99331 99404 99556 99990 99110 99226 99331 99446 99556 99999 99110 99236 99339 99344 99566 99999 99111 99236 99344 99446 99589 99999 99113 99244 99344 99448 99448 99660 | 99048 | 99199 | 99290 | 99375 | 99488 | 99810 |
| 99051 99202 99293 99378 99495 99821 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99056 99207 99298 99383 99500 99884 99056 99208 99299 99384 99501 99879 99060 99208 99299 99384 99501 99877 99063 99208 99299 99384 99501 99877 99065 9920A 99300 99386 99502 99889 99070 9920A 99300 99386 99503 99901 99071 09921 99302 99391 99505 99907 99071 09921 99302 99391 99505 99907 99074 99211 99304 99393 99506 99910 99075 99212 99305 99394 99506 99910 99076 99213 99306 99394 99506 99910 99077 99210 99307 99399 99507 99078 99214 99307 99399 99509 99914 99079 99215 99306 99399 99509 99914 99079 99216 99309 99399 99510 99919 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99939 99080 99218 99311 99401 99554 99991 99080 99218 99311 99401 99552 99940 99080 99216 99315 99404 99539 99942 99099 99221 99315 99408 99555 99949 99099 99222 99317 9940 99555 99949 99099 99223 99316 9940 99555 99999 99010 99224 99323 99411 99556 99999 99110 99226 99327 9940 99555 99999 99110 99226 99327 9940 99555 99999 99110 99227 99331 99406 99555 99999 99110 99228 99331 99406 99555 99999 99110 99228 99331 99406 99555 99999 99110 99228 99331 99432 99566 99999 99111 99231 99332 99446 99556 99999 99111 99231 99331 99446 99566 99999 99114 99246 99344 99446 99593 99214 99133 | 99049 | 99200 | 99291 | 99376 | 99489 | 99811 |
| 99051 99202 99293 99378 99495 99821 99052 99203 99294 99379 99496 99833 99053 99204 99295 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99206 99297 99382 99499 99881 99056 99207 99298 99383 99500 99884 99056 99208 99299 99384 99501 99879 99060 99208 99299 99384 99501 99877 99063 99208 99299 99384 99501 99877 99065 9920A 99300 99386 99502 99889 99070 9920A 99300 99386 99503 99901 99071 09921 99302 99391 99505 99907 99071 09921 99302 99391 99505 99907 99074 99211 99304 99393 99506 99910 99075 99212 99305 99394 99506 99910 99076 99213 99306 99394 99506 99910 99077 99210 99307 99399 99507 99078 99214 99307 99399 99509 99914 99079 99215 99306 99399 99509 99914 99079 99216 99309 99399 99510 99919 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99939 99080 99218 99311 99401 99554 99991 99080 99218 99311 99401 99552 99940 99080 99216 99315 99404 99539 99942 99099 99221 99315 99408 99555 99949 99099 99222 99317 9940 99555 99949 99099 99223 99316 9940 99555 99999 99010 99224 99323 99411 99556 99999 99110 99226 99327 9940 99555 99999 99110 99226 99327 9940 99555 99999 99110 99227 99331 99406 99555 99999 99110 99228 99331 99406 99555 99999 99110 99228 99331 99406 99555 99999 99110 99228 99331 99432 99566 99999 99111 99231 99332 99446 99556 99999 99111 99231 99331 99446 99566 99999 99114 99246 99344 99446 99593 99214 99133 | | | | | | |
| 99052 99203 99294 99295 99380 99497 99840 99054 99205 99286 99381 99498 99841 99056 99206 99297 99382 99499 99881 99058 99207 99298 99383 99500 99844 99060 99208 99299 99384 99501 9987 99063 39209 99300 99385 99502 99899 99065 9920A 99300 99386 99503 99897 99065 9920A 99301 99387 99503 99899 99070 9920X 99301 99387 99504 99902 99071 09210 99302 99391 99505 99907 99072 99210 99303 99387 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 9934 99508 999 | | | | | | |
| 99053 99204 9925 99380 99497 99840 99054 99205 99296 99381 99499 99881 99056 99207 99288 99383 99500 99884 99063 99209 99300 99385 99501 99897 99063 9920A 99300 99386 99502 99899 99070 9920A 99300 99386 99503 99901 99071 09921 99301 99387 99504 99902 99071 09921 99302 99393 99505 99907 99072 99210 99303 99393 99505 99907 99074 99211 99304 99393 99507 99910 99075 99212 99305 99393 99507 99912 99076 99212 99305 99334 99508 99913 99078 99212 99307 9936 99510 9907 <t< td=""><td></td><td></td><td></td><td></td><td></td><td></td></t<> | | | | | | |
| 99056 99206 99297 99381 99498 99811 99056 99206 99297 99382 99499 99881 99058 99207 99298 99383 99500 99894 99060 99208 99299 99384 99501 99887 99063 99208 99299 99384 99501 99887 99065 9920A 99300 99385 99502 99899 99075 9920K 99301 99387 99505 99907 99070 9920K 99301 99387 99505 99907 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99508 99914 99078 99214 99306 99395 99509 99914 99079 99215 99308 99397 99511 99920 99078 99216 99308 99397 99511 99920 99078 99216 99308 99397 99511 99920 99078 99216 99308 99399 99512 9921 99077 99217 99308 99399 99512 9921 99078 99216 99309 99399 99512 9921 99079 99216 99309 99399 99512 9921 99078 99216 99309 99399 99512 9921 99079 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99082 9921F 99313 99401 99523 99940 99082 9921F 99313 99404 99539 9942 99090 99220 99317 99407 99552 9949 99091 99220 99317 99407 99553 99949 99091 99220 99317 99407 99555 99949 99091 99220 99317 99409 99554 9959 99091 99220 99317 99409 99554 99999 99011 99225 99324 99412 99557 99999 99104 99227 99326 99429 99559 99999 99104 99227 99326 99429 99559 99999 99104 99226 99327 99446 99559 99999 99110 99238 99347 99447 99566 99999 99112 99238 99347 99447 99566 99999 99124 99339 99447 99566 99999 99124 99344 99349 99447 99560 99999 9913 99246 99344 99447 99660 | | | | | | |
| 99056 99206 99297 99382 99499 99841 99058 99208 99298 99383 99500 99894 99060 99208 99299 99384 99501 99897 99063 99200 9930 99385 99502 99899 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99071 09921 99303 99393 99505 99907 99072 99210 99303 99393 99505 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99334 99508 99913 99076 99213 99306 99339 99509 99914 99078 99214 99307 99396 99510 99919 99078 99216 99309 99399 99512 99921 | 99053 | 99204 | 99295 | 99380 | 99497 | 99840 |
| 99058 99207 99298 99383 99500 99894 99060 99208 99299 99384 99501 99887 99063 99209 9930 99385 99502 99899 99065 9920A 99300 99386 99503 99901 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99073 99211 99304 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99306 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99395 99509 99914 99079 99215 99308 99397 99511 99920 99078 99216 99309 99309 99319 99512 99078 99216 99309 99319 99510 99919 99078 99216 99309 99319 99510 99919 99078 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99311 99082 9921F 99313 99402 99523 99940 99082 9921F 99313 99402 99530 99941 99089 99216 99317 99316 99404 99539 99941 99090 99215 99318 99316 99404 99539 99940 99089 99216 99317 99316 99404 99539 99940 99089 99216 99317 99318 99407 99551 99943 99090 99215 99318 99316 99404 99539 99940 99090 99215 99318 99316 99404 99539 99940 99090 99215 99318 99316 99404 99539 99940 99090 99215 99318 99404 99551 99943 99091 99220 99317 99407 99552 99949 99091 99221 99318 99408 99553 99949 99091 99222 99321 99318 99408 99553 99949 99091 99222 99321 99318 99408 99553 99959 99091 99222 99321 99318 99408 99553 99994 99091 99223 99324 99331 99408 99555 99949 99091 99223 99324 99324 99408 99555 99940 99091 99223 99324 99324 99408 99555 99961 9910 99223 99324 99324 99408 99555 99996 9910 99224 99331 99408 99555 99990 99110 99236 99325 99408 99556 99990 99111 99236 99326 99327 99426 99566 99999 99110 99236 99338 99349 99442 99566 99999 99110 99236 99338 99349 99442 99566 99999 99110 99236 99338 99349 99442 99566 99999 99111 99236 99338 99349 99444 99566 99999 99112 99236 99338 99344 99348 99566 99999 99113 99244 99339 99442 99569 99999 99124 99339 99444 99568 99999 99125 99344 99344 99568 99999 99124 99344 99344 99569 99999 9913 99244 99344 99344 99560 99999 9913 99444 99546 99344 99546 99593 99991 | 99054 | 99205 | 99296 | 99381 | 99498 | 99841 |
| 99060 99208 99299 99384 99501 9987 99063 99209 9930 99385 99502 99899 99070 9920A 99300 99387 99504 99901 99071 099210 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99910 99912 99076 99213 99305 99910 99912 99076 99213 99306 99393 99507 99912 99076 99213 99307 99396 99914 9907 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99319 99512 9902 9907 99216 <td>99056</td> <td>99206</td> <td>99297</td> <td>99382</td> <td>99499</td> <td>99881</td> | 99056 | 99206 | 99297 | 99382 | 99499 | 99881 |
| 99060 99208 99299 99384 99501 9987 99063 99209 9930 99385 99502 99899 99070 9920A 99300 99387 99504 99901 99071 099210 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99910 99912 99076 99213 99305 99910 99912 99076 99213 99306 99393 99507 99912 99076 99213 99307 99396 99914 9907 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99319 99512 9902 9907 99216 <td></td> <td>99207</td> <td></td> <td>99383</td> <td></td> <td></td> | | 99207 | | 99383 | | |
| 99063 99209 9930 99385 99502 99899 99065 9920A 99300 99385 99502 99899 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99392 99506 99910 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99395 99509 99914 99079 99215 99308 99397 99511 99920 99079 99215 99308 99399 99512 99921 99076 99217 99310 99400 99513 99922 99078 99218 99311 99400 99513 99925 99080 99218 99311 99401 99514 99931 99082 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99082 99217 99310 99402 99523 99940 99082 99217 99313 99402 99523 99940 99082 99217 99313 99403 99530 99941 99089 99216 99315 99404 99533 99942 99090 99215 99316 99400 99551 99940 99080 99218 99311 99402 99523 99940 99081 99219 99312 99402 99523 99940 99082 99217 99313 99403 99530 99941 99080 99218 99316 99404 99553 99940 99081 99219 99316 99400 99551 99940 99082 99216 99316 99400 99551 99961 99909 99090 99215 99316 99404 99553 99940 99090 99215 99316 99400 99551 99949 99091 99220 99317 99407 99552 99949 99097 99221 99318 99409 99554 99959 99097 99221 99318 99409 99554 99960 99079 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99318 99409 99554 99959 99091 99222 99321 99338 99409 99554 99960 99091 99224 99338 99409 99554 99960 99091 99225 99324 99400 99556 99999 99110 99226 99327 99426 99559 99999 99110 99236 99337 99426 99560 99999 99110 99236 99337 99426 99560 99999 99111 99236 99337 99441 99566 99999 99111 99236 99337 99441 99566 99999 99111 99236 99337 99441 99566 99999 99112 99236 99337 99444 99568 99999 99113 99234 99339 99344 99566 99999 99114 99236 99337 99444 99568 99999 99114 99236 99337 99444 99568 99999 99114 99236 99337 99444 99569 99999 99114 99236 99337 99444 99569 99999 99124 99349 99444 99569 99999 99124 99349 99444 99569 99999 99135 99244 99344 99446 99593 99214 | | | | | | |
| 99065 9920A 99300 99386 99503 99901 99070 9920K 99301 99387 9950A 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99333 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99926 99078 99218 99311 99400 99513 99925 99080 99218 99311 99400 99513 99925 99080 99218 99311 99400 99513 99925 99082 9921F 99313 99402 99523 9940 99082 9921F 99313 99403 99530 99941 99089 99099 99212 99315 99404 99539 99942 99099 99212 99315 99404 99539 99942 99090 99215 99316 99404 99539 99949 99090 99215 99316 99406 99551 9943 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99099 99221 99321 99408 99553 99969 99099 99222 99321 99408 99553 99969 99099 99222 99321 99409 99554 99960 99079 99221 99318 99408 99553 99969 99099 99222 99321 99409 99554 99960 99099 99222 99321 99409 99554 99960 99099 99222 99321 99409 99556 99969 9910 99226 99325 99324 99412 99555 99961 9910 99226 99325 99326 99329 99411 99556 99969 9910 99229 99321 99329 99409 99558 99999 9910 99229 99321 99409 99558 99969 9910 99229 99329 99329 99409 99556 99969 9910 99229 99329 99329 99409 99556 99999 9910 99229 99329 99329 99409 99556 99999 9910 99229 99329 99329 99409 99556 99999 9910 99229 99329 99329 99409 99559 99999 9910 99229 99329 99329 99329 99409 99559 99999 9910 99229 99329 99329 99329 99409 99559 99999 9910 99229 99329 99329 99329 99409 99559 99999 9910 99229 99329 99 | | | | | | |
| 99070 9920X 99301 99387 99504 99902 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99512 99921 99078 99217 99310 99400 99513 99925 99081 99218 99311 99401 99514 99931 99082 99218 99311 99401 99514 99931 99082 9921F 99312 99402 99523 99940 99089 99216 99315 99404 99539 99542 99099 99215 99316 99404 99539 99941 99099 99215 99316 99404 99539 99942 99099 99215 99316 99404 99553 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99599 99099 99222 99321 99408 99553 99599 99091 99220 99317 99407 99552 99949 99091 99220 99317 99408 99553 99959 99099 99221 99318 99408 99553 99959 99099 99221 99318 99408 99553 99959 99099 99221 99318 99408 99553 99959 99099 99221 99318 99408 99553 99960 99091 99220 99317 99407 99552 99949 99091 99220 99317 99407 99552 99949 99099 99221 99318 99408 99553 99959 99099 99222 99321 99408 99553 99960 99099 99224 99323 99419 99556 99968 99101 99226 99326 99326 99409 99554 99960 99110 99226 99326 99326 99429 99559 99999 99110 99227 99326 99326 99429 99559 99999 99110 99228 99329 99324 99412 99557 99970 99110 99230 99327 99426 99560 99999 99110 99230 99327 99426 99560 99999 99110 99230 99337 99426 99560 99999 99110 99230 99337 99446 99566 99999 99111 99236 99338 99336 99431 99566 99999 99111 99236 99338 99336 99440 99566 99999 99112 99239 99337 99441 99568 99999 99112 99236 99339 99337 99441 99568 99999 99110 99236 99338 99336 99444 99569 99999 99111 99236 99339 99344 99446 99569 99999 99112 99236 99337 99444 99569 99999 99124 99244 99340 99446 99598 99999 99124 99245 99343 99447 99600 9913 99246 99344 99344 99446 99593 99214 | | | | | | |
| 99071 09921 99302 99391 99505 99907 99072 99210 99303 99392 99506 99910 99074 99211 99304 99508 99912 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99214 99307 99511 99920 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99079 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99218 99311 99401 99523 99940 99081 99219 99312 99402 99523 99941 99089 99216 99315 99403 99539 99942 99089 99216 | 99065 | 9920A | 99300 | 99386 | 99503 | 99901 |
| 99072 99210 99303 99392 99506 99910 99074 99211 99304 99333 99507 99912 99075 99212 99306 99394 99508 99913 99076 99213 99306 99395 99500 99914 99078 99214 99307 99396 99510 99919 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99078 99216 99309 99399 99511 99920 99078 99216 99309 99319 99511 99921 99078 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 9982 99216 99315 99402 99530 99941 | 99070 | 9920X | 99301 | 99387 | 99504 | 99902 |
| 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99078 99213 99306 99395 99510 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99512 99921 99078 99216 99300 99313 99921 99078 99216 99300 99313 99921 99079 99217 99310 99400 99513 99921 9907 99217 99310 99401 99514 99931 99080 99218 99311 99401 99514 99931 99082 99217 99315 99402 9953 99942 99091 99216 99315 99406 99551 99943 99091 99220 99317 </td <td>99071</td> <td>09921</td> <td>99302</td> <td>99391</td> <td>99505</td> <td>99907</td> | 99071 | 09921 | 99302 | 99391 | 99505 | 99907 |
| 99074 99211 99304 99393 99507 99912 99075 99212 99305 99394 99508 99913 99078 99213 99306 99395 99510 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99512 99921 99078 99216 99300 99313 99921 99078 99216 99300 99313 99921 99079 99217 99310 99400 99513 99921 9907 99217 99310 99401 99514 99931 99080 99218 99311 99401 99514 99931 99082 99217 99315 99402 9953 99942 99091 99216 99315 99406 99551 99943 99091 99220 99317 </td <td>99072</td> <td>99210</td> <td>99303</td> <td>99392</td> <td>99506</td> <td>99910</td> | 99072 | 99210 | 99303 | 99392 | 99506 | 99910 |
| 99075 99212 99305 99394 99508 99913 99076 99213 99306 99395 99509 99914 99078 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 9921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99081 99219 99312 99402 99523 99940 99082 99216 99313 99403 99530 99941 99089 99216 99315 99404 99539 99942 99090 99215 99316 99406 99551 99943 99090 99215 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 | | | | | | |
| 99076 99213 99306 99395 99509 99914 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99339 99512 99921 99078 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 99215 99316 99404 99539 99942 99001 99220 99317 99407 99551 99949 99007 99215 99318 99408 99551 99949 99097 99221 99318 99408 99553 99959 | | | | | | |
| 99078 99214 99307 99396 99510 99919 99079 99215 99308 99397 99511 99920 99078 99216 99309 99399 99512 99921 99076 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 9931 99081 99219 99312 99402 99533 99940 99082 99216 99313 99403 99530 99941 99089 99216 99315 99404 99539 99942 99090 99215 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99409 99554 9960 99057 99221 9931 99409 99554 9966 <tr< td=""><td></td><td></td><td></td><td></td><td></td><td></td></tr<> | | | | | | |
| 99079 99215 99308 99397 99511 99920 9907B 99216 99309 99319 99512 99921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99408 99554 99960 9957 99223 99321 99408 99555 99961 | 99076 | 99213 | 99306 | 99395 | 99509 | 99914 |
| 9907B 99216 99309 99399 99512 99921 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99408 99553 99959 99097 99221 99321 99409 99554 99960 99057 99223 99321 99409 99554 99960 99057 99223 99324 99419 99556 99961 | 99078 | 99214 | 99307 | 99396 | 99510 | 99919 |
| 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 9922O 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99407 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 99409 99554 99960 99057 99223 99322 99409 99555 99961 99100 99224 99323 99411 99557 99970 | 99079 | 99215 | 99308 | 99397 | 99511 | 99920 |
| 9907E 99217 99310 99400 99513 99925 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 9922O 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99097 99221 99318 99407 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 99409 99554 99960 99057 99223 99322 99409 99555 99961 99100 99224 99323 99411 99557 99970 | 9907B | 99216 | 99309 | 99399 | 99512 | 99921 |
| 99080 99218 99311 99401 99514 99931 99081 99219 99312 99402 99523 99940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 9943 99091 99220 99317 99407 99552 9949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99408 99553 99959 99097 99221 99318 99408 99553 99959 99099 99222 99321 99408 99554 99960 99007 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 < | 9907F | | 99310 | 99400 | 99513 | 99925 |
| 99081 99219 99312 99402 99523 9940 99082 9921F 99313 99403 99530 99941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9988 99104 99227 99326 99420 99558 99989 99110 99230 99327 99426 99560 99990 < | | | | | | |
| 99082 9921F 99313 99403 99530 9941 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 9960 990ST 99223 99322 9940A 99555 9961 99100 99224 99323 99411 99556 9996 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99420 99558 9989 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 | | | | | | |
| 99089 9921G 99315 99404 99539 99942 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99999 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 | | | | | | |
| 99090 9921S 99316 99406 99551 99943 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99999 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 | 99082 | 9921F | 99313 | 99403 | 99530 | 99941 |
| 99091 99220 99317 99407 99552 99949 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 99057 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 99989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99332 99331 99432 99562 99992 99113 99233 99332 99433 99564 99994 99115 99234 99333 99435 99564 99994 | 99089 | 9921G | 99315 | 99404 | 99539 | 99942 |
| 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 9905T 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 <t< td=""><td>99090</td><td>9921S</td><td>99316</td><td>99406</td><td>99551</td><td>99943</td></t<> | 99090 | 9921S | 99316 | 99406 | 99551 | 99943 |
| 99097 99221 99318 99408 99553 99959 99099 99222 99321 99409 99554 99960 9905T 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 9968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 <t< td=""><td>99091</td><td>99220</td><td>99317</td><td>99407</td><td>99552</td><td>99949</td></t<> | 99091 | 99220 | 99317 | 99407 | 99552 | 99949 |
| 99099 99222 99321 99409 99554 99960 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 9991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 9994 99116 99235 99344 99436 99565 99995 99119 99236 99335 99438 99566 99996 <tr< td=""><td></td><td></td><td></td><td></td><td></td><td></td></tr<> | | | | | | |
| 990ST 99223 99322 9940A 99555 99961 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 9991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 < | | | | | | |
| 99100 99224 99323 99411 99556 99968 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99344 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99999 | | | | | | |
| 99101 99225 99324 99412 99557 99970 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 | | | | | | |
| 99102 99226 99325 99420 99558 9989 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 9993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 < | 99100 | | 99323 | 99411 | 99556 | 99968 |
| 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V | 99101 | 99225 | 99324 | 99412 | 99557 | 99970 |
| 99104 99227 99326 99429 99559 09999 99110 99230 99327 99426 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V | 99102 | 99226 | 99325 | 99420 | 99558 | 99989 |
| 99110 99230 99327 9942G 99560 99990 99111 99231 99328 99431 99561 99991 99112 99232 9931 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 | | | 99326 | | 99559 | |
| 99111 99231 99328 99431 99561 99991 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99344 99448 99600 | | | | | | |
| 99112 99232 99331 99432 99562 99992 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99113 99233 99332 99433 99563 99993 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 99996 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99115 99234 99333 99435 99564 99994 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99113 | 99233 | 99332 | 99433 | 99563 | 99993 |
| 99116 99235 99334 99436 99565 99995 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99115 | 99234 | 99333 | 99435 | 99564 | 99994 |
| 99119 99236 99335 99438 99566 99996 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99116 | 99235 | 99334 | 99436 | 99565 | 99995 |
| 99120 99238 99336 99440 99567 99997 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | 99236 | | | 99566 | |
| 99121 99239 99337 99441 99568 99998 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99123 99241 99339 99442 99569 99999 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99714 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99124 99242 99340 99443 99580 9999G 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99214 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | | | | | |
| 99125 99243 99341 99444 99588 9999V 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | | 99241 | 99339 | 99442 | 99569 | 99999 |
| 09913 99244 99342 99446 99593 99Z14 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99124 | 99242 | 99340 | 99443 | 99580 | 9999G |
| 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 99125 | 99243 | 99341 | 99444 | 99588 | 9999V |
| 99135 99245 99343 99447 99600 09914 99246 99344 99448 99601 | 09913 | 99244 | 99342 | 99446 | 99593 | 99Z14 |
| 09914 99246 99344 99448 99601 | | | | | | |
| 99140 99345 99449 99602 | | | | | | |
| | 99140 | 99248 | 99345 | 99449 | 99602 | |



# Appendix A Healthcare utilization measures

| 86140 | 86141 |
|-------|-------|

#### Number of serum creatinine tests

| CPT | |
|-------|-------|
| 80048 | 80054 |
| 80049 | 80069 |
| 80053 | 82565 |

### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| ntestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality Disorders, And Other Nonpsychotic Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.800, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.283, F16.288, F16.980, F16.983, F16.983, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.950, F19.951, F19.96, F19.282, F19.91, F19.982, F19.984, F19.950, F19.950, F19.951, F19.96, F19.282, F19.91, F19.982, F19.984, F19.950, F19.950, F19.951, F19.96, F19.282, F19.91, F19.982, F19.984, F19.950, F19.950, F19.951, F19.96, F19.282, F19.921, F19.982, F19.984, F19.950, F19.950, F19.951, F19.96, F19.282, F19.921, F19.982, F19.984, F19.950, F19.950, F19.951, F19.96, F19.282, F19.939, F19.94, F19.950, F19.951, F19.96, F19.282, F19.951, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, F19.282, F19.951, F19.982, F19.944, F19.950, F19.951, F19.96, F19.282, F19.951, F19.982, F19.951, F19.950, F19.951, F19.96, F19.281, F19.952, F19.951, F19.952, F19.950, F19.951, F19.96, F19.282, F19.951, F19.952, | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-<br>G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | J30-J39 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36<br>(excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | S81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

Osteoporosis

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| encounter and extradural hemorrh consciousness S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | of skull with subarachnoid, subdural, |
|---|---|
| S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | nage unenecified state of |
| S065X0A 80120 Traumatic subdural hemorrhage without loss of consciousness, initial encounter and extradural hemorrh | lage, unspecified state of |
| consciousness, initial encounter and extradural hemorrh | af alvelles ithe authorise has in a subalvisal |
| | · |
| | nage, unspecified state of |
| consciousness | |
| S066X0A 80120 Traumatic subarachnoid hemorrhage without loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, unspecified state of |
| consciousness | |
| S02109A 80121 Fracture of base of skull, unspecified side, initial encounter Closed fracture of base | of skull with subarachnoid, subdural, |
| | nage, with no loss of consciousness |
| | iage, men no ross er consciousness |
| S064X0A 80121 Epidural hemorrhage without loss of consciousness, initial Closed fracture of base | of skull with subarachnoid, subdural, |
| | nage, with no loss of consciousness |
| and extradular nemorn | lage, with no loss of consciousness |
| COCCYOA 20121 Traumatic subdural homographore without loss of Closed fracture of hose | of clault with cubora shootd cubdural |
| | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, with no loss of consciousness |
| | of skull with subarachnoid, subdural, |
| consciousness, initial encounter and extradural hemorrh | nage, with no loss of consciousness |
| | of skull with subarachnoid, subdural, |
| for closed fracture and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S064X1A 80122 Epidural hemorrhage with loss of consciousness of 30 minutes Closed fracture of base | of skull with subarachnoid, subdural, |
| or less, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| | of skull with subarachnoid, subdural, |
| | nage, with brief [less than one hour] |
| loss of consciousness | lage, with bire fless than one floar |
| | af alvelles ith as because the side as the decide |
| | of skull with subarachnoid, subdural, |
| | nage, with brief [less than one hour] |
| loss of consciousness | |
| S065X2A 80122 Traumatic subdural hemorrhage with loss of consciousness of Closed fracture of base | of skull with subarachnoid, subdural, |
| 31 minutes to 59 minutes, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S066X1A 80122 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| consciousness of 30 minutes or less, initial encounter and extradural hemorrh | nage, with brief [less than one hour] |
| loss of consciousness | |
| S066X2A 80122 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base | of skull with subarachnoid, subdural, |
| <u> </u> | nage, with brief [less than one hour] |
| | lage, with bire fless than one hoar] |
| loss of consciousness S03100A 90133 Eracture of base of skull unspecified side initial ensembles. Closed fracture of base | of ckull with subarasbasid subdume |
| | of skull with subarachnoid, subdural, |
| | nage, with moderate [1-24 hours] los |
| of consciousness | |
| ' | of skull with subarachnoid, subdural, |
| hours 59 minutes, initial encounter and extradural hemorrh | nage, with moderate [1-24 hours] los |
| of consciousness | |
| S064X4A 80123 Epidural hemorrhage with loss of consciousness of 6 hours to Closed fracture of base | of skull with subarachnoid, subdural, |
| 24 hours, initial encounter and extradural hemorrh | nage, with moderate [1-24 hours] los |
| of consciousness | |
| | of skull with subarachnoid, subdural, |
| - 2002/201 - COTES - FILAMINATIC SAPANTAL HEIDOLTHAGE WITH 1033 OF CONSCIONACION ACTURE OF DATE | nage, with moderate [1-24 hours] los |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh | |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness | of clault with cubarachasid subdiving |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of Closed fracture of base of the consciousness of Closed fracture of the consciousness of Closed fracture of Closed fracture of Closed fracture of Closed fra | |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh | · |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness | nage, with moderate [1-24 hours] los |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness S066X3A 80123 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base of consciousness | nage, with moderate [1-24 hours] lost |
| 1 hour to 5 hours 59 minutes, initial encounter and extradural hemorrh of consciousness S065X4A 80123 Traumatic subdural hemorrhage with loss of consciousness of 6 hours to 24 hours, initial encounter and extradural hemorrh of consciousness S066X3A 80123 Traumatic subarachnoid hemorrhage with loss of Closed fracture of base of consciousness | of skull with subarachnoid, subdural, nage, with moderate [1-24 hours] loss of skull with subarachnoid, subdural, nage, with moderate [1-24 hours] loss |


| | | T |
|---|---|---|
| 8083 | Fracture of superior rim of left pubis, initial encounter for open fracture | Open fracture of pubis |
| 8083 | Fracture of superior rim of unspecified pubis, initial encounter for open fracture | Open fracture of pubis |
| 8083 | Other specified fracture of right pubis, initial encounter for | Open fracture of pubis |
| 8083 | Other specified fracture of left pubis, initial encounter for | Open fracture of pubis |
| 8083 | Other specified fracture of unspecified pubis, initial encounter | Open fracture of pubis |
| 80841 | Unspecified fracture of right ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | Unspecified fracture of left ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | Displaced avulsion fracture of right ilium, initial encounter | Closed fracture of ilium |
| 80841 | Displaced avulsion fracture of left ilium, initial encounter for | Closed fracture of ilium |
| 80841 | closed fracture Displaced avulsion fracture of unspecified ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Nondisplaced avulsion fracture of right ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Nondisplaced avulsion fracture of left ilium, initial encounter | Closed fracture of ilium |
| 80841 | for closed fracture Nondisplaced avulsion fracture of unspecified ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Other fracture of right ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | fracture Other fracture of left ilium, initial encounter for closed | Closed fracture of ilium |
| | fracture | Closed fracture of ilium |
| | closed fracture | |
| | closed fracture | Closed fracture of ischium |
| | closed fracture | Closed fracture of ischium |
| 80842 | for closed fracture | Closed fracture of ischium |
| 80842 | Displaced avulsion fracture of left ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Displaced avulsion fracture of unspecified ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of right ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of left ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of unspecified ischium, initial | Closed fracture of ischium |
| 80842 | Other specified fracture of right ischium, initial encounter for | Closed fracture of ischium |
| 80842 | Other specified fracture of left ischium, initial encounter for | Closed fracture of ischium |
| 80842 | Other specified fracture of unspecified ischium, initial | Closed fracture of ischium |
| 80849 | Fracture of unspecified parts of lumbosacral spine and pelvis, | Closed fracture of other specified part of pelvis |
| 80851 | Unspecified fracture of right ilium, initial encounter for open | Open fracture of ilium |
| 80851 | Unspecified fracture of left ilium, initial encounter for open | Open fracture of ilium |
| 80851 | Displaced avulsion fracture of right ilium, initial encounter | Open fracture of ilium |
| | 8083<br>8083<br>8083<br>8083<br>8083<br>80841<br>80842 | open fracture 8083 Fracture of superior rim of unspecified pubis, initial encounter for open fracture 8083 Other specified fracture of right pubis, initial encounter for open fracture 8083 Other specified fracture of left pubis, initial encounter for open fracture 8083 Other specified fracture of unspecified pubis, initial encounter for open fracture 80841 Unspecified fracture of right ilium, initial encounter for closed fracture 80841 Unspecified fracture of left ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of left ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of unspecified ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of unspecified ilium, initial encounter for closed fracture 80841 Other fracture of right ilium, initial encounter for closed fracture 80841 Other fracture of right ilium, initial encounter for closed fracture 80841 Other fracture of unspecified ilium, initial encounter for closed fracture 80842 Unspecified fracture of right ischium, initial encounter for closed fracture 80842 Unspecified fracture of right ischium, initial encounter for closed fracture 80842 Unspecified fracture of left ischium, initial encounter for closed fracture 80842 Displaced avulsion fracture of right ischium, initial encounter for closed fracture 80842 Displaced avulsion fracture of right ischium, initial encounter for closed fracture 80842 Other specified fracture of left ischium, initial encounter for closed fracture 80842 Nondisplaced avulsion fracture of unspecified ischium, initial encounter for closed fracture 80842 Other specified fracture of right ischium, initial encounter for closed fracture 80843 Unspecified fracture of |


# Appendix A Frailty markers


Falls


# Appendix A Frailty markers

## Combined Comorbidity Score for Claims Data

Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her Q. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


# Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

## Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

# Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| Anti epitepite non mood stabilizers | |
|-------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

## Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

## Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

# Selective serotonin reuptake inhibitor

| NDC Generic Name | |
|---------------------------|-----------------------------------------|
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

# Tricyclic antidepressants

| NDC Generic Name | |
|------------------------------------|--------------------------------|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL |
| AMOXAPINE | DOXEPIN HCL |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL |

# Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

# Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM, PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM,PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM, PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| Antiplatelet agents | |
|---|---|
| NDC Generic Name | |
| ABCIXIMAB | CILOSTAZOL |
| ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | VORAPAXAR SULFATE |
| NDC Brand Name | |
| ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

## Angiotensin II Receptor Blockers

| NDC Generic Name | |
|---|---|
| ALISKIREN/VALSARTAN | LOSARTAN POTASSIUM |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE/VALSARTAN | OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZID |
| AZILSARTAN MEDOXOMIL | OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE | TELMISARTAN |
| CANDESARTAN CILEXETIL | TELMISARTAN/AMLODIPINE BESYLATE |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE | TELMISARTAN/HYDROCHLOROTHIAZIDE |
| IRBESARTAN | VALSARTAN |

| IRBESARTAN/HYDROCHLOROTHIAZIDE | VALSARTAN/HYDROCHLOROTHIAZIDE |
|--------------------------------|--------------------------------|
| NDC Brand Name | · |
| AMLODIPINE-VALSARTAN | EXFORGE HCT |
| ATACAND | HYZAAR |
| ATACAND HCT | IRBESARTAN |
| AVALIDE | IRBESARTAN-HYDROCHLOROTHIAZIDE |
| AVAPRO | LOSARTAN POTASSIUM |
| AZOR | LOSARTAN-HYDROCHLOROTHIAZIDE |
| BENICAR | MICARDIS |
| BENICAR HCT | MICARDIS HCT |
| CANDESARTAN CILEXETIL | TELMISARTAN |
| CANDESARTAN-HYDROCHLOROTHIAZID | TELMISARTAN-AMLODIPINE |
| COZAAR | TELMISARTAN-HYDROCHLOROTHIAZID |
| DIOVAN | TRIBENZOR |
| DIOVAN HCT | TWYNSTA |
| EDARBI | VALSARTAN |
| EDARBYCLOR | VALSARTAN-HYDROCHLOROTHIAZIDE |
| EXFORGE | VALTURNA |

| Angiotensin Converting Enzyme inhibitors | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | LISINOPRIL |
| BENAZEPRIL HCL | LISINOPRIL/HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE | MOEXIPRIL HCL |
| CAPTOPRIL | MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | PERINDOPRIL ERBUMINE |
| ENALAPRIL MALEATE | QUINAPRIL HCL |
| ENALAPRIL MALEATE/FELODIPINE | QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE | RAMIPRIL |
| ENALAPRILAT DIHYDRATE | TRANDOLAPRIL |
| FOSINOPRIL SODIUM | TRANDOLAPRIL/VERAPAMIL HCL |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ACCUPRIL | LOTREL |
| ACCURETIC | LYTENSOPRIL |
| ACEON | LYTENSOPRIL-90 |
| ALTACE | MAVIK |
| AMLODIPINE BESYLATE-BENAZEPRIL | MOEXIPRIL HCL |
| BENAZEPRIL HCL | MOEXIPRIL-HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL-HCTZ | MONOPRIL |
| BENAZEPRIL-HYDROCHLOROTHIAZIDE | MONOPRIL HCT |
| CAPOTEN | PERINDOPRIL ERBUMINE |
| CAPOZIDE | PRINIVIL |
| CAPTOPRIL | PRINZIDE |
| CAPTOPRIL-HYDROCHLOROTHIAZIDE | QUINAPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | QUINAPRIL HCL |
| ENALAPRIL MALEATE | QUINAPRIL-HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE-HCTZ | QUINARETIC |
| ENALAPRIL MALEATE/HCTZ | RAMIPRIL |
| ENALAPRIL-HYDROCHLOROTHIAZIDE | TARKA |
| ENALAPRILAT | TRANDOLAPRIL |
| EPANED | TRANDOLA PRIL-VERA PAMIL |
| FOSINOPRIL SODIUM | UNIRETIC |
| FOSINOPRIL-HYDROCHLOROTHIAZIDE | UNIVASC |
| LEXXEL | VASERETIC |
| LISINOPRIL | VASOTEC |
| LISINOPRIL-HCTZ | VASOTEC I.V. |
| LISINOPRIL-HYDROCHLOROTHIAZIDE | ZESTORETIC |
| LOTENSIN | ZESTRIL |
| LOTENSIN HCT | |

#### Beta blockers

| Deta Blockers | |
|-------------------------|------------------------------------------|
| NDC Generic Name | |
| ACEBUTOLOL HCL | ESMOLOL HCL |
| ATENOLOL | LABETALOL HCL |
| ATENOLOL/CHLORTHALIDONE | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| BISOPROLOL FUMARATE | METOPROLOL TARTRATE |

| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE | METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
|---|---|
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE | NEBIVOLOL HCL |
| CARTEOLOL HCL | SOTALOL HCL |
| CARVEDILOL | TIMOLOL |
| CARVEDILOL PHOSPHATE | TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE | TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF | TIMOLOL MALEATE/PF |
| NDC Brand Name | |
| ACEBUTOLOL HCL | ISTALOL |
| ATENOLOL | KERLONE |
| ATENOLOL W/CHLORTHALIDONE | LABETALOL HCL |
| ATENOLOL-CHLORTHALIDONE | LOPRESSOR |
| BETAPACE | LOPRESSOR HCT |
| BETAPACE AF | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL TARTRATE |
| BETIMOL | METOPROLOL-HYDROCHLOROTHIAZIDE |
| BETOPTIC | NORMODYNE |
| BETOPTIC S | OCUPRESS |
| BISOPROLOL FUMARATE | SECTRAL |
| BISOPROLOL FUMARATE-HCTZ | SENORMIN |
| BISOPROLOL FUMARATE/HCTZ | SORINE |
| BISOPROLOL-HYDROCHLOROTHIAZIDE | SOTALOL |
| BLOCADREN | SOTALOL AF |
| BREVIBLOC | SOTALOL HCL |
| BYSTOLIC | TENORETIC 100 |
| CARTEOLOL HCL | TENORETIC 50 |
| CARTROL | TENORMIN |
| CARVEDILOL | TENORMIN CALENDAR PAK |
| COMBIGAN | TIMOLIDE |
| COREG | TIMOLOL MALEATE |
| COREG CR | TIMOPTIC |
| COSOPT | TIMOPTIC OCUDOSE |
| COSOPT PF | TIMOPTIC-XE |
| DORZOLAMIDE-TIMOLOL | TOPROL XL |
| DUTOPROL | TRANDATE |
| ESMOLOL HCL | ZEBETA |
| HYPERTENSOLOL | ZIAC |

# Calcium channel blockers

| Calcium channel blockers | |
|---|---|
| HCPCS | |
| C9248 | |
| NDC Generic Name | |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE | BEPRIDIL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE | CLEVIDIPINE BUTYRATE |
| AMLODIPINE BESYLATE | DILTIAZEM HCL |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | DILTIAZEM MALATE |
| AMLODIPINE BESYLATE/VALSARTAN | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |

| CARDIZEM CD | NYMALIZE |
|-------------------|------------------------|
| CARDIZEM LA | PLENDIL |
| CARDIZEM SR | POSICOR |
| CARTIA XT | PROCARDIA |
| CLEVIPREX | PROCARDIA XL |
| COVERA-HS | SULAR |
| DILACOR XR | TARKA |
| DILT-CD | TAZTIA XT |
| DILT-XR | TEKAMLO |
| DILTIA XT | TELMISARTAN-AMLODIPINE |
| DILTIAZEM 24HR CD | TIAMATE |
| DILTIAZEM 24HR ER | TIAZAC |
| DILTIAZEM ER | TRANDOLAPRIL-VERAPAMIL |
| DILTIAZEM HCL | TRIBENZOR |
| DILTIAZEM HCL-NS | TWYNSTA |
| DILTIAZEM XR | VASCOR |
| DILTIAZEM-D5W | VERAPAMIL ER |
| DILTZAC ER | VERAPAMIL ER PM |
| DYNACIRC | VERAPAMIL HCL |
| DYNACIRC CR | VERAPAMIL SR |
| EXFORGE | VERELAN |
| EXFORGE HCT | VERELAN PM |
| FELODIPINE ER | |

## Diuretics

| NDC Generic Name | |
|-----------------------------------|---------------------|
| AMILORIDE HCL | HYDROCHLOROTHIAZIDE |
| AMILORIDE HCL/HYDROCHLOROTHIAZIDE | HYDROFLUMETHIAZIDE |
| BENDROFLUMETHIAZIDE | INDAPAMIDE |
| BUMETANIDE | METHYCLOTHIAZIDE |
| CHLOROTHIAZIDE | METOLAZONE |
| CHLORTHALIDONE | POLYTHIAZIDE |
| EPLERENONE | SPIRONOLACTONE |
| ETHACRYNATE SODIUM | TORSEMIDE |
| ETHACRYNIC ACID | TRIAMTERENE |
| FUROSEMIDE | TRICHLORMETHIAZIDE |

# Nitrates

| Nitrates | |
|---|---|
| NDC Generic Name | |
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL | NITROGLYCERIN/DEXTROSE 5 % IN WATER |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |
| DILATRATE-SR | NITROCINE |
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 | NITROMIST |
| ISOREX-2.5 | NITRONAL |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |

| ISOTRATE ER | NITROSTAT IV |
|--------------------------|-----------------|
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| Lipid lowering drugs | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | METHYLTETRAHYDROFOLATE GLUCOSAMINE/NIACINAMIDE/CUPRIC &ZN OX |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA | NIACIN |
| ATORVASTATIN CALCIUM | NIACIN (INOSITOL NIACINATE) |
| BETA-CAROTENE(A) W-C & E/NIACINAMIDE/VIT B2/LUT/MIN/GLU-ONE | NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| CERAMIDES 1,3,6-11/NIACINAMIDE | NIACIN/LOVASTATIN |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID | NIACIN/SIMVASTATIN |
| CHOLESTYRAMINE | NIACINAMIDE |
| CHOLESTYRAMINE (WITH SUGAR) | NIACINAMIDE ASCORBATE |
| CHOLESTYRAMINE/ASPARTAME | NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| COLESEVELAM HCL | NIACINAMIDE/RIBOFLAVIN/BETA-CAROTENE(A) W-C & E/MINERALS |
| COLESTIPOL HCL | NIACINAMIDE/VIT B6/VIT C/FA/COPPER/MG CIT/ZN GLUC/ALIP ACID |
| EZETIMIBE | PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| EZETIMIBE/ATORVASTATIN CALCIUM | PITAVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN | POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| FENOFIBRATE | PRAVASTATIN SODIUM |
| FENOFIBRATE NANOCRYSTALLIZED | ROSUVASTATIN CALCIUM |
| FENOFIBRATE, MICRONIZED | SIMVASTATIN |
| FLUVASTATIN SODIUM | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| FOLIC ACID/NIACINAMIDE/ZINC | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| GEMFIBROZIL | THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| INOSITOL NIACINATE | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |

## Non-insulin diabetes medications

| Non-mount diabetes medications | |
|--------------------------------------|-------------------------------------|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL | PIOGLITAZONE HCL/METFORMIN HCL |
| CANAGLIFLOZIN/METFORMIN HCL | REPAGLINIDE |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |

| GLYBURIDE | SAXAGLIPTIN HCL |
|---|---|
| GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | TOLAZAMIDE |
| METFORMIN/CAFFEINE/AMINO ACIDS#7/HERBAL COMB#125/CHOLINE BIT | TOLBUTAMIDE |
| NDC Brand Name | |
| ACARBOSE | ICN-TOLAM |
| ACETOHEXAMIDE | INSULASE |
| ACTOPLUS MET | INVOKAMET |
| ACTOPLUS MET XR | JANUMET |
| ACTOS | JANUMET XR |
| AMARYL | JANUVIA |
| APPFORMIN | JENTADUETO |
| APPFORMIN-D | JUVISYNC |
| AVANDAMET | KAZANO |
| AVANDARYL | KOMBIGLYZE XR |
| AVANDIA | METAGLIP |
| CHLORABETIC 250 | METFORMIN HCL |
| CHLORPROPAMIDE | METFORMIN HCL ER |
| DIABETA | MICRONASE |
| DIABINESE | NATEGLINIDE |
| DIBATROL | NESINA |
| DUETACT | ONGLYZA |
| DYMELOR | ORIBETIC |
| FORTAMET | ORINASE |
| GLIMEPIRIDE | OSENI |
| GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCAMIDE | PRANDIN |
| GLUCOPHAGE | PRECOSE |
| GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOTROL | RIOMET |
| GLUCOTROL XL | RONASE |
| GLUCOVANCE | SK-TOLBUTAMIDE |
| GLUMETZA | STARLIX |
| GLYBURIDE | TOLAMIDE |
| GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| GLYCRON | TOLINASE |
| GLYNASE | TRADJENTA |
| GLYSET | |

# Insulin


| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
|-----------------------------|--------------------------------|
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| HUMALOG MIX 50/50 | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | |

#### Antidepressants

| HCPCS | |
|---|---|
| J1320 | |
| NDC Generic Name | |
| AMITRIPTYLINE HCL | IMIPRAMINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEV OMILNA CIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT, MISC. COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE | VORTIOXETINE HYDROBROMIDE |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |

| AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
|---|---|
| AMOXAPINE | MIRTAZAPINE ANHYDROUS |
| ANAFRANIL | NARDIL |
| APLENZIN | NEFAZODONE HCL |
| APPBUTAMONE | NORFRANIL |
| APPBUTAMONE-D | NORPRAMIN |
| ASENDIN | NORTRIPTYLINE HCL |
| AVENTYL HCL | OLANZAPINE-FLUOXETINE HCL |
| BRINTELLIX | OLEPTRO ER |
| BRISDELLE | PAMELOR |
| BUDEPRION SR | PAROXETINE HCL |
| BUDEPRION XL | PAXIL |
| BUPROBAN | PAXIL CR |
| BUPROPION HCL | PER-TRIP |
| BUPROPION HCL ER | PERPHENAZINE-AMITRIPTYLINE |
| BUPROPION HCL SR | PEXEVA |
| BUPROPION XL | PHENELZINE SULFATE |
| CELEXA | PRISTIQ ER |
| CHLORDIAZEPOXIDE-AMITRIPTYLINE | PROTRIPTYLINE HCL |
| CITALOPRAM | PROZAC |
| CITALOPRAM HBR | PROZAC WEEKLY |
| CLOMIPRAMINE HCL | PRUDOXIN |
| CYMBALTA | Q.E.L |
| DECONIL | RAPIFLUX |
| DESIPRAMINE HCL | RE-LIVE |
| DESVENLAFAXINE ER | REMERON |
| DESVENDATAXINE EIX DESVENDATAXINE FUMARATE ER | SARAFEM |
| DESYREL | SELFEMRA |
| DOXEPIN HCL | SENTROXATINE |
| DULOXETINE HCL | SERTRALINE HCL |
| E-VILL 10 | SERZONE |
| L VILL 10 | SEINZOINE |
| E-VIII 100 | SILENOR |
| E-VILL 100 | SILENOR<br>SINFOLIAN |
| E-VILL 25 | SINEQUAN |
| E-VILL 25<br>E-VILL 50 | SINEQUAN<br>SK-AMITRIPTYLINE |
| E-VILL 25 E-VILL 50 E-VILL 75 | SINEQUAN<br>SK-AMITRIPTYLINE<br>SK-PRAMINE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VIIBRYD |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VIBRYD VIVACTIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VELBUTRIN |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL WELLBUTRIN WELLBUTRIN |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5-4 TRIAVIL 2-5-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-6 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN SR WELLBUTRIN XL ZOLOFT |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5-4 TRIAVIL 2-5-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |

# Colchicine

| NDC Brand Name | |
|-----------------------|--------------------------|
| COLCRYS | |
| NDC Generic Name | |
| COLCHICINE | COLCHICINE/RHUS EXTRACTS |
| PROBENECID/COLCHICINE | |

# **NSAIDs and Coxibs**

| NDC Generic Name | |
|------------------|------------|
| CELECOXIB | NABUMETONE |
| DIFLUNISAL | NAPROXEN |
| ETODOLAC | OXAPROZIN |
| FLURBIPROFEN | PIROXICAM |
| IBUPROFEN | ROFECOXIB |
| INDOMETHACIN | SULINDAC |
| KETOPROFEN | VALDECOXIB |
| MELOXICAM | |

# Opioids

| NDC Brand Name LCOF DH LIQUIHISTINE CS ABC COMPOUND W/CODEINE #3 LORCET ABERTUSS HC LORCET 10-650 ASSTRAL LORCET 10-650 ACAHISTINE LORCET HD ACETA W/CODEINE ACETAMINOPH-CAFF-DIHYDROCODEIN LORCIDE ACETAMINOPHEN W-CODEINE LORTAB ASA ACETAMINOPHEN W-CODEINE LORTAB ASA ACETAMINOPHEN-CODEINE LORTUSS EX ACTAGEN-C LORTUSS HC ACTIFED WITH CODEINE LYNOX ACTIO M-CLEAR ADOL M-CLEAR IR AIRACOF ALA-HIST AC ALA-HIST AC ALA-HIST DHC ALA-HIST DHC ALLERFIM W/CODEINE ALLERFIM W-CODEINE AMBIED CD AMBARCOF GB AMAPHEN AMAPHEN AMAPHEN AMARCOP AMAPHEN AMARCOP AMBIED CD AMARCOP AMBIED CD AMARCOP AMBIED CD AMBIED CD AMARCOP AMBIED CD AMARCOP AMARCOP AMARCOP AMARCOP AMBIED CD AMARCOP AMARCOP AMARCOP AMARCOP AMARCOP AMBIED CD AMARCOP AMAR | Opioids | |
|---|---|---|
| ABC COMPOUND W/CODEINE #3 ABERTUSS HC ABERTUSS HC LORCET 10-650 ABSTRAL LORCET 10-650 ACAHISTINE LORCET HD ACETA W/CODEINE ACETAMINOPHE-CAFF-DIHYDROCODEIN ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN-CODEINE LORTUSS EX ACTAGEN-C LORTUSS HC ACTIGED WITH CODEINE LORTUSS HC ACTIGED WITH CODEINE ADOL M-CLEAR ADOL M-CLEAR ADOL M-CLEAR WC ALA-HIST AC ALA-HIST AC ALA-HIST DHC ALLEFT M-END MAX ALLEFT M-END MAX ALLEFT M-END MAX ALLEFT M-END MAX ALLEFT M-END MAX ALLEFT M-END WC ALLEFRIM W/CODEINE ALLEF CD ALLEF CD M-END W-ESSIC ALLEF CD M-END W-ESSIC ALLEF CD M-ESSIC ALLEF CD M-ARACOF BP AMACODONE MAR-COF BP AMACODONE MAR-COF CD MARGESIC AMBIEFD CD MARGESIC MARGES | NDC Brand Name | |
| ABER-TUSS HC ABSTRAL LORCET 10/650 ACAHISTINE LORCET HD ACETA W/CODEINE LORCET PLUS ACETAMINOPH-CAFF-DIHYDROCODEIN ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W/CODEINE LORTAB ASA ACETAMINOPHEN W/CODEINE LORTUSS EX ACTAGENC LORTUSS HC ACTIGED WITH CODEINE LYNOX ACTIQ M-CLEAR ADOL M-CLEAR IR ADOL M-CLEAR WC ALAHIST AC ALAHIST AC ALAHIST DHC M-END MAX ALCET M-END MAX ALCET M-END MAX ALLER IM-END PE ALLER IM-END WC ALLER IM-END W | A-COF DH | LIQUIHISTINE CS |
| ABSTRAL ACATAISTINE LORCET HD ACETA W/CODEINE LORCET PLUS ACETAMINOPH-CAFF-DIHYDROCODEIN ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W-CODEINE LORTAB ASA ACETAMINOPHEN W-CODEINE LORTAS ASA ACETAMINOPHEN-CODEINE LORTUSS EX ACTAGEN-C LORTUSS HC ACTIGE WITH CODEINE LYNOX ACTIQ M-CLEAR ADOL M-CLEAR IR AIRACOF M-CLEAR IR AIRACOF M-CLEAR IN M-END ALAHIST ACC M-END MAX ALCET M-END MAX ALCET M-END MAX ALLEFER MW/CODEINE M-END MC ALLEFEN CD M-END DE ALLEFEN CD M-END WC ALLEFEN CD M-END WC ALLEFEN CD M-END WC ALLEFEN CD M-END WC ALLEFEN CD M-M-CLEAR M-M-COF CB M-MAR-COF CB M-MAR-COF C | ABC COMPOUND W/CODEINE #3 | LORCET |
| ACAHISTINE ACETA W/CODEINE LORCET PLUS ACETAMINOPH-CAFF-DIHYDROCODEIN LORCIDE ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W/CODEINE LORTAB ASA ACETAMINOPHEN-CODEINE LORTUSS EX ACETAMINOPHEN-CODEINE LORTUSS EX ACTAGEN-C LORTUSS HC ACTIGED WITH CODEINE LYNOX ACTIQ ADOL M-CLEAR ACACIQ ADOL M-CLEAR IR ARACOF M-CLEAR WC ALA-HIST AC M-END ALA-HIST AC M-END ALA-HIST AC ALLAY M-END MAX ALCET M-END MAX ALLEF M-END MAX ALLEF M-END WC ALLEFRIM W/CODEINE M-END PE ALLERFRIM W/CODEINE M-END WC ALLEFN CD M-GESIC ALPHEN M-COF BP MAR-COF CG MARPHEN W/CODEINE NAR-COF CG MARPHEN W/CODEINE NAR-COF CG MARPHEN W/CODEINE NAR-COF CG MARPHEN W/CODEINE NAR-COF CG MARPED CD MAR-COF CG MARGESIC COMPOUND MAR-COF CG MARGESIC COMPOUND MARGESIC COMPOUND MARGESIC COMPOUND MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC IMPROVED MARHED-G CD MARGESIC IMPROVED MARHED-G CD MARHED-G CD MARHED-G CD MARHED-G CD MARHED-G CD MARLED-G CD MARLED-G CD MARLED-G CD MARLED-G CD MARLED-G CD MARLED-C CD MARLED- | ABER-TUSS HC | LORCET 10-650 |
| ACETA W/CODEINE ACETAMINOPH-CAFF-DIHYDROCODEIN LORCIDE ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W-CODEINE LORTAB ACETAMINOPHEN W-CODEINE LORTUSS EX ACTAGEN-C LORTUSS EX ACTAGEN-C LORTUSS HC ACTIGE WITH CODEINE LUNDOX ACTIQ ACTIQ ACTIQ ACTIQ ACTICA ACTICA ACODEINE ALA-HIST AC ALA-HIST BC ALLAY ALERT AC ALLAY ALLAY ALLAY ALLER BC ALLER BC ALLER BC ALLER BC ALLER BC ALLER BC ALLER BC ALLER CD AMAGNACET ALLER CD AMACODONE AMACODONE AMACODONE AMACODONE AMACODO C AMABISTISTION AMARCOF AMBISTISTION AMARCOF AMBISTO-G CD AMARESIC COMPOUND AMBISTO-G CD AMARIED CD AMARIED CD AMARIED CD AMARIED CD AMARIED CD AMARIED CD AMASITUSS HCC AMBOPHEN AMAI-TUSS HCC AMBOPHEN AMAI-TUSS HCC AMASIPED CD AM | ABSTRAL | LORCET 10/650 |
| ACETAMINOPH-CAFF-DIHYDROCODEINE ACETAMINOPHEN W-CODEINE ACETAMINOPHEN W-CODEINE LORTAB ASA ACETAMINOPHEN-CODEINE LORTUSS EX ACETAMINOPHEN-CODEINE LORTUSS EX ACTIAGEN-C LORTUSS HC ACTIGE WITH CODEINE LLYNOX ACTIQ M-CLEAR ADOL M-CLEAR IR ADOL M-CLEAR WC ALA-HIST AC ALA-HIST AC ALA-HIST OHC ALA-HIST OHC ALLER M-END MAX ALLET M-END MAX ALLET M-END MAX ALLET M-END WC ALLERRIM W/CODEINE M-END WC ALLERRIM W/CODEINE M-END WC ALLER COX M-TUSS ALOR M-MAGNACET ALPHEN MAR-COF BP MARACOF CG MARACOF BP MARACOF CG MARACOF BP MARACOF CG MARAGESIC AMBIEST JS JOO MARGESIC COMPOUND MARGESIC COMPOUND MARGESIC MARCOF MARGESIC COMPOUND MA | ACAHISTINE | LORCET HD |
| ACETAMINOPHEN W-CODEINE ACETAMINOPHEN W/CODEINE LIORTUSS ASA ACETAMINOPHEN CODEINE LIORTUSS EX ACTAGEN-C LIORTUSS HC ACTICED WITH CODEINE LLYNOX ACTIQ ACTICED WITH CODEINE LLYNOX ACTIQ M-CLEAR ADOL M-CLEAR JR ADOL AIRACOF M-CLEAR WC ALA-HIST AC ALA-HIST AC ALA-HIST DHC M-END MAX ALCET M-END MAX ALCET M-END MAX ALCET M-END MAX D ALLERFIM W/CODEINE M-END WC ALLERRIM W/CODEINE M-END WC ALLER NC ALIFEN CD M-GESIC ALIFEN CD M-GESIC ALIFEN CD M-GESIC ALIFEN M-COF BP AMACODONE MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 AMBINST AMBINST MARGESIC AMBIEC CD MARGESIC MARGESIC AMBIEC CD MARGESIC MARG | ACETA W/CODEINE | LORCET PLUS |
| ACETAMINOPHEN W-CODEINE ACETAMINOPHEN W/CODEINE LIORTUSS ASA ACETAMINOPHEN CODEINE LIORTUSS EX ACTAGEN-C LIORTUSS HC ACTICED WITH CODEINE LLYNOX ACTIQ ACTICED WITH CODEINE LLYNOX ACTIQ M-CLEAR ADOL M-CLEAR JR ADOL AIRACOF M-CLEAR WC ALA-HIST AC ALA-HIST AC ALA-HIST DHC M-END MAX ALCET M-END MAX ALCET M-END MAX ALCET M-END MAX D ALLERFIM W/CODEINE M-END WC ALLERRIM W/CODEINE M-END WC ALLER NC ALIFEN CD M-GESIC ALIFEN CD M-GESIC ALIFEN CD M-GESIC ALIFEN M-COF BP AMACODONE MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 AMBINST AMBINST MARGESIC AMBIEC CD MARGESIC MARGESIC AMBIEC CD MARGESIC MARG | ACETAMINOPH-CAFF-DIHYDROCODEIN | LORCIDE |
| ACETAMINOPHEN-CODEINE ACTAGEN-C LORTUSS HC ACTIGED WITH CODEINE LLYNOX ACTIQ M-CLEAR ADOL M-CLEAR IR AIRACOF ALA-HIST AC ALA-HIST AC ALLER IN ALLER IN M-END ALLER IN M-END MAX ALCET M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END WC ALLER IN ALLER IN ALLER IN ALLER IN M-END WC ALLER IN ALLER IN ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC M-END WC M | | |
| ACETAMINOPHEN-CODEINE ACTAGEN-C LORTUSS HC ACTIGED WITH CODEINE LLYNOX ACTIQ M-CLEAR ADOL M-CLEAR IR AIRACOF ALA-HIST AC ALA-HIST AC ALLER IN ALLER IN M-END ALLER IN M-END MAX ALCET M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END MAX ALLER IN M-END WC ALLER IN ALLER IN ALLER IN ALLER IN M-END WC ALLER IN ALLER IN ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC ALLER IN ALLER IN M-END WC M-END WC M | ACETAMINOPHEN W/CODEINE | LORTAB ASA |
| ACTAGEN-C ACTIFED WITH CODEINE LYNOX ACTIQ M-CLEAR ADOL M-CLEAR JR AIRACOF ALA-HIST AC ALA-HIST AC ALA-HIST DHC ALLERRIM W/CODEINE M-END MAX ALLERRIM W/CODEINE ALLERRIM W/CODEINE ALLER DX ALLER DX M-END MARCOF BP AMARCOF BP AMARCOF BP AMARGESIC AMBIFED CD MARGESIC MARGESIC MARCOF MARCOF MARCOF MARCOF MARCOF MARCOF MARGESIC | | LORTUSS EX |
| ACTIFED WITH CODEINE ACTIQ ACTIQ M-CLEAR M-CLEAR M M-CLEAR WC ALACHIST AC ALA-HIST AC ALAHIST DHC ALLET M-END MAX ALCET M-END MAX D ALLERFRIM W/CODEINE ALLEFRIM W/CODEINE ALLEFN CD ALLEFN CD ALLEFN CD ALLEFN CD M-END MAX M-END WC ALLEPN CDX M-TUSS ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBISTAS/100 MARGESIC MARGESIC MARGESIC MARGESIC MARGESIC MARCOF CG MARACOP BP AMACODONE MARCOF CG AMAPHEN W/CODEINE NO.3 MARGESIC AMBISTAS/100 MARGESIC MARGESI | ACTAGEN-C | |
| ADOL M-CLEAR JR AIRACOF M-CLEAR WC ALA-HIST AC M-END ALAHIST DHC M-END MAX ALCET M-END MAX ALLEY M-END PE ALLERRIM W/CODEINE M-END WC ALLER CD M-END WC ALLER CDX M-GESIC ALLPHEN MACODENE MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARGESIC AMBI S/15/100 MARGESIC AMBIFED CD MAXIFTUSS HC AMBIFED CD MAXI-TUSS HC AMBIFED CD MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCX AMACONA MAXIFED CD ANACIN-3 W/CODEINE ANACIN-3 W/CODEINE ANACIPAC MAXIFED CDX | | |
| ADOL M-CLEAR JR AIRACOF M-CLEAR WC ALA-HIST AC M-END ALAHIST DHC M-END MAX ALCET M-END MAX ALLEY M-END PE ALLERRIM W/CODEINE M-END WC ALLER CD M-END WC ALLER CDX M-GESIC ALLPHEN MACODENE MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARGESIC AMBI S/15/100 MARGESIC AMBIFED CD MAXIFTUSS HC AMBIFED CD MAXI-TUSS HC AMBIFED CD MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCX AMACONA MAXIFED CD ANACIN-3 W/CODEINE ANACIN-3 W/CODEINE ANACIPAC MAXIFED CDX | | |
| AIRACOF ALA-HIST AC ALAHIST DHC ALAHIST DHC ALAHIST DHC M-END MAX ALCET M-END MAX D ALLAY M-END PE ALLERFRIM W/CODEINE M-END WC ALLER CD ALLER CD ALLER CD ALLER CD ALLER CDX ALOR ALOR ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBIS/15/100 MARGESIC AMBIS/15/100 MARGESIC AMBIS-DIS-COMPOUND AMBIFED CD MARGESIC COMPOUND AMBIFED-G CD MARGESIC MAX HC AMBIFED-G CD MAX HC AMBIFED-G CD MAX HC AMBIFED-G CD MAX HC AMBIFED-G CD MAXI-TUSS HC AMBOPHEN MAXI-TUSS HC AMACON MAX | • | |
| ALA-HIST AC ALAHIST DHC ALAHIST DHC M-END MAX ALCET M-END MAX M-END MX ALLAY M-END MY ALLAY M-END WC ALLEFIND WC ALLEFEN CD M-GESIC ALLFEN CDX M-TUSS ALOR MARCOF AMPICO AMPICO AMARCOF AMACODONE AMACOF AMACOF AMARCOF AMARCOF AMBI 5/15/100 MARGESIC AMBI 5/15/100 MARGESIC AMBIFED CD MARGESIC AMBIFED CD MARGESIC AMBIFED-G CDX MARGESIC AMBIFED-G CDX MARGESIC AMBIFED-G CDX MARGESIC AMBIFED-G CDX MARGESIC AMBIFED-G CDX MARGESIC MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCX AMBOPHEN MAXI-TUSS HCX ANA-BATE MAXIONE ANACIN-3 W/CODEINE MAXIFED CD MAXIFED CD MAXIFED CD ANAIFED CD MAXIFED CD ANAIFED CD MAXIFED CD | | |
| ALAHIST DHC ALCET M-END MAX D ALLAY M-END PE ALLEFRIM W/CODEINE M-END WC ALLEFR CD M-GESIC ALLEFR CDX M-TUSS ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARGOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC AMBIFED CD MARGESIC AMBIFED CD MARGESIC COMPOUND AMBIFED CD MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC MAX HC AMBIFED-G CDX MANI-TUSS HC AMBOPHEN MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMSATE MAXIOONE MAXIFED CD | | |
| ALCET M-END MAX D ALLAY M-END PE ALLERFRIM W/CODEINE M-END WC ALLFEN CD M-GESIC ALLFEN CDX M-TUSS ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC AMBIFED CD MARGESIC COMPOUND AMBIFED CD MARGESIC IMPROVED AMBIFED CD MAX HC AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCS AMACONA MAXI-TUSS HCS AMACON | | |
| ALLAY ALLEFRIM W/CODEINE ALLEFRIM W/CODEINE ALLEFN CD ALLEFN CDX ALOR MAGNACET ALPHEN AMACODONE AMAR-COF EBP AMARCOF AMAPHEN W/CODEINE NO.3 AMBENYL AMBI 5/15/100 AMBIFED CD AMBIFED CD AMBIFED CDX AMBIFED CDX AMBIFED G CD AMBIFED G CD AMBIFED G CDX AMAXI-TUSS HC AMBOPHEN AMAXI-TUSS HCC AMAXI-TUSS H | | |
| ALLERFRIM W/CODEINE ALLER CD ALLER CDX ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE AMAPHEN W/CODEINE NO.3 AMBENYL AMBIS/15/100 AMBIS/15/100 MARGESIC AMBIFED CD AMBIFED CD AMBIFED CDX MARGESIC IMPROVED AMBIFED G CD AMBIFED G CD AMSHIFED G CDX AMSHIFED CDX AMSHIFED CDX AMSHIFED CDX AMSHIFED CDX AMSHIFED CDX AMSHIFED CDX ANACIN-3 W/CODEINE ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE MAXIFED CDX ANAXIFED CDX | | |
| ALLFEN CD M-GESIC ALLFEN CDX M-TUSS ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC AMBIFED CD MARGESIC COMPOUND AMBIFED CD MARGESIC H AMBIFED CDX MARGESIC IMPROVED AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCC AMBOPHEN MAXI-TUSS HCC AMBOPHEN MAXI-TUSS HCX AN-ABATE MAXIONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CD ANAIFED CDX | | |
| ALLFEN CDX M-TUSS ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC COMPOUND AMBIFED CD MARGESIC IMPROVED AMBIFED CDX MARGESIC IMPROVED AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| ALOR MAGNACET ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC COMPOUND AMBIFED CD MARGESIC H AMBIFED CDX MARGESIC IMPROVED AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXI-TUSS HCX AN-ABATE MAXI-TUSS HCX ANAIFED CD ANACIN-3 W/CODEINE MAXIFED CD ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED CDX ANAIFED-G CD | | |
| ALPHEN MAR-COF BP AMACODONE MAR-COF CG AMAPHEN W/CODEINE NO.3 MARCOF AMBENYL MARGESIC AMBI 5/15/100 MARGESIC COMPOUND AMBIFED CD MARGESIC IMPROVED AMBIFED CDX MARGESIC IMPROVED AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED-G CD | | |
| AMACODONE AMAPHEN W/CODEINE NO.3 AMBENYL AMBI 5/15/100 AMBIFED CD AMBIFED CD AMBIFED CDX AMBIFED-G CD AMBIFED-G CDX AMBIFED-G CDX AMBOPHEN AMSOPHEN AMSOPHEN AMSOPHEN AMSOPHEN ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE ANACIN-3 WITH CODEINE ANACIN-3 WASTED-G CD MARGESIC COMPOUND MARGESIC COMPOUND MARGESIC IMPROVED MARGESIC IMPROVED MARGESIC IMPROVED MAXI-TUSS HC MAXI-TUSS HC MAXI-TUSS HC MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXIFED CD MAXIFED CD MAXIFED CD MAXIFED CDX MAXIFED-G CD | | |
| AMAPHEN W/CODEINE NO.3 AMBENYL AMBENYL AMBI 5/15/100 AMBIFED CD AMBIFED CD AMBIFED CDX AMBIFED-G CD AMBIFED-G CD AMBIFED-G CDX AMBIFED-G CDX AMBIFED-G CDX AMSIFED-G CDX ANAI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX ANABATE ANAIDONE ANAIDONE ANAIN-3 W/CODEINE ANAIFED CD ANAIFED CDX ANAIFED-G CD | AMACODONE | |
| AMBENYL MARGESIC AMBI 5/15/100 MARGESIC COMPOUND AMBIFED CD MARGESIC H AMBIFED CDX MARGESIC IMPROVED AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| AMBIFED CD AMBIFED CDX AMBIFED-G CD AMBIFED-G CD AMBIFED-G CDX AMBIFED-G CDX AMBIFED-G CDX AMBIFED-G CDX AMSI-TUSS HC AMBOPHEN AMGENAL AN-ABATE ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE ANAPLEX HD MARGESIC IMPROVED MAXI-TUSS HCX MAXI-TUSS HC MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXIFED CD MAXIFED CD MAXIFED CDX MAXIFED CDX MAXIFED-G CD | | |
| AMBIFED CD AMBIFED CDX AMBIFED-G CD AMBIFED-G CD AMBIFED-G CDX AMBIFED-G CDX AMBIFED-G CDX AMBIFED-G CDX AMSI-TUSS HC AMBOPHEN AMGENAL AN-ABATE ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE ANAPLEX HD MARGESIC IMPROVED MAXI-TUSS HCX MAXI-TUSS HC MAXI-TUSS HCX MAXI-TUSS HCX MAXI-TUSS HCX MAXIFED CD MAXIFED CD MAXIFED CDX MAXIFED CDX MAXIFED-G CD | AMBI 5/15/100 | MARGESIC COMPOUND |
| AMBIFED CDX AMBIFED-G CD AMBIFED-G CDX AMBIFED-G CDX AMBOPHEN AMBOPHEN AMGENAL AN-ABATE ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE ANAPLEX HD MAXIFED-G CDX MAXIFED-G CD MAXIFED-G CD MAXIFED-G CD | | |
| AMBIFED-G CD MAX HC AMBIFED-G CDX MAXI-TUSS HC AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| AMBIFED-G CDX AMBOPHEN MAXI-TUSS HCG AMGENAL AN-ABATE ANACIN-3 W/CODEINE ANACIN-3 WITH CODEINE ANAPLEX HD MAXIFED-G CD MAXIFED-G CD | | |
| AMBOPHEN MAXI-TUSS HCG AMGENAL MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| AMGENAL MAXI-TUSS HCX AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| AN-ABATE MAXIDONE ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| ANACIN-3 W/CODEINE MAXIFED CD ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| ANACIN-3 WITH CODEINE MAXIFED CDX ANAPLEX HD MAXIFED-G CD | | |
| ANAPLEX HD MAXIFED-G CD | | |
| TANATUSS WALGUEINE TWAXIEED-G CDX | ANATUSS W/CODEINE | MAXIFED-G CDX |

| ANEXSIA | MAXIFLU CD |
|---|---|
| ANODYNOS-DHC | MAXIFLU CDX |
| ANOLOR DH-5 | MAXIPHEN CD |
| APOKYN | MAXIPHEN CDX |
| APOMORPHINE HCL | MAXITUSS HC |
| ASA-BUTALB-CAFFEINE-CODEINE | MC COUGH |
| ASCOMP W/CODEINE # 3 | MC JR COUGH |
| ASCOMP WITH CODEINE | MED-HIST |
| ASPIRIN W/CODEINE | MED-HIST-HC |
| ASPIRIN WITH CODEINE | MEDCODIN |
| ASPIRIN WITH CODEINE ASPIRIN-CAFFEINE-DIHYDROCODEIN | MEDICAP HD |
| ASTRAMORPH-PF | MEDICAF IID MEDIPAIN 5 |
| ATROPINE W/DEMEROL | MEDTUSS HD |
| ATUSS EX | MEGAGESIC |
| ATUSS G | MEGAMOR |
| ATUSS HC | MEPERGAN |
| ATUSS HD | MEPERGAN FORTIS |
| ATUSS HS | MEPERIDINE HCL |
| ATUSS HX<br>ATUSS MR | MEPERIDINE HCL-0.9% NACL MEPERIDINE HCL-NS |
| ATUSS MS | MEPERIDINE HCL-NS MEPERIDINE HCL/NS |
| ATUSS NX | MEPERIDINE W/PROMETHAZINE |
| AVINZA | MEPERIDINE W/PROMETHAZINE MEPERIDINE-PROMETHAZINE |
| AZDONE | |
| - | MEDROZINE |
| B-TUSS | MEPROZINE |
| BALACET 325 | MESEHIST WC |
| BALTUSSIN | MI-CODE |
| BALTUSSIN HC | MI-DECON |
| BANCAP HC | MINTEX HC |
| BAYCOMINE | MINTUSS EX |
| BAYCOMINE PEDIATRIC | MINTUSS G |
| BAYHISTINE | MINTUSS HC |
| BEXOPHENE | MINTUSS HD |
| BIOTUSSIN AC | MINTUSS MR |
| BIOTUSSIN DAC | MINTUSS MS |
| BIPHETANE-DC | MINTUSS NX |
| BITEX | MONTE-G HC |
| IDDM DELIC | NACHITETI I I I C |
| BPM PEHC | MONTEFLU HC |
| BROM-CORT-DC | MORPHINE SULF/D5W |
| BROM-CORT-DC<br>BROMANATE DC | MORPHINE SULF/D5W MORPHINE SULF/NS |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE | MORPHINE SULF/D5 W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMOTUSS W/CODEINE BROMPHEN-DC | MORPHINE SULF/D5W MORPHINE SULF/NS MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHEN-DC BROMPHENEX HD | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE DC | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMCOMP HC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMCOMP HC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-DC W/CODEINE BROMPHENIRAMINE-DC | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMCOMP HC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHEN-DC BROMPHENIRAMINE DC BROMPHENIRAMINE-DC | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE IN JECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE/D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR |
| BROM-CORT-DC BROMANATE DC BROMANATE-DC BROMANYL BROMAREST DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPLEX HD BRON-TUSS | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS MYBANIL |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-HYDROCOD-PSE BROMPLEX HD BRON-TUSS BRONKISAN A/C BRONTEX | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-BROCOD-PSE | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-BROWDE BROMPHENIRAMINE-BROWDE BROMPHENIRAMINE-BROWDE BROMPHENIRAMINE-BROWDE BROWDEX HD BRON-TUSS BRONKISAN A/C BRONTEX BROVEX CB | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 MYHYDROMINE |
| BROM-CORT-DC BROMANATE DC BROMANYL BROMAREST DC BROMATANE-DC BROMCOMP HC BROMODIPHENHYDRAMINE HCL BROMODIPHENHYDRAMINE W/CODEINE BROMOTUSS W/CODEINE BROMPHEN-DC BROMPHENEX HD BROMPHENIRAMINE DC BROMPHENIRAMINE-DC BROMPHENIRAMINE-BROCOD-PSE | MORPHINE SULF/D5W MORPHINE SULFATE MORPHINE SULFATE MORPHINE SULFATE CONCENTRATE MORPHINE SULFATE CR MORPHINE SULFATE ER MORPHINE SULFATE IN DEXTROSE MORPHINE SULFATE INJECTION MORPHINE SULFATE SELECT-A-JET MORPHINE SULFATE-0.9% NACL MORPHINE SULFATE-D5W MORPHINE SULFATE/D5W MORPHINE SULFATE/NS MS CONTIN MS/L MS/S MSIR MULTI-HIST CS MYBANIL MYCI-GC MYGRANOL W/CODEINE #3 |

| BROVEX PB CX | MYTUSSIN AC |
|---|---|
| BUTALB-ACETAMINOPH-CAFF-CODEIN | MYTUSSIN AC |
| BUTALB-CAFF-ACETAMINOPH-CODEIN | NALDECON-CX ADULT |
| BUTALBITAL COMPOUND W/CODEINE | NALEX |
| BUTALBITAL COMPOUND-CODEINE | NALEX AC |
| BUTALBITAL-CAFF-APAP-CODEINE | NALEX DH |
| BUTALBITAL/CAFF/APAP/CODEINE | NARCOF |
| BUTINAL W/CODEINE #3 | NARIZ HC |
| C-TUSSIN | NARVOX |
| CALCIDRINE | NASATUSS |
| CALCIUM IODIDE W/CODEINE | NASOTUSS |
| CANGES-HC | NAZARIN HC |
| CANGES-HC NR | NEO AC |
| CANGES-XP | NEO HC |
| CAPCOF | NORCET |
| CAPITAL W-CODEINE | NORCET 7.5MG |
| CAPITAL W/CODEINE | NORCO |
| CARISOPRODOL COMPOUND-CODEINE | NOTUSS |
| CARISOPRODOL-ASPIRIN-CODEINE | NOTUSS AC |
| CENTUSSIN DHC | NOTUSS DC |
| CETA-PLUS | NOTUSS PD |
| CGU WC | NOTUSS-FORTE |
| CHEMDAL | NOTUSS-PORTE<br>NOTUSS-NX |
| CHEMERGAN W/CODEINE | NOTUSS-NXD |
| CHERACOL | NOTUSS-PE |
| CHERATUSSIN AC | NOVADYNE |
| CHERATUSSIN AC CHERATUSSIN DAC | NOVADYNE DH |
| CHLORPHEN HD | NOVAGEST |
| CHLORPHENIRAMINE-CODEINE | NOVAGEST DH |
| CLEARTUSS DH | NOVAHISTINE |
| CO-GESIC | NOVAHISTINE DH |
| CO-HISTINE | NOVARISTINE DR |
| CO-HISTINE DH | NUCOCHEM |
| COASTALDYNE | NUCODINE SYR |
| COCET | NUCOFED |
| COCET PLUS | NUCOTUSS |
| CODACA NO.3 | NUDAL-HD |
| CODACA NO.4 | NUMORPHAN |
| CODAFED | OMS |
| CODAL-DH | ONCET |
| CODAMINE | ONCET 5 |
| CODAMINE PEDIATRIC | ONCET 7 |
| CODAPHEN | ONSOLIS |
| CODAR AR | OPANA |
| CODAR AR CODAR D | OPANA ER |
| | ORAMORPH SR |
| CODEEN CODEEN | |
| CODEFEN CODEGEST | ORGADIN-TUSS OXECTA |
| CODEINE COUGH SYRUP CODEINE PHOSPHATE | OXYCODONE CONCENTRATE OXYCODONE HCL |
| I CODEINE CHI EATE | |
| CODEINE CHAIFFNICH | OXYCODONE HCL ER |
| CODEINE-GUAIFENESIN | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH CODIMAL PH | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN OXYCODONE W/ASPIRIN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH CODIMAL PH CODITUSS DH | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN OXYCODONE W/ASPIRIN OXYCODONE W/ASPIRIN HALF-STR |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH CODIMAL PH CODITUSS DH CODOTUSS | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN OXYCODONE W/ASPIRIN OXYCODONE W/ASPIRIN HALF-STR OXYCODONE-ACETAMINOPHEN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH CODIMAL PH CODITUSS DH CODOTUSS COLDCOUGH | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN OXYCODONE W/ASPIRIN OXYCODONE W/ASPIRIN HALF-STR OXYCODONE-ACETAMINOPHEN OXYCODONE-ASPIRIN |
| CODEINE-GUAIFENESIN CODEINE/PHENYLPROP/GUAIFENESIN CODEMINE CODICLEAR DH CODIMAL DH CODIMAL PH CODITUSS DH CODOTUSS | OXYCODONE HCL ER OXYCODONE HCL-ACETAMINOPHEN OXYCODONE HCL-ASPIRIN OXYCODONE HCL-IBUPROFEN OXYCODONE HYDROCHLORIDE OXYCODONE W/ACETAMINOPHEN OXYCODONE W/ASPIRIN OXYCODONE W/ASPIRIN HALF-STR OXYCODONE-ACETAMINOPHEN |

| COLDCOLICITICM | OVVEACT |
|---|---|
| COLDCOUGH HCM | OXYFAST |
| COLDCOUGH PD | OXYIR OXYMADRIUONE LICE |
| COLDCOUGH XP | OXYMORPHONE HCL |
| COLDTUSS COLREX COMPOUND | OXYMORPHONE HCL ER |
| | P-EPD HCL/HCOD BT/CARBINOX |
| COMPLICED IIC | P-EPHED HCL/HYDROCOD BIT/CP |
| COMPASIN HC | P-TUSS |
| CONDASIN CONTRACTOR FINE | P-TUSS D |
| CONEX W/CODEINE | P-V-TUSSIN |
| CONZIP | PALLADONE |
| COPUENE VP | PANACET |
| COPHENE XP | PANADOL W/CODEINE NO.4 |
| COPHENE-S | PANADOL W/CODEINE NO.4 |
| COTAD A | PANASAL |
| COTAB A | PANCET |
| COTAB AX | PANCOF |
| COTABFLU | PANCOF EXP |
| COTUSS EX | PANCOF HC |
| COTUSS HD | PANCOF PD |
| COTUSS MS | PANCOF XP |
| COTUSS-V | PANLOR |
| COUGHTUSS | PANLOR DC |
| CPB WC | PANLOR SS |
| CRANTEX HC | PAPA-DEINE NO.4 |
| CYCOFED | PC-CAP |
| CYNDAL | PEDIACOF |
| CYTUSS HC | PEDIATEX HC |
| CYTUSS-HC | PEDITUSS |
| D-TANN HC | PERCOCET |
| DAMASON-P | PERCODAN |
| DARVOCET A500 | PERCODAN DEMI |
| DARVOCET-N 100 | PERCOLONE |
| DARVOCET-N 100<br>DARVOCET-N 50 | PERCOLONE<br>PERLOXX |
| DARVOCET-N 100 DARVOCET-N 50 DARVON | PERCOLONE PERLOXX PHANATUSS HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON | PERCOLONE PERLOXX PHANATUSS HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC |
| DARVOCET-N 100 DARVOCET-N 50 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS |
| DARVOCET-N 100 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE |
| DARVOCET-N 100 DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR DE-CHLOR MR DE-CHLOR NX | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DE-CHLOR NX DE-CHLOR NX | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENFLU CD PHENFLU CD |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/TODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENHIST |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECONAMINE CX | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DH DECONAMINE CX DECONGEST | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR DE-CHLOR MR DE-CHLOR MX DECOHISTINE DECOHISTINE DH DECONGEST DECTUSS C | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR DE-CHLOR MR DE-CHLOR MX DECOHISTINE DH DECONAMINE CX DECTUSS C DELHISTINE CS | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR MR DE-CHLOR MR DE-CHLOR MX DECOHISTINE DECOHISTINE DH DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DEMEROL DEPODUR | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CD PHENFLU CDX PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DEPODUR DESPEC-EXP | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-EXP DESPEC-PD | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE DH PHENYLPROPANOLAMINE PHENYLPROPANOLAMINE PHENYLPROPANOLAMINE PHENYLPROPANOLAMINE/HYDROCODON |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-PD DESPEC-PD DESPEC-PD DESPEC-PDC | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE DH PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR MX DECOHISTINE DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-EXP DESPEC-PD DESPEC-PDC DETUSS | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR MX DECOHISTINE DECOHISTINE DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-EXP DESPEC-PD DESPEC-PD DESPEC-PD DESPEC-PDC DETUSS DETUSS N | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-HCOD BT-CP PHENYLEPHRINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHURATUSS |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DH DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-PD DESPEC-PD DESPEC-PD DESPEC-PDC DETUSS DETUSS IN DEX-TUSS DEXPHEN W-C | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-HCOD BT-CP PHENYLEPHSTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DH DECONAMINE CX DECNGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-EXP DESPEC-PD DESPEC-PD DESPEC-PD DETUSS DETUSSIN DEX-TUSS DEXPHEN W-C DIABETIC TUSSIN C | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN VC WITH CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-RINE HD PHENYLHISTINE PHENYLHISTINE DH PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE/HYDROCODON PHRENILIN W/CAFFEINE & CODEINE PLURATUSS PNAP PNEUMOTUSSIN PNEUMOTUSSIN |
| DARVOCET-N 100 DARVON DARVON DARVON COMPOUND DARVON COMPOUND 32 DARVON COMPOUND-65 DARVON-N DAZIDOX DE-CHLOR G DE-CHLOR HC DE-CHLOR HD DE-CHLOR MR DE-CHLOR NX DECOHISTINE DECOHISTINE DH DECONAMINE CX DECONGEST DECTUSS C DELHISTINE CS DEMEROL DESPEC-PD DESPEC-PD DESPEC-PD DESPEC-PDC DETUSS DETUSS IN DEX-TUSS DEXPHEN W-C | PERCOLONE PERLOXX PHANATUSS HC PHEN/CHLOR HC PHENA-HC PHENAPHEN W/CODEINE PHENDACOF HC PHENDACOF PLUS PHENERGAN VC W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN W/CODEINE PHENERGAN WITH CODEINE PHENERGAN WITH CODEINE PHENFLU CD PHENFLU CD PHENFLU CDX PHENHIST PHENYLCODONE PEDIATRIC PHENYLEPH-HCOD BT-CP PHENYLEPH-HCOD BT-CP PHENYLEPHINE HD PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLHISTINE PHENYLPROP/COD/BR-PHENIRAMINE PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE DC PHENYLPROPANOLAMINE & CODEINE PHRENILIN W/CAFFEINE & CODEINE PHRENILIN-CAFFEINE-CODEINE PLURATUSS PNAP PNEUMOTUSSIN |

| | I |
|---|---|
| DIHISTINE DH | POLY HIST HC |
| DIHYDRO-CP | POLY HIST NC |
| DIHYDRO-GP | POLY-CS |
| DIHYDRO-PE | POLY-HISTINE |
| DIHYDROCODEINE COMP MOD | POLY-HISTINE CS |
| DIHYDROCODEINE COMPOUND | POLY-TUSSIN |
| DIHYDROCODEINE-BPM-PE | POLY-TUSSIN AC |
| DIHYDROXCODEINE COMPOUND | POLY-TUSSIN D |
| DILAUDID | POLY-TUSSIN DHC |
| DILAUDID STRIP PACKS | POLY-TUSSIN EX |
| DILAUDID-5 | POLY-TUSSIN HD |
| DILAUDID-HP | POLY-TUSSIN XP |
| DIMETANE-DC | POLYGESIC |
| DOLACET | POLYTINE CS |
| DOLAGESIC | POT GUAIACO-HYDROCODONE BIT |
| DOLENE | PP-CAP |
| DOLENE AP-65 | PRIMALEV |
| DOLENE COMPOUND-65 | PRIMLEV |
| DOLFEN | PRO POX 65 |
| DOLO PAP | PRO-CLEAR |
| DOLO-PAP | PRO-CLEAR AC |
| DOLOREX FORTE | PRO-CLEAR CAPS |
| DOLPHEN | PRO-COF |
| DONATUSS DC | PRO-COF D |
| DONATUSSIN DC | PRO-RED |
| DONATUSSIN MAX | PRO-RED AC |
| DORAPHEN-65 | PROCET |
| DOXAPAP N-100 | PROLEX DH |
| DRITUSS HD | PROMETHAZINE VC W/CODEINE |
| DROCON-CS | PROMETHAZINE VC-CODEINE PROMETHAZINE VC-CODEINE |
| DROTUSS | PROMETHAZINE WCODEINE PROMETHAZINE WCODEINE |
| DROTUSS-CP | PROMETHAZINE W/CODEINE PROMETHAZINE-CODEINE |
| DUOCET | PROPACET PROPACET |
| DOUCEI | PROPACEI |
| DUQUIST DU | IDDODACHEM |
| DUOHIST DH | PROPACHEM PEDIATRIC |
| DURADAL | PROPACHEM PEDIATRIC |
| DURADAL<br>DURADAL HD | PROPACHEM PEDIATRIC PROPAIN HC |
| DURADAL DURADAL HD DURADAL HD PLUS | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE W/APAP PROPOXYPHENE NAPSYLATE-APAP |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNEX HD | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-SYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNATUSS HC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-SYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNEX HD | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-SYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNATUSS HC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-SYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTESS PROTUSS-D PROVAL NO.3 |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNATUSS HCG DYNATUSS HC DYNATUSS HC DYNATUSS HCG DYNATUSS HC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTUSS- PROTUSS-D |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS DF DYNATUSS HC DYNATUSS HCG DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC ED-TLC | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTESS PROTUSS-D PROVAL NO.3 |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HCG DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC EFASIN | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE W/APAP PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC ED-TLC EFASIN EFASIN-HD | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE W/APAP PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTUSS PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE W/APAP PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.3 | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/CODEINE |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HCG DYNEX HD DYTAN-HC E-LOR ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.4 | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HC ED TUSS HC ED TUSS HC ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.3 EMCODEINE NO.3 EMCODEINE NO.3 | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HC ED TUSS HC ED TUSS HC ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.4 EMPIRIN W/CODEINE | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HC ED TUSS HC ED TUSS HC ED TUSS HC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.3 EMPRACET W/CODEINE NO.4 EMPRACET W/CODEINE NO.4 | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HC EDYNATUSS HC EDTUSS HC ED TUSS HC ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.4 EMPIRIN W/CODEINE EMPRACET W/CODEINE NO.4 ENDACOF ENDACOF | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE W/APAP PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTEX PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL |
| DURADAL DURADAL HD DURADAL HD PLUS DURADYNE DHC DURAGANIDIN NR DURAGESIC DURAMORPH DURATUSS HD DYNATUSS HC DYNATUSS HC DYNATUSS HC EDYNATUSS HC ELOR ED TUSS HC ED-TLC EFASIN EFASIN-HD EMBEDA EMCODEINE NO.4 EMPRACET W/CODEINE NO.4 ENDACOF | PROPACHEM PEDIATRIC PROPAIN HC PROPOXACET-N 100 PROPOXYPHENE HCL PROPOXYPHENE HCL COMPOUND PROPOXYPHENE HCL W/APAP PROPOXYPHENE HCL-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAP-ACETAMINOPHEN PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE PROPOXYPHENE NAPSYLATE-APAP PROTEX PROTEX PROTEX PROTUSS PROTUSS PROTUSS-D PROVAL NO.3 PSE BPM HD PSEUDATEX HC PSEUDOEPHEDRINE W/CODEINE PSEUDOEPHEDRINE W/HYDROCODONE PSEUDOEPHEDRINE-CODEINE Q-V TUSSIN QUAL-TUSSIN DC QUALA-HC QUINDAL |

| END ACCE DI | DEL ACON LICAID |
|----------------------------|------------------------------|
| ENDACOF-UC | RELACON-HC NR |
| ENDACOF-PLUS | RELASIN HC RELASIN-HCX |
| ENDACOF-PLOS ENDACOF-XP | RELATUSS HC |
| ENDAGEN-HD | RELCOF C |
| ENDAL | REPREXAIN |
| ENDAL CD | RESCUDOSE |
| ENDAL HD | REX-A-HIST |
| ENDAL-HD | REZIRA |
| ENDAL-HD PLUS | RHINACON DH |
| ENDOCET ENDOCET | RID-A-PAIN W/CODEINE |
| ENDOCODONE | RINDAL HD |
| ENDODAN | RINDAL HD PLUS |
| ENDOTUSS | RINDAL HID FEOS |
| ENPLUS-HD | RMS-SUPPOSITORY |
| ENTEX HC | RO-CET-N 100 |
| ENTUSS | ROBAFEN AC |
| ENTUSS-D | ROBAFEN-DAC |
| ESGIC W/CODEINE | ROBICHEM AC |
| ETH-OXYDOSE | ROBITUSSIN A-C |
| EXALGO | ROBITUSSIN-DAC |
| EXCOF | ROGESIC #3 |
| EXCOF-SF | ROMILAR AC |
| EXECLEAR | ROXANOL |
| EXECLEAR-C | ROXANOL SR |
| EXECOF-XP | ROXANOL UD |
| EXETUSS-HC | ROXANOL-T |
| EXTENDRYL HC | ROXICET |
| FARBITAL W/CODEINE #3 | ROXICODONE |
| FEBRIDYNE | ROXICODONE INTENSOL |
| FENTANYL | ROXIPRIN |
| FENTANYL BASE | RYBIX ODT |
| FENTANYL CITRATE | RYDEX |
| FENTANYL CITRATE-0.9% NACL | RYNA-C |
| FENTANYL CITRATE-D5W | RYNA-CX |
| FENTANYL CITRATE-NS | RYZOLT |
| FENTANYL CITRATE/NS | S-T FORTE 2 |
| FENTANYL ORALET | SENEFEN III |
| FENTANYL W/DROPERIDOL | SIMUC-HD |
| FENTANYL WITH DROPERIDOL | SINODEINE |
| FENTANYL-BUPIVACAINE-NS | SK-65 |
| FENTANYL-ROPIVACAINE-NS | SK-65 APAP |
| FENTANYL/NS | SK-65 COMPOUND |
| FENTORA | SK-APAP W/CODEINE |
| FENTUSS | SK-OXYCODONE W/ACETAMINOPHEN |
| FIORICET W/CODEINE | SK-OXYCODONE W/ASPIRIN |
| FIORICET WITH CODEINE | SOMA COMPOUND W/CODEINE |
| FIORINAL W/CODEINE #3 | SOMA COMPOUND WITH CODEINE |
| FIORINAL WITH CODEINE #3 | SPEN-HISTINE |
| FIORMOR W/CODEINE #3 | STAGESIC |
| FIORTAL W/CODEINE #3 | STAGESIC-10 |
| FLUTUSS HC | STATUSS |
| FLUTUSS XP | STATUSS GREEN |
| G-TUSS | STERAPHEN W/CODEINE |
| GANI-TUSS NR | STOPAYNE |
| GECIL | SU-TUSS HD |
| GENAGESIC | SUBLIMAZE |
| GENECOF-HC | SUBSYS |
| GENECOF-XP | SUDATUSS-2 |
| GENTEX HC | SUDATUSS-SF |
| GESIC-5<br>GESIC-HD | SUTTAR-2 |
| | SUTTAR-SF |

| OFFITHER HE | CVAATAN |
|---|---|
| GESTUSS-HC | SYMTAN CONSTANT A |
| GILTUSS HC | SYMTAN A |
| GILTUSS PED-C | SYNALGOS-DC |
| GLYDEINE | SYNGESIC DC |
| GUA C<br>GUA PC | SYNGESIC-DC<br>T-GESIC |
| GUAIATUSSIN AC | T-GESIC FORTE |
| GUAIFEN-C | THERACODOPHEN 650 |
| GUAIFENESIN A.C. GUAIFENESIN AC | THERACODOPHEN-650 THERACODOPHEN-LOW-90 |
| GUAIFENESIN DAC<br>GUAIFENESIN NR | THERATRAMADOL-60 THERATRAMADOL-90 |
| | TL-HIST CD |
| GUAIFENESIN W-CODEINE GUAIFENESIN W/CODEINE | TL-HIST CM |
| GUAIFENESIN W/CODEINE GUAIFENESIN-CODEINE | |
| GUAIFENESIN-CODEINE GUAIFENESIN-P-EPHEDRINE-COD | TOURO HC TRAMADOL HCL |
| GUAIFENESIN-P-EPHEDRINE-COD GUAIFENESIN-PHENYLEPHRINE-HCOD | TRAMADOL HCL TRAMADOL HCL ER |
| GUAIFENESIN/CODEINE PHOSPHATE | TRAMADOL HCL-ACETAMINOPHEN |
| GUAIFENESIN/CODEINE PHOSPHATE GUAIFENESIN/P-EPHED HCL/HCOD | TREZIX |
| GUAIFENESIN/P-EPHED HCL/HCOD GUAIFENESIN/P-EPHEDRINE/COD | TRI-VENT HC |
| GUAITENESIN/P-EPHEDRINE/COD GUAITUSSIN AC | TRIACIN C |
| GUAITUSSIN AC<br>GUAITUSSIN DAC | TRIACIN C |
| GUAL-CO | TRIAFED WITH CODEINE |
| GUAPETEX HC | TRIAMINIC DH |
| GUIADEX DH | TRIAMINIC DH TRIAMINIC W/CODEINE |
| | · |
| GUIAOLEX HC | TRIANT-HC |
| GUIATUSS AC<br>GUIATUSS DAC | TRICODE AR TRICODE GF |
| GUIATUSSIN DAC | TRICODE GF TRICODENE W/CODEINE |
| GUIATUSSIN DAC<br>GUIATUSSIN W/CODEINE | TRICOPENE W/CODEINE |
| H-C TUSSIVE | TRICOF EXP |
| 1 1 - 1 1 1 1 1 N N | |
| H-C TUSSIVE-D | TRICOF PD |
| H-C TUSSIVE-D<br>HALOTUSSIN AC | TRICOF PD TRIDAL |
| H-C TUSSIVE-D<br>HALOTUSSIN AC<br>HALOTUSSIN-AC | TRICOF PD TRIDAL TRIDAL HD |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX PV HISTUSS HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTUSSINE HC HISTUSSINE HC HISTUSSINE HC HISTUSSINE HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN HC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL C TUSNEL-HC TUSS-AX TUSS-DS |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSS HC HISTUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX HC HISTINEX HC HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP HY-PHEN | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-PD |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX HC HISTINEX HC HISTIUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP HY-PHEN HYCET | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-PD TUSS-S |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-6XP HY-PHEN HYCET HYCO-PAP | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-PD TUSS-S TUSS-PD TUSS-S TUSS-BUSS-BUSS-BUSS-BUSS-BUSS-BUSS-BUSS- |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSS HC HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-6XP HY-PHEN HYCET HYCO-PAP HYCODAN | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIFIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-PD TUSS-S TUSS-B TUSSADUR-HD TUSSAFED-HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTINEX HC HISTINEX HC HISTINEX HC HISTIUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP HY-PHEN HYCET HYCO-PAP HYCODAN HYCODAPHEN | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-PD TUSS-S TUSSADUR-HD TUSSAFED-HC TUSSAFED-HC TUSSAFED-HC TUSSAFED-HC TUSSAFED-HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN D HY-5 HY-KXP HY-PHEN HYCET HYCO-PAP HYCODAN HYCODAPHEN HYCOFED | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-PD TUSS-S TUSS-PD TUSS-S TUSSADUR-HD TUSSAFED-HC TUSSAFED-HCG TUSSAR-2 |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP HY-PHEN HYCOFED HYCOGESIC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-HC TUSS-PD TUSS-S TUSSAPED-HC TUSSAFED-HC TUSSAR-2 TUSSAFED-HCG TUSSAR-2 TUSSAR-2 TUSSAR-2 TUSSCOUGH DHC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-FAXP HY-PHEN HYCET HYCODAN HYCODAPHEN HYCOFED HYCOGESIC HYCOMAL DH | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-HC TUSS-PD TUSS-S TUSSADUR-HD TUSSAFED-HC TUSSAR-2 TUSSCOUGH DHC TUSSCOUGH HC |
| H-C TUSSIVE-D HALOTUSSIN AC HALOTUSSIN-AC HALOTUSSIN-DAC HBA HC TUSSIVE-D HC-GUAI HC-PE-DBROM HIST-HC HIST-PLUS HISTAFED-C HISTEX HC HISTINEX HC HISTINEX PV HISTUSSIN D HISTUSSIN D HISTUSSIN D HISTUSSIN HC HPB MAX HPR END HY-5 HY-KXP HY-PHEN HYCOFED HYCOGESIC | TRICOF PD TRIDAL TRIDAL HD TRIDAL HD PLUS TRIFED-C TRIHIST-CS TRIPOSED W/CODEINE TRIPROLIDINE-C TRIPROLIDINE/P-EPHED/CODEINE TRITUSSIN TRYCET TRYMINE CG TUSANA-D TUSDEC-HC TUSNEL C TUSNEL PED-C TUSNEL-HC TUSS-AX TUSS-DS TUSS-ES TUSS-HC TUSS-PD TUSS-S TUSSAPED-HC TUSSAFED-HC TUSSAR-2 TUSSAFED-HCG TUSSAR-2 TUSSAR-2 TUSSAR-2 TUSSCOUGH DHC |

| LIVCOMINE COMPOUND | THIS CONCANIDINALD |
|---|---|
| HYCOMINE COMPOUND | TUSSI-ORGANIDIN NR |
| HYCOPHEN | TUSSI-ORGANIDIN-S NR |
| HYCOSIN | TUSSICAPS |
| HYCOTAB | TUSSICLEAR DH |
| HYCOTUSS | TUSSIDEN C |
| HYDEX PD | TUSSIDIN NR |
| HYDONE | TUSSIGON |
| HYDRO GP | TUSSIN AC |
| HYDRO PC II | TUSSINAL 12 |
| HYDRO PRO | TUSSINATE |
| HYDRO PRO D | TUSSIONEX |
| HYDRO-DP | TUSSIREX |
| HYDRO-PC | TUSSIVE HC |
| HYDRO-PC II PLUS | TUSSO-C |
| HYDRO-PROPANOLAMINE PEDIATRIC | TUSSO-DF |
| HYDRO-TUSS | TUSSO-HC |
| HYDRO-TUSSIN DHC | TUSSPLEX |
| HYDRO-TUSSIN EXP | TY-PAP W/CODEINE |
| HYDRO-TUSSIN HC | TY-TAB W/CODEINE |
| HYDRO-TUSSIN HD | TYLAGESIC 3 |
| HYDRO-TUSSIN HG | TYLENOL W/CODEINE |
| HYDRO-TUSSIN XP | TYLENOL W/CODEINE NO.2 |
| HYDROCET | TYLENOL W/CODEINE NO.3 |
| HYDROCOD BIT-PHENYLEPHRINE-CP | TYLENOL W/CODEINE NO.4 |
| HYDROCOD-CPM-PSEUDOEPHEDRINE | TYLENOL-CODEINE NO.3 |
| HYDROCOD/CARBINOX/PSEUDOEPHED | TYLENOL-CODEINE NO.4 |
| HYDROCODONE | TYLOX |
| HYDROCODONE BIT-HOMATROPINE MB | UGESIC |
| HYDROCODONE BIT-IBUPROFEN | ULTRACET |
| HYDROCODONE BITARTRATE | ULTRAGESIC |
| LIVEROCODONE DE LIONANTRODINE NADR | LUTDANA |
| HYDROCODONE BT-HOMATROPINE MBR | ULTRAM |
| HYDROCODONE BI-HOMATROPINE MBR HYDROCODONE COMPOUND | ULTRAM ER |
| HYDROCODONE COMPOUND | ULTRAM ER |
| HYDROCODONE COMPOUND<br>HYDROCODONE CP | ULTRAM ER<br>UMI-APAP |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF | ULTRAM ER UMI-APAP UNI MULTIHIST CS |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV |
| HYDROCODONE COMPOUND HYDROCODONE GP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-EV UNI-TRICOF HC |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOR |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE WACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE WACETAMINOPHEN HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-IBUPROFEN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VAZOTUSS HC |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-IBUPROFEN HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-IBUPROFEN HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/HOMATROPINE HYDROCODONE/HOMATROPINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PENYLEPH/PYRILAM | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-EV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE ACETAMINOPHEN HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN HYDROCODONE/HOMATROPINE HYDROCODONE/HOMATROPINE HYDROCODONE/HOMATROPINE HYDROCODONE/HOMATROPINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-EV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN HYDROCODONE/HOMATROPINE HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPOPANOLAMIN | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN VICODIN ES |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE HD HYDROCODONE WACETAMINOPHEN HYDROCODONE WACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROFED HYDROGESIC | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PHENYLPROPEN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMET | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLPROPANOLAMIN HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMET HYDROMINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOR VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN VIHISTINE |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMINE HYDROMINE HYDROMINE HYDROMINE | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOR VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN VIHISTINE VIRTUSSIN AC |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE MBR HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMET HYDROMINE HYDROMORPHONE ER | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN VIHISTINE VIRTUSSIN AC VISVEX HC |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE PA HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/PHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-BUPROFEN HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCODONE/PHENYLEPH/PYRILAM HYDROCOF-HC HYDROFED HYDROGESIC HYDROMET HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOR VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN TUSS VICOPROFEN VIHISTINE VIRTUSSIN AC VISVEX HC VITAPAP W/CODEINE |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMET HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN VIHISTINE VISVEX HC VITAPAP W/CODEINE VITUSSIN |
| HYDROCODONE COMPOUND HYDROCODONE GF HYDROCODONE HD HYDROCODONE WACETAMINOPHEN HYDROCODONE-ACETAMINOPHEN HYDROCODONE-ACETAMINOPHEN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-HOMATROPINE MBR HYDROCODONE-BUPROFEN HYDROCODONE/ACETAMINOPHEN HYDROCODONE/ACETAMINOPHEN HYDROCODONE/ACETAMINOPHEN HYDROCODONE/PHENYLEPH/PYRILAM HYDROMORPHONE HCL INJECTION HYDROMORPHONE HCL-D5W | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI-COF UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN TUSS VICOPROFEN VIHISTINE VISVEX HC VITAPAP W/CODEINE VITUSSIN VITUZ |
| HYDROCODONE COMPOUND HYDROCODONE CP HYDROCODONE GF HYDROCODONE HD HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W-ACETAMINOPHEN HYDROCODONE W/GUAIFENESIN HYDROCODONE W/FHENYLPROP HYDROCODONE-ACETAMINOPHEN HYDROCODONE-GUAIFENESIN HYDROCODONE-HOMATROPINE HYDROCODONE-HOMATROPINE MBR HYDROCODONE-BUPROFEN HYDROCODONE-POT GUAIACOSULFON HYDROCODONE/ACETAMINOPHEN HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPPH/PYRILAM HYDROCODONE/PHENYLPROPANOLAMIN HYDROCOF-HC HYDROGESIC HYDROMET HYDROMINE HYDROMORPHONE ER HYDROMORPHONE HCL | ULTRAM ER UMI-APAP UNI MULTIHIST CS UNI TUSS HC UNI-COF UNI-COF EXP UNI-LEV UNI-TRICOF HC VANACET VANACOF CD VANACON VANEX GRAPE VANEX HD VAZOTUSS HC VENDONE VERDROCET VI-Q-TUSS VICOCLEAR DH VICODIN HP VICODIN TUSS VICOPROFEN VIHISTINE VIRTUSSIN VISVEX HC VITAPAP W/CODEINE VITUSSIN |

| LIVEROMORPHONE HVEROCHLORIDE | WELL THECHO |
|---|---|
| HYDROMORPHONE HYDROCHLORIDE | WELL-TUSS HD |
| HYDROMORPHONE-BUPIVACAINE HYDROMORPHONE-BUPIVACAINE-NS | WELLTUSS EXP WELLTUSS HC |
| HYDROMORPHONE/BUPIVACAINE | WYGESIC |
| HYDRON CP | XARTEMIS XR |
| HYDRON EX | XODOL 10-300 |
| HYDRON KGS | XODOL 10/300<br>XODOL 10/300 |
| | XODOL 10/300<br>XODOL 5-300 |
| HYDRON PSC | XODOL 5-300<br>XODOL 7.5-300 |
| HYDROPHEN | XOLOX |
| HYDROPHEN PEDIATRIC | XPECT-HC |
| HYDROPHENE DH | |
| | XYLON 10 Z-COF HC |
| HYDROSTAT<br>HYPHED | Z-COF HCX |
| HYPHEN-HD | Z-TUSS 2 |
| HYTAN | Z-TUSS AC |
| IBUDONE | Z-TUSS E |
| IDENAL W/CODEINE | ZAMICET |
| INFUMORPH | ZERLOR<br>ZHIST |
| INNOVAR<br>IODAL HD | ZODRYL AC 25 |
| IOFEN-C NF | ZODRYL AC 25 ZODRYL AC 30 |
| IOPHEN | |
| IOPHEN C-NR | ZODRYL AC 35<br>ZODRYL AC 40 |
| IOPHEN-C NR IOTUSSIN D | ZODRYL AC 50<br>ZODRYL AC 60 |
| IOTUSSIN HC | |
| | ZODRYL AC 80 |
| ISOBUTAL W/CODEINE ISOLIN W/CODEINE | ZODRYL DAC 25<br>ZODRYL DAC 30 |
| ISOLLYL W/CODEINE | |
| J-CET | ZODRYL DAG 40 |
| J-COF DHC | ZODRYL DAC 50 |
| J-MAX DHC | ZODRYL DAC 50<br>ZODRYL DAC 60 |
| J-TAN D HC | ZODRYL DAC 80 |
| JAYCOF | ZODRYL DAC 80 ZODRYL DEC 25 |
| JAYCOF-HC | ZODRYL DEC 25 ZODRYL DEC 30 |
| JAYCOF-NC<br>JAYCOF-XP | ZODRYL DEC 35 |
| KADIAN | ZODRYL DEC 35 ZODRYL DEC 40 |
| KG-DAL HD | ZODRYL DEC 40 ZODRYL DEC 50 |
| KG-DAL HD PLUS | ZODRYL DEC 30 ZODRYL DEC 60 |
| KG-FED | ZODRYL DEC 80 |
| KG-FED PEDIATRIC | ZOHYDRO ER |
| KG-TUSS HD<br>KG-TUSSIN | ZOLVIT<br>ZOTEX-C |
| KGS-HC | ZOTEX-C |
| KWELCOF | ZTUSS |
| LAZANDA | ZTUSS ZT |
| LEVALL | ZUTRIPRO |
| | ZYDONE |
| LEVALL 5.0 | |
| LEXUSS 210 | ZYMINE HC |
| LIQUICET LIQUICOUGH HC | ZYRPHEN-HC |
| NDC Generic Name | |
| | WEDEBIDINE HOLIN O.9 & SODILIM CHI OBIDE |
| BROMPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MEPERIDINE HCL /NE |
| BROMPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | MEPERIDINE HCL/PF |
| BROMPHENIRAMINE MALEATE/PHENYLEPHRINE | MEPERIDINE HCL/PROMETHAZINE HCL |
| BROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE | MORPHINE SULFATE IN O. 0. % CODILINA CILL ODIDE |
| BROMPHENIRAMINE/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE | MORPHINE SULFATE IN 0.9 % SODIUM CHLORIDE |
| BUTALBITAL/ACETAMINOPHEN/CAFFEINE/CODEINE PHOSPHATE | MORPHINE SULFATE UNOSOMAL/DE |
| CHLORCYCLIZINE HCL/CODEINE PHOSPHATE | MORPHINE SULFATE LIPOSOMAL/PF |
| TE DI CIDE VELLZINIE DEL ZUDENIVI EDDUDINE DEL JETA MANDENIE DUCCOUATE | |
| CHLORCYCLIZINE HCL/PHENYLEPHRINE HCL/CODEINE PHOSPHATE CHLORCYCLIZINE HCL/PSEUDOEPHEDRINE HCL/CODEINE | MORPHINE SULFATE/DEXTROSE 5 % IN WATER MORPHINE SULFATE/DEXTROSE 5% WATER/PF |

| To the second se | T |
|---|---|
| CHLORPHENIRAMINE MALEATE/CODEINE PHOSPHATE | MORPHINE SULFATE/NALTREXONE HCL |
| CHLORPHENIRAMINE MALEATE/CODEINE | MORPHINE SULFATE/PF |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE | OXYCODONE HCL |
| CHLORPHENIRAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE | OXYCODONE HCL/ACETAMINOPHEN |
| CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN | OXYCODONE/ASPIRIN |
| CODEINE PHOSPHATE/PYRILAMINE MALEATE | OXYMORPHONE HCL |
| CODEINE SULFATE | PHENYLEPHRINE HCL/CODEINE PHOSPHATE |
| CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE |
| CODEINE/CALCIUM IODIDE | PHENYLEPHRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| DEXBROMPHENIRAMINE MALEATE/PSEUDOEPHEDRINE | PHENYLEPHRINE |
| DEXCHLORPHENIRAMINE MALEATE/PHENYLEPHRINE | PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE |
| DIHYDROCODEINE BITARTRATE/ACETAMINOPHEN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE/CHLORPHENIRAMINE/POTASSIUM |
| DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE | PHENYLEPHRINE HCL/CODEINE/PYRILAMINE |
| DIHYDROCODEINE BITARTRATE/GUAIFENESIN | PHENYLEPHRINE HCL/DIHYDROCODEINE BITARTRATE |
| DIHYDROCODEINE/ASPIRIN/CAFFEINE | PHENYLEPHRINE HCL/DIHYDROCODEINE |
| DIPHENHYDRAMINE HCL/PHENYLEPHRINE HCL/CODEINE | PHENYLEPHRINE HCL/DIHYDROCODEINE |
| FENTANYL | PHENYLEPHRINE HCL/PPA |
| FENTANYL CITRATE | PHENYLEPHRINE TANNATE/HYDROCODONE |
| FENTANYL CITRATE IN 0.9 % SODIUM CHLORIDE/PF | PHENYLEPHRINE/HYDROCODONE |
| FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM | PHENYLEPHRINE/HYDROCODONE/BROMPHENIRAMINE TANNATES |
| FENTANYL CITRATE/DEXTROSE 5% WATER/PF | PHENYLEPHRINE/HYDROCODONE/DEXCHLORPHENIRAMINE |
| FENTANYL CITRATE/DROPERIDOL | PHENYLPROPANOLAMINE HCL/CODEINE/BROMPHENIRAMINE |
| FENTANYL CITRATE/PF | POTASSIUM GUAIACOLSULFONATE/PSEUDOEPHEDRINE |
| FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE 0.9%/PF | PROMETHAZINE HCL/CODEINE |
| GUAIFENESIN/CODEINE PHOSPHATE | PROMETHAZINE/PHENYLEPHRINE HCL/CODEINE |
| GUAIFENESIN/HYDROCODONE BITARTRATE | PROPOXYPHENE HCL |
| GUAIFENESIN/PHENYLEPHRINE HCL/HYDROCODONE | PROPOXYPHENE HCL/ACETAMINOPHEN |
| GUAIFENESIN/PHENYLPROPANOLAMINE HCL/CODEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| GUAIFENESIN/PHENYLPROPANOLAMINE | PROPOXYPHENE NAPSYLATE |
| GUAIFENESIN/PSEUDOEPHEDRINE HCL/DIHYDROCODEINE | PROPOXYPHENE NAPSYLATE/ACETAMINOPHEN |
| GUAIFENESIN/PSEUDOEPHEDRINE | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE |
| HYDROCODONE BITARTRATE | PSEUDOEPHEDRINE HCL/CODEINE |
| HYDROCODONE BITARTRATE/ACETAMINOPHEN | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/GUAIFENESIN |
| HYDROCODONE BITARTRATE/ACETAMINOPHEN/DIETARY | PSEUDOEPHEDRINE HCL/CODEINE PHOSPHATE/TRIPROLIDINE |
| HYDROCODONE BITARTRATE/ASPIRIN | PSEUDOEPHEDRINE HCL/CODEINE/CHLORPHENIRAMINE |
| HYDROCODONE BITARTRATE/CHLORPHENIRAMINE MALEATE | PSEUDOEPHEDRINE HCL/DIHYDROCODEINE |
| HYDROCODONE BITARTRATE/HOMATROPINE METHYLBROMIDE | PSEUDOEPHEDRINE HCL/HYDROCODONE BITARTRATE |
| HYDROCODONE TANNATE/CHLORPHENIRAMINE TANNATE | PSEUDOEPHEDRINE HCL/HYDROCODONE |
| HYDROCODONE/IBUPROFEN | PSEUDOEPHEDRINE TANNATE/HYDROCODONE TANNATE |
| HYDROMORPHONE HCL | PSEUDOEPHEDRINE/HYDROCODONE/BROMPHENIRAMINE |
| HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE | PSEUDOEPHEDRINE/HYDROCODONE/CHLORPHENIRAMINE |
| HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF | PYRILAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE PHOSPHATE |
| HYDROMORPHONE HCL IN DEXTROSE 5 % WATER/PF | PYRILAMINE MALEATE/PHENYLEPHRINE HCL/CODEINE PHOSPHATE PYRILAMINE MALEATE/PHENYLEPHRINE HCL/DIHYDROCODEINE BT |
| HYDROMORPHONE HCL/BUPIVACAINE HCL IN 0.9% SODIUM | PYRILAMINE MALEATE/PRENTLEPHRINE HCL/CODEINE PYRILAMINE MALEATE/PSEUDOEPHEDRINE HCL/CODEINE |
| HYDROMORPHONE HCL/PF | TRAMADOL HCL |
| IBUPROFEN/OXYCODONE HCL | TRAMADOL HCL/ACETAMINOPHEN |
| · | INAIVIADOL TICL/ACLIAIVIIIVOFTILIV |
| MEPERIDINE HCL | |

#### Glucocorticoids

| diacocorticolas | |
|---------------------------|----------------------|
| Ingredient code | |
| P5AR - prednisone | P5BC - dexamethasone |
| P5CB - triamcinolone | P5BB - betamethasone |
| P5AM - methylprednisolone | P5BL - budesonide |
| P5AB - hydrocortisone | P5AH - prednisolone |
| P5AA - cortisone | |

# Uric acid tests

| CPT |
|-------|
| 84550 |

**Atrial Fibrillation** 


| Coronary | <b>Artery</b> | Disease |
|----------|---------------|---------|


Heart Failure


| Dilation of Left Subdavian Artery with Four or More Intraluminal Devices, Open Approach— Dilation of Left Subdavian Artery, Bifurcation, Open Approach— Dilation of Left Subdavian Artery, Open Approach— Dilation of Left Subdavian Artery with Drug-eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Subdavian Artery with Two Drug-eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Subdavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Subdavian Artery with Two Intraluminal Device, Percutaneous Approach— Dilation of Left Subdavian Artery, With Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, With Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, With Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, With Tree Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subdavian Artery, Percutaneous Approach— Dilation of Left Subdavi |
|---|
| Dilation of Left Subclavian Artery, Bifurcation, Open Approach— Dilation of Left Subclavian Artery, Open Approach— Dilation of Left Subclavian Artery, Open Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach- Dilation of Left Subclavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach- Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of |
| 0374322 Dilation of Left Subclavian Artery, Open Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach—Intraluminal Device, Percutaneous Approach—Intraluminal Device, Percutaneous Approach—Intraluminal Device, Percutaneous Approach—Intraluminal Device, Percutaneous Approach—Intraluminal Devices, Percutaneous Endoscopic Approach—Intraluminal Devices, Percutaneous Endoscopic Approach—Intraluminal Devices, Percutaneous Endoscopic Approach—Intraluminal Devices, Percutaneous Endoscopic Approach—Intralu |
| Dilation of Left Subclavian Artery, Open Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percuta |
| Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Two Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left |
| Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery with Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subdavian Artery, Percutaneous Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Subdavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Dev |
| Intraluminal Device, Percutaneous Approach |
| Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery with Two Intraluminal Device, Percutaneous Approach Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach Dilation of Left Subclavian Artery, Percutaneous Approach Dilation of Left Subclavian Artery, Percutaneous Approach Dilation of Left Subclavian Artery, Percutaneous Approach Dilation of Left Subclavian Artery, Percutaneous Approach Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach |
| Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery with Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery with Two Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, Percutaneous Approach Dilation of Left Subdavian Artery, Percutaneous Approach- Dilation of Left Subdavian Artery, Percutaneous Approach- Dilation of Left Subdavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Approach |
| Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intral |
| Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subdavian Artery with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Subdavian Artery with Intraluminal Device, Percutaneous Approach- Dilation of Left Subdavian Artery with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Subdavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Subdavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Approach |
| Dilation of Left Subclavian Artery with Four or More Drugeluting Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting In |
| eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Intraluminal Devices, Percutaneous Approach |
| Dilation of Left Subclavian Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Intraluminal Device, Percutaneous Approach— |
| Dilation of Left Subclavian Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| 03743DZ Percutaneous Approach— Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Eluting Intraluminal Devices, Percutaneous End |
| Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or O3743G6 More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous |
| Intraluminal Devices, Percutaneous Approach— |
| Dilation of Left Subclavian Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approac |
| Dilation of Left Subclavian Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices Intraluminal Device |
| Dilation of Left Subclavian Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| O3743GZ Intraluminal Devices, Percutaneous Approach— Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— O3743Z6 Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery, Bifurcation, Percutaneous Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| O3743ZE Approach— Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery, Percutaneous Approach— Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Subclavian Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| O37444Z Approach Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Subclavian Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 037445Z Approach Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Subclavian Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| , |
| 037446Z Approach |
| Dilation of Left Subclavian Artery with Four or More Drug- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| Approach-eluting Intraluminal Devices, Percutaneous |
| 037447Z Endoscopic Approach |
| Dilation of Left Subclavian Artery, Bifurcation, with |
| 03744D6 Intraluminal Device, Percutaneous Endoscopic Approach— |
| Dilation of Left Subclavian Artery with Intraluminal Device, |
| 03744DZ Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery with Two Intraluminal 03744EZ Devices, Percutaneous Endoscopic Approach— Dilation of Left Subclavian Artery, Bifurcation, with Three 03744F6 Intraluminal Devices, Percutaneous Endoscopic Approach— |


| Dilation of Loft Internal Corptial Autory, Differentian with | T |
|---|---|
| •• | |
| , , | |
| , | |
| · | |
| , | |
| · | |
| 1 1 11 | |
| • | |
| • | |
| · | |
| i ii | |
| •• | |
| • | |
| Dilation of Left Internal Carotid Artery with Three | |
| Intraluminal Devices, Open Approach- | |
| Dilation of Left Internal Carotid Artery, Bifurcation, with | |
| Four or More Intraluminal Devices, Open Approach— | |
| Dilation of Left Internal Carotid Artery with Four or More | |
| Intraluminal Devices, Open Approach– | |
| Dilation of Left Internal Carotid Artery, Bifurcation, Open | |
| 2: | |
| i ii | |
| , , , | |
| · | |
| _ · | |
| Dilation of Right External Carotid Artery, Biflircation, with | |
| Dilation of Right External Carotid Artery, Bifurcation, with<br>Three Drug-eluting Intraluminal Devices, Open Approach- | |
| | Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery with Four or More Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, Open Approach— Dilation of Right External Carotid Artery, Bifurcation, with Drug-eluting Intraluminal Device, Open Approach— Dilation of Right External Carotid Artery with Drug-eluting Intraluminal Device, Open Approach Dilation of Right External Carotid Artery with Drug-eluting Intraluminal Device, Open Approach— Dilation of Right External Carotid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Open Approach— Dilation of Right External Carotid Artery with Two Drug-eluting Intraluminal Devices, Open Approach— Dilation of Right External Carotid Artery with Two Drug-eluting Intraluminal Devices, Open Approach—eluting Intraluminal Devices, Open Approach— |


| Insertion of Intraluminal Device into Left Internal Carotid | |
|---|---|
| 71 | |
| 71 | |
| S | |
| 1 11 | |
| 27 1 11 | |
| 1 11 | |
| · · · | |
| · | |
| • • | |
| · · I | |
| • • | |
| · · I | |
| · | |
| • • | |
| • • • • | |
| • • | |
| Percutaneous Approach- | |
| Insertion of Intraluminal Device into Left Temporal Artery, | |
| Percutaneous Endoscopic Approach- | |
| Insertion of Intraluminal Device into Right Thyroid Artery, | |
| Open Approach- | |
| Insertion of Intraluminal Device into Right Thyroid Artery, | |
| Percutaneous Approach- | |
| Insertion of Intraluminal Device into Right Thyroid Artery, | |
| Percutaneous Endoscopic Approach- | |
| Insertion of Intraluminal Device into Left Thyroid Artery, | |
| Open Approach- | |
| Insertion of Intraluminal Device into Left Thyroid Artery, | |
| | Insertion of Intraluminal Device into Left Temporal Artery, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Right Thyroid Artery, Open Approach— Insertion of Intraluminal Device into Right Thyroid Artery, Percutaneous Approach— Insertion of Intraluminal Device into Right Thyroid Artery, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Left Thyroid Artery, |


| Dilation of Right Renal Artery, Bifurcation, with Intraluminal | |
|---|---|
| Device, Percutaneous Endoscopic Approach | |
| i ii | |
| _ · | |
| , | |
| - ' | |
| · | |
| · · | |
| Endoscopic Approach- | |
| · | |
| · · | |
| , | |
| · | |
| 1 - 1 | |
| , | |
| Devices, Open Approach | |
| Dilation of Left Renal Artery, Bifurcation, with Three Drug- | |
| Intraluminal Devices, Open Approach | |
| Dilation of Left Renal Artery with Three Drug-eluting | |
| Intraluminal Devices, Open Approach-eluting Intraluminal | |
| Devices, Open Approach | |
| Dilation of Left Renal Artery, Bifurcation, with Four or More | |
| Drug-eluting Intraluminal Devices, Open Approach-eluting | |
| Intraluminal Devices, Open Approach | |
| Dilation of Left Renal Artery with Four or More Drug-eluting | |
| Intraluminal Devices, Open Approach-eluting Intraluminal | |
| Devices, Open Approach | |
| Dilation of Left Renal Artery, Bifurcation, with Intraluminal | |
| Device, Open Approach– | |
| Dilation of Left Renal Artery with Intraluminal Device, Open | |
| Approach- | |
| Dilation of Left Renal Artery, Bifurcation, with Two | |
| Intraluminal Devices, Open Approach- | |
| Dilation of Left Renal Artery with Two Intraluminal Devices, | |
| Open Approach | |
| Dilation of Left Renal Artery, Bifurcation, with Three | |
| Intraluminal Devices, Open Approach- | |
| Dilation of Left Renal Artery with Three Intraluminal | |
| Devices, Open Approach— | |
| Dilation of Left Renal Artery, Bifurcation, with Four or More | |
| Intraluminal Devices, Open Approach– | |
| Devices, Open Approach– | |
| | Dilation of Right Renal Artery, Percutaneous Endoscopic Approach— Dilation of Left Renal Artery, Bifurcation, with Drug-eluting Intraluminal Device, Open Approach-eluting Intraluminal Device, Open Approach—Dilation of Left Renal Artery with Drug-eluting Intraluminal Device, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery with Two Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery with Two Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery with Three Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Intraluminal Device, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Two Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Two Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Three Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Three Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Three Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Three Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach—Dilation of Left Renal Artery, Bifurcation, with Four |


| Dilation of Left Foot Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intralu |
|---|
| eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutane |
| D47W446 Approach Dilation of Left Foot Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Interlemental Device |
| Dilation of Left Foot Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approac |
| Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Turo Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Turo Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Itwo Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Itwo Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Itwo Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Device, Percutaneous Endoscopic Approach |
| Dilation of Left Foot Artery, Bifurcation, with Two Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, With Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Wifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Wifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Wifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal |
| Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Dilation of Left Foot Artery, Bifurcation, with Two Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, With Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery, Bifurcation, with Three Drug- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047W472 Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach-Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach-Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic A |
| Dilation of Left Foot Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two U47W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047W46Z Approach Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic 047W47Z Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal 047W4D6 Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic 047W47Z Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal 047W4D6 Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two O47W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047W476 Endoscopic Approach Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic 047W47Z Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- O47W4E6 Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— O47W4E6 |
| 047W47Z Approach Dilation of Left Foot Artery, Bifurcation, with Intraluminal 047W4D6 Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, 047W4DZ Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery, Bifurcation, with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two O47W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| 047W4DZ Percutaneous Endoscopic Approach— Dilation of Left Foot Artery, Bifurcation, with Two 047W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery, Bifurcation, with Two O47W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| 047W4E6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery with Two Intraluminal Devices, |
| 047W4EZ Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery, Bifurcation, with Three |
| 047W4F6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery with Three Intraluminal Devices, |
| 047W4FZ Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery, Bifurcation, with Four or More |
| 047W4G6 Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Foot Artery with Four or More Intraluminal |
| 047W4GZ Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Foot Artery, Bifurcation, Percutaneous |
| 7 11 |
| Dilation of Left Foot Artery, Percutaneous Endoscopic |
| 047W4ZZ Approach— |
| Dilation of Lower Artery, Bifurcation, with Drug-eluting |
| Intraluminal Device, Open Approach-eluting Intraluminal |
| 047Y046 Device, Open Approach |
| Dilation of Lower Artery with Drug-eluting Intraluminal |
| Device, Open Approach-eluting Intraluminal Device, Open |
| 047Y04Z Approach |


| Supplement Hemiazygos Vein with Autologous Tissue | |
|---|---|
| i ii | |
| 1 11 | |
| 1 '' | |
| 1 '' | |
| * * | |
| , | |
| • • | |
| 1 '' | |
| 1 '' | |
| , , , | |
| i ii | |
| 1 11 | |
| - | |
| 1 11 | |
| * * | |
| , , | |
| · | |
| • • • | |
| i ii | |
| 1 1 11 | |
| l | |
| 1 11 | |
| Supplement Left Innominate Vein with Synthetic Substitute, | |
| Percutaneous Approach | |
| Supplement Left Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Approach- | |
| Supplement Left Innominate Vein with Autologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach- | |
| Supplement Left Innominate Vein with Synthetic Substitute, | |
| Percutaneous Endoscopic Approach– | |
| Supplement Left Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Endoscopic Approach- | |
| Substitute, Open Approach- | |
| Substitute, Open Approach- | |
| Supplement Right Subclavian Vein with Synthetic | |
| | Percutaneous Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Innominate Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Innominate Vein with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Innominate Vein with Nonautologous |


| _ |
|---|


| | Revision of Extraluminal Device in Lower Vein, Percutaneous | |
|---|---|---|
| 06WY4CZ | Endoscopic Approach— | |
| | Revision of Intraluminal Device in Lower Vein, Percutaneous | |
| 06WY4DZ | Endoscopic Approach– | |
| HCPCS | | |
| 35256 | | |
| 35286 | | |
| 35351 | | |
| 35355 | | |
| 35361 | | |
| 35363 | | |
| 35371 | | |
| 35372 | | |
| 35381 | | |
| 35454 | | |
| 35456 | | |
| 35459 | | |
| 35470 | | |
| 35473 | | |
| 35474 | | |
| 35482 | | |
| 35483 | | |
| 35485 | | |
| 35492 | | |
| 35493 | | |
| 35495 | | |
| 35521 | | |
| 35533 | | |
| 35556 | | |
| 35558 | | |
| 35563 | | |
| 35565 | | |
| 35566 | | |
| 35571 | | |
| 35621 | | |
| 35623 | | |
| 35641 | | |
| 35646 | | |
| 35647 | | |
| 35650 | | |
| 35651 | | |
| 35654 | | |
| 35656 | | |
| 35661 | | |
| 35663 | | |
| 35666 | | |
| 35671 | I | |
| Hypertension | | |
| ICD10 Dx | ICD9 Dx LongDesICD10 | LongDesICD9 |

| 110 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
|---|---|---|---|
| 110 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| 110 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| 1160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| 1161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| 1169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| 1119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| l110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| 1119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| 1110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive chronic kidney disease, malignant, with chroni kidney disease stage I through stage IV, or unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic kidney disease or end stage renal disease | Hypertensive chronic kidney disease, malignant, with chroni kidney disease stage V or end stage renal disease |
| 1129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| 1123 | 40310 | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| 1120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| • | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| 1129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| 1123 | 40330 | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40201 | | |
| 1120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| 14040 | 40400 | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| 11310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| 11311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| 1132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end stage | with heart failure and with chronic kidney disease stage V o |
| | | renal disease | end stage renal disease |
| 11310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I through |
| | | or unspecified chronic kidney disease | stage IV, or unspecified |
| 11311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| .1011 | .0.112 | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| 1132 | 40413 | | heart failure and chronic kidney disease stage V or end stage |
| | | failure and with stage 5 chronic kidney disease, or end stage | , , , |
| 11210 | 40400 | renal disease | renal disease |
| 11310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| 11311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | i | stage renal disease | V or end stage renal disease |

| l132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
|---|---|---|---|
| | | failure and with stage 5 chronic kidney disease, or end stage | with heart failure and chronic kidney disease stage V or end |
| | | renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| I150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| l151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| I152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| I158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| I159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

Diabetes


Hyperlipidem ia

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| E780 | 2720 | Pure hypercholesterolemia | PURE HYPERCHOLESTEROLEMIA |
| E7800 | 2722 | | MIXED HYPERLIPIDEMIA |
| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| | | | _ |
|---|---|---|---|
| M10372 | 40410 | Gout due to renal impairment, left ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M10379 | 40411 | Gout due to renal impairment, unspecified ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M1038 | 40412 | Gout due to renal impairment, vertebrae | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | · · · | BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M1039 | 40413 | Gout due to renal impairment, multiple sites | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| 1011033 | 40413 | dout due to renar impairment, multiple sites | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | 1010 | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M3214 | 4049 | Glomerular disease in systemic lupus erythematosus | UNSPECIFIED HYPERTENSIVE HEART AND KIDNEY DISEASE |
| M3215 | 40490 | Tubulo-interstitial nephropathy in systemic lupus | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | erythematosus | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | | KIDNEY DISEASE STAGE I THROUGH STAGE IV OR |
| | | | UNSPECIFIED |
| M3504 | 40491 | Sicca syndrome with tubulo-interstitial nephropathy | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| N000 | 40492 | Acute nephritic syndrome with minor glomerular | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | .5.52 | abnormality | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | abilornanty | |
| NOOA | 40403 | A control of the control of the food and accounted | KIDNEY DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N001 | 40493 | Acute nephritic syndrome with focal and segmental | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | glomerular lesions | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N002 | 4533 | Acute nephritic syndrome with diffuse membranous | EMBOLISM AND THROMBOSIS OF RENAL VEIN |
| | | glomerulonephritis | |
| N003 | 5800 | Acute nephritic syndrome with diffuse mesangial | ACUTE GLOMERULONEPHRITIS WITH LESION OF |
| | | proliferative glomerulonephritis | PROLIFERATIVE GLOMERULONEPHRITIS |
| N004 | 5804 | Acute nephritic syndrome with diffuse endocapillary | ACUTE GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | proliferative glomerulonephritis | PROGRESSIVE GLOMERULONEPHRITIS |
| N005 | 5808 | Acute nephritic syndrome with diffuse mesangiocapillary | ACUTE GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| | | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N006 | 5809 | Acute nephritic syndrome with dense deposit disease | ACUTE GLOMERULONEPHRITIS WITH UNSPECIFIED |
| | 5005 | The state map in the symmetric with defined deposit disease | PATHOLOGICAL LESION IN KIDNEY |
| N007 | 581 | Acute nephritic syndrome with diffuse crescentic | NEPHROTIC SYNDROME |
| 14007 | 361 | glomerulonephritis | NEFTINOTIC STNDROWL |
| NOOO | 5040 | | NEDUDOTIC CVAID DOME MUTIL LECION OF PROLIFERATIVE |
| N008 | 5810 | Acute nephritic syndrome with other morphologic changes | NEPHROTIC SYNDROME WITH LESION OF PROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N009 | 5811 | Acute nephritic syndrome with unspecified morphologic | NEPHROTIC SYNDROME WITH LESION OF MEMBRANOUS |
| | | changes | GLOMERULONEPHRITIS |
| N010 | 5812 | Rapidly progressive nephritic syndrome with minor | NEPHROTIC SYNDROME WITH LESION OF |
| | | glomerular abnormality | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N011 | 5813 | Rapidly progressive nephritic syndrome with focal and | NEPHROTIC SYNDROME WITH LESION OF MINIMAL CHANG |
| | | segmental glomerular lesions | GLOMERULONEPHRITIS |
| N012 | 5818 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH OTHER SPECIFIED |
| · | | membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N013 | 58181 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME IN DISEASES CLASSIFIED |
| 14013 | 30101 | mesangial proliferative glomerulonephritis | |
| NO4.4 | 50400 | | ELSEWHERE |
| N014 | 58189 | Rapidly progressive nephritic syndrome with diffuse | OTHER NEPHROTIC SYNDROME WITH SPECIFIED |
| | | endocapillary proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED PATHOLOGICA |
| | | mesangiocapillary glomerulonephritis | LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense deposit | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | disease | PROLIFERATIVE GLOMERULONEPHRITIS |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | CHRONIC GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| 11010 | 3024 | morphologic changes | PROGRESSIVE GLOMERULONEPHRITIS |
| | | וווטו אווטוטבור נוומוובכים | I HOGHESSIVE GEOIVIERGEOIVEFIINITIS |

| N020 | 5828 | Recurrent and persistent hematuria with minor glomerular abnormality | CHRONIC GLOMERULONEPHRITIS WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
|---|---|---|---|
| N021 | 5829 | Recurrent and persistent hematuria with focal and segmental glomerular lesions | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| 11022 | 3030 | membranous glomerulonephritis | OR CHRONIC WITH LESION OF PROLIFERATIVE |
| | | membranous gromer aronephiners | GLOMERULONEPHRITIS |
| N023 | 5831 | Recurrent and persistent hematuria with diffuse mesangial | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| 11023 | 3031 | proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOUS |
| | | promerative gromerationeprints | GLOMERULONEPHRITIS |
| N024 | 5832 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | 3332 | endocapillary proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOPROLIFERATIVE |
| | | endocapinary promerative giorner dioneprintis | GLOMERULONEPHRITIS |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| 14025 | 3034 | mesangiocapillary glomerulonephritis | OR CHRONIC WITH LESION OF RAPIDLY PROGRESSIVE |
| | | mesangiocapinary giorner dioneprintis | GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| INUZU | 3630 | | |
| NO27 | F027 | disease | OR CHRONIC WITH LESION OF RENAL CORTICAL NECROSIS |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse crescentic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | glomerulonephritis | OR CHRONIC WITH LESION OF RENAL MEDULLARY NECROSIS |
| N028 | 5838 | Recurrent and persistent hematuria with other morphologic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | changes | OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESION |
| | | | IN KIDNEY |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | morphologic changes | OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN |
| | | mer priorogic ditainges | KIDNEY |
| N030 | 5846 | Chronic nephritic syndrome with minor glomerular | ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL |
| | 33.3 | abnormality | NECROSIS |
| N031 | 5847 | Chronic nephritic syndrome with focal and segmental | ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLAR |
| NOSI | 3047 | glomerular lesions | (PAPILLARY) NECROSIS |
| N032 | 5848 | Chronic nephritic syndrome with diffuse membranous | ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED |
| | | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N033 | 5849 | Chronic nephritic syndrome with diffuse mesangial | ACUTE KIDNEY FAILURE UNSPECIFIED |
| | | proliferative glomerulonephritis | |
| N034 | 5851 | Chronic nephritic syndrome with diffuse endocapillary | CHRONIC KIDNEY DISEASE STAGE I |
| | | proliferative glomerulonephritis | |
| N035 | 5852 | Chronic nephritic syndrome with diffuse mesangiocapillary | CHRONIC KIDNEY DISEASE STAGE II (MILD) |
| .1000 | 3332 | glomerulonephritis | |
| N036 | 5853 | Chronic nephritic syndrome with dense deposit disease | CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N037 | 5854 | Chronic nephritic syndrome with diffuse crescentic | CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| | | glomerulonephritis | , , |
| N038 | 5855 | Chronic nephritic syndrome with other morphologic changes | CHRONIC KIDNEY DISEASE STAGE V |
| N039 | 5856 | Chronic nephritic syndrome with unspecified morphologic | END STAGE RENAL DISEASE |
| | | changes | |
| N040 | 5859 | Nephrotic syndrome with minor glomerular abnormality | CHRONIC KIDNEY DISEASE UNSPECIFIED |
| N041 | 86600 | Nephrotic syndrome with focal and segmental glomerular | UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND |
| | | lesions | INTO CAVITY |
| N042 | 86601 | Nephrotic syndrome with diffuse membranous | HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE |
| | | glomerulonephritis | WITHOUT OPEN WOUND INTO CAVITY |
| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative | INJURY TO KIDNEY WITH OPEN WOUND INTO CAVITY |
| | | glomerulonephritis | |
| N044 | | Nephrotic syndrome with diffuse endocapillary proliferative | |
| | | glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic | |
| | I | glomerulonephritis | |
| | | giornei dionephiritis | |
| N048 | | Nephrotic syndrome with other morphologic changes | |

| | | Т |
|--------|---------------------------------------------------------------|---|
| N050 | Unspecified nephritic syndrome with minor glomerular | |
| | abnormality | _ |
| N051 | Unspecified nephritic syndrome with focal and segmental | |
| | glomerular lesions | |
| N052 | Unspecified nephritic syndrome with diffuse membranous | |
| | glomerulonephritis | |
| N053 | Unspecified nephritic syndrome with diffuse mesangial | |
| | proliferative glomerulonephritis | |
| N054 | Unspecified nephritic syndrome with diffuse endocapillary | |
| | proliferative glomerulonephritis | |
| N055 | Unspecified nephritic syndrome with diffuse | |
| | mesangiocapillary glomerulonephritis | |
| N056 | Unspecified nephritic syndrome with dense deposit disease | |
| N057 | Unspecified nephritic syndrome with diffuse crescentic | |
| | glomerulonephritis | |
| N058 | Unspecified nephritic syndrome with other morphologic | |
| | changes | |
| N059 | Unspecified nephritic syndrome with unspecified | |
| | morphologic changes | |
| N060 | Isolated proteinuria with minor glomerular abnormality | |
| N061 | Isolated proteinuria with focal and segmental glomerular | |
| .,,,,, | lesions | |
| N062 | Isolated proteinuria with diffuse membranous | 1 |
| 14002 | glomerulonephritis | |
| N063 | | |
| 11003 | Isolated proteinuria with diffuse mesangial proliferative | |
| NOCA | glomerulonephritis | - |
| N064 | Isolated proteinuria with diffuse endocapillary proliferative | |
| | glomerulonephritis | |
| N065 | Isolated proteinuria with diffuse mesangiocapillary | |
| | glomerulonephritis | |
| N066 | Isolated proteinuria with dense deposit disease | |
| N067 | Isolated proteinuria with diffuse crescentic | |
| | glomerulonephritis | |
| N068 | Isolated proteinuria with other morphologic lesion | |
| N069 | Isolated proteinuria with unspecified morphologic lesion | |
| N070 | Hereditary nephropathy, not elsewhere classified with | |
| | minor glomerular abnormality | |
| N071 | Hereditary nephropathy, not elsewhere classified with focal | |
| | and segmental glomerular lesions | |
| N072 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse membranous glomerulonephritis | |
| N073 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangial proliferative glomerulonephritis | |
| N074 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse endocapillary proliferative glomerulonephritis | |
| N075 | Hereditary nephropathy, not elsewhere classified with | 1 |
| - 1 | diffuse mesangiocapillary glomerulonephritis | |
| N076 | Hereditary nephropathy, not elsewhere classified with | |
| 1.07.5 | dense deposit disease | |
| N077 | Hereditary nephropathy, not elsewhere classified with | |
| 14077 | diffuse crescentic glomerulonephritis | |
| N078 | Hereditary nephropathy, not elsewhere classified with | 1 |
| NU/O | , , , , , | |
| NO70 | other morphologic lesions | + |
| N079 | Hereditary nephropathy, not elsewhere classified with | |
| NOO | unspecified morphologic lesions | |
| N08 | Glomerular disorders in diseases classified elsewhere | |
| N140 | Analgesic nephropathy | |
| N141 | Nephropathy induced by other drugs, medicaments and | |
| | biological substances | |
| N142 | Nephropathy induced by unspecified drug, medicament or | |
| | biological substance | |
| N143 | Nephropathy induced by heavy metals | |


## Appendix A Comorbid conditions

| 90964 |
|-------|
| 90965 |
| 90966 |
| 90967 |
| 90968 |
| 90969 |
| 90970 |
| 90989 |
| 90993 |
| 99512 |
| 99559 |


| K7581 | Nonalcoholic steatohepatitis (NASH) |
|-------|---------------------------------------------------|
| K7589 | Other specified inflammatory liver diseases |
| K759 | Inflammatory liver disease, unspecified |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K761 | Chronic passive congestion of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K765 | Hepatic veno-occlusive disease |
| K766 | Portal hypertension |
| K767 | Hepatorenal syndrome |
| K7681 | Hepatopulmonary syndrome |
| K7689 | Other specified diseases of liver |
| K769 | Liver disease, unspecified |
| K77 | Liver disorders in diseases classified elsewhere |

## **Asthma**


Ischemic heart disease


## Appendix A Comorbid conditions


COPD

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| J40 | 490 | Bronchitis, not specified as acute or chronic | BRONCHITIS NOT SPECIFIED AS ACUTE OR CHRONIC |
| J410 | 491 | Simple chronic bronchitis | CHRONIC BRONCHITIS |
| J411 | 4910 | Mucopurulent chronic bronchitis | SIMPLE CHRONIC BRONCHITIS |
| J418 | 4911 | Mixed simple and mucopurulent chronic bronchitis | MUCOPURULENT CHRONIC BRONCHITIS |
| J42 | 4912 | Unspecified chronic bronchitis | OBSTRUCTIVE CHRONIC BRONCHITIS |
| J430 | 49120 | Unilateral pulmonary emphysema [MacLeod's syndrome] | OBSTRUCTIVE CHRONIC BRONCHITIS WITHOUT |
| | | | EXACERBATION |
| J431 | 49121 | Panlobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH (ACUTE) |
| | | | EXACERBATION |
| J432 | 49122 | Centrilobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH ACUTE |
| | | | BRONCHITIS |
| J438 | 4918 | Other emphysema | OTHER CHRONIC BRONCHITIS |
| J439 | 4919 | Emphysema, unspecified | UNSPECIFIED CHRONIC BRONCHITIS |
| J440 | 492 | Chronic obstructive pulmonary disease with acute lower | EMPHYSEMA |
| | | respiratory infection | |
| J441 | 4920 | Chronic obstructive pulmonary disease with (acute) | EMPHYSEMATOUS BLEB |
| | | exacerbation | |
| J449 | 4928 | Chronic obstructive pulmonary disease, unspecified | OTHER EMPHYSEMA |
| J470 | 494 | Bronchiectasis with acute lower respiratory infection | BRONCHIECTASIS |
| J471 | 4940 | Bronchiectasis with (acute) exacerbation | BRONCHIECTASIS WITHOUT ACUTE EXACERBATION |
| J479 | 4941 | Bronchiectasis, uncomplicated | BRONCHIECTASIS WITH ACUTE EXACERBATION |
| | 496 | | CHRONIC AIRWAY OBSTRUCTION NOT ELSEWHERE |
| | | | CLASSIFIED |

Occurence of malignancy

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| C000 | 140 | Malignant neoplasm of external upper lip | MALIGNANT NEOPLASM OF LIP |
| C001 | 1400 | Malignant neoplasm of external lower lip | MALIGNANT NEOPLASM OF UPPER LIP VERMILION BORDER |
| C002 | 1401 | Malignant neoplasm of external lip, unspecified | MALIGNANT NEOPLASM OF LOWER LIP VERMILION BORDER |
| C003 | 1403 | Malignant neoplasm of upper lip, inner aspect | MALIGNANT NEOPLASM OF UPPER LIP INNER ASPECT |
| C004 | 1404 | Malignant neoplasm of lower lip, inner aspect | MALIGNANT NEOPLASM OF LOWER LIP INNER ASPECT |
| C005 | 1405 | Malignant neoplasm of lip, unspecified, inner aspect | MALIGNANT NEOPLASM OF LIP UNSPECIFIED INNER ASPECT |
| C006 | 1406 | Malignant neoplasm of commissure of lip, unspecified | MALIGNANT NEOPLASM OF COMMISSURE OF LIP |
| C008 | 1408 | Malignant neoplasm of overlapping sites of lip | MALIGNANT NEOPLASM OF OTHER SITES OF LIP |
| C009 | 1409 | Malignant neoplasm of lip, unspecified | MALIGNANT NEOPLASM OF LIP UNSPECIFIED VERMILION |
| | | | BORDER |
| C01 | 141 | Malignant neoplasm of base of tongue | MALIGNANT NEOPLASM OF TONGUE |
| C020 | 1410 | Malignant neoplasm of dorsal surface of tongue | MALIGNANT NEOPLASM OF BASE OF TONGUE |
| C021 | 1411 | Malignant neoplasm of border of tongue | MALIGNANT NEOPLASM OF DORSAL SURFACE OF TONGUE |
| C022 | 1412 | Malignant neoplasm of ventral surface of tongue | MALIGNANT NEOPLASM OF TIP AND LATERAL BORDER OF |
| | | | TONGUE |

| C023 | 1413 | Malignant neoplasm of anterior two-thirds of tongue, part unspecified | MALIGNANT NEOPLASM OF VENTRAL SURFACE OF TONGUE |
|---|---|---|---|
| C024 | 1414 | Malignant neoplasm of lingual tonsil | MALIGNANT NEOPLASM OF ANTERIOR TWO-THIRDS OF TONGUE PART UNSPECIFIED |
| C028 | 1415 | Malignant neoplasm of overlapping sites of tongue | MALIGNANT NEOPLASM OF JUNCTIONAL ZONE OF TONGUE |
| C029 | 1416 | Malignant neoplasm of tongue, unspecified | MALIGNANT NEOPLASM OF LINGUAL TONSIL |
| C030 | 1418 | Malignant neoplasm of upper gum | MALIGNANT NEOPLASM OF OTHER SITES OF TONGUE |
| C031 | 1419 | Malignant neoplasm of lower gum | MALIGNANT NEOPLASM OF TONGUE UNSPECIFIED |
| C039 | 142 | Malignant neoplasm of gum, unspecified | MALIGNANT NEOPLASM OF MAJOR SALIVARY GLANDS |
| C040 | 1420 | Malignant neoplasm of anterior floor of mouth | MALIGNANT NEOPLASM OF PAROTID GLAND |
| C041 | 1421 | Malignant neoplasm of lateral floor of mouth | MALIGNANT NEOPLASM OF SUBMANDIBULAR GLAND |
| C048 | 1422 | Malignant neoplasm of overlapping sites of floor of mouth | MALIGNANT NEOPLASM OF SUBLINGUAL GLAND |
| C049 | 1428 | Malignant neoplasm of floor of mouth, unspecified | MALIGNANT NEOPLASM OF OTHER MAJOR SALIVARY GLANDS |
| C050 | 1429 | Malignant neoplasm of hard palate | MALIGNANT NEOPLASM OF SALIVARY GLAND UNSPECIFIED |
| C051 | 143 | Malignant neoplasm of soft palate | MALIGNANT NEOPLASM OF GUM |
| C052 | 1430 | Malignant neoplasm of uvula | MALIGNANT NEOPLASM OF UPPER GUM |
| C058 | 1431 | Malignant neoplasm of overlapping sites of palate | MALIGNANT NEOPLASM OF LOWER GUM |
| C059 | 1438 | Malignant neoplasm of palate, unspecified | MALIGNANT NEOPLASM OF OTHER SITES OF GUM |
| C060 | 1439 | Malignant neoplasm of cheek mucosa | MALIGNANT NEOPLASM OF GUM UNSPECIFIED |
| C061 | 144 | Malignant neoplasm of vestibule of mouth | MALIGNANT NEOPLASM OF FLOOR OF MOUTH |
| C062 | 1440 | Malignant neoplasm of retromolar area | MALIGNANT NEOPLASM OF ANTERIOR PORTION OF FLOOR OF MOUTH |
| C0680 | 1441 | Malignant neoplasm of overlapping sites of unspecified parts of mouth | MALIGNANT NEOPLASM OF LATERAL PORTION OF FLOOR OF MOUTH |
| C0689 | 1448 | Malignant neoplasm of overlapping sites of other parts of mouth | MALIGNANT NEOPLASM OF OTHER SITES OF FLOOR OF MOUTH |
| C069 | 1449 | Malignant neoplasm of mouth, unspecified | MALIGNANT NEOPLASM OF FLOOR OF MOUTH PART UNSPECIFIED |
| C07 | 145 | Malignant neoplasm of parotid gland | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF MOUTH |
| C080 | 1450 | Malignant neoplasm of submandibular gland | MALIGNANT NEOPLASM OF CHEEK MUCOSA |
| C081 | 1451 | Malignant neoplasm of sublingual gland | MALIGNANT NEOPLASM OF VESTIBULE OF MOUTH |
| C089 | 1452 | Malignant neoplasm of major salivary gland, unspecified | MALIGNANT NEOPLASM OF HARD PALATE |
| C090 | 1453 | Malignant neoplasm of tonsillar fossa | MALIGNANT NEOPLASM OF SOFT PALATE |
| C091 | 1454 | Malignant neoplasm of tonsillar pillar (anterior) (posterior) | MALIGNANT NEOPLASM OF UVULA |
| C098 | 1455 | Malignant neoplasm of overlapping sites of tonsil | MALIGNANT NEOPLASM OF PALATE UNSPECIFIED |
| C099 | 1456 | Malignant neoplasm of tonsil, unspecified | MALIGNANT NEOPLASM OF RETROMOLAR AREA |
| C100 | 1458 | Malignant neoplasm of vallecula | MALIGNANT NEOPLASM OF OTHER SPECIFIED PARTS OF MOUTH |
| C101 | 1459 | Malignant neoplasm of anterior surface of epiglottis | MALIGNANT NEOPLASM OF MOUTH UNSPECIFIED |
| C102 | 146 | Malignant neoplasm of lateral wall of oropharynx | MALIGNANT NEOPLASM OF OROPHARYNX |
| C103 | 1460 | Malignant neoplasm of posterior wall of oropharynx | MALIGNANT NEOPLASM OF TONSIL |
| C104 | 1461 | Malignant neoplasm of branchial cleft | MALIGNANT NEOPLASM OF TONSILLAR FOSSA |
| C108 | 1462 | Malignant neoplasm of overlapping sites of oropharynx | MALIGNANT NEOPLASM OF TONSILLAR PILLARS (ANTERIOR) (POSTERIOR) |
| C109 | 1463 | Malignant neoplasm of oropharynx, unspecified | MALIGNANT NEOPLASM OF VALLECULA EPIGLOTTICA |
| C110 | 1464 | Malignant neoplasm of superior wall of nasopharynx | MALIGNANT NEOPLASM OF ANTERIOR ASPECT OF EPIGLOTTIS |
| C111 | 1465 | Malignant neoplasm of posterior wall of nasopharynx | MALIGNANT NEOPLASM OF JUNCTIONAL REGION OF OROPHARYNX |
| C112 | 1466 | Malignant neoplasm of lateral wall of nasopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF<br>OROPHARYNX |
| C113 | 1467 | Malignant neoplasm of anterior wall of nasopharynx | MALIGNANT NEOPLASM OF POSTERIOR WALL OF OROPHARYNX |
| C118 | 1468 | Malignant neoplasm of overlapping sites of nasopharynx | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF OROPHARYNX |
| C119 | 1469 | Malignant neoplasm of nasopharynx, unspecified | MALIGNANT NEOPLASM OF OROPHARYNX UNSPECIFIED SITE |
| C12 | 147 | Malignant neoplasm of pyriform sinus | MALIGNANT NEOPLASM OF NASOPHARYNX |

| C130 | 1470 | Malignant neoplasm of postcricoid region | MALIGNANT NEOPLASM OF SUPERIOR WALL OF |
|---|---|---|---|
| | | | NASOPHARYNX |
| C131 | 1471 | Malignant neoplasm of aryepiglottic fold, hypopharyngeal aspect | MALIGNANT NEOPLASM OF POSTERIOR WALL OF NASOPHARYNX |
| C132 | 1472 | Malignant neoplasm of posterior wall of hypopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF NASOPHARYNX |
| C138 | 1473 | Malignant neoplasm of overlapping sites of hypopharynx | MALIGNANT NEOPLASM OF ANTERIOR WALL OF |
| C130 | 1175 | Wanghane neoplasm of overlapping siees of mypopharym | NASOPHARYNX |
| C139 | 1478 | Malignant neoplasm of hypopharynx, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | , , , , , , | NASOPHARYNX |
| C140 | 1479 | Malignant neoplasm of pharynx, unspecified | MALIGNANT NEOPLASM OF NASOPHARYNX UNSPECIFIED SITE |
| C142 | 148 | Malignant neoplasm of Waldeyer's ring | MALIGNANT NEOPLASM OF HYPOPHARYNX |
| C148 | 1480 | Malignant neoplasm of overlapping sites of lip, oral cavity | MALIGNANT NEOPLASM OF POSTCRICOID REGION OF |
| | | and pharynx | HYPOPHARYNX |
| C153 | 1481 | Malignant neoplasm of upper third of esophagus | MALIGNANT NEOPLASM OF PYRIFORM SINUS |
| C154 | 1482 | Malignant neoplasm of middle third of esophagus | MALIGNANT NEOPLASM OF ARYEPIGLOTTIC FOLD |
| | | | HYPOPHARYNGEAL ASPECT |
| C155 | 1483 | Malignant neoplasm of lower third of esophagus | MALIGNANT NEOPLASM OF POSTERIOR HYPOPHARYNGEAL |
| | | | WALL |
| C158 | 1488 | Malignant neoplasm of overlapping sites of esophagus | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | HYPOPHARYNX |
| C159 | 1489 | Malignant neoplasm of esophagus, unspecified | MALIGNANT NEOPLASM OF HYPOPHARYNX UNSPECIFIED |
| | | | SITE |
| C160 | 149 | Malignant neoplasm of cardia | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES |
| | | | WITHIN THE LIP ORAL CAVITY AND PHARYNX |
| C161 | 1490 | Malignant neoplasm of fundus of stomach | MALIGNANT NEOPLASM OF PHARYNX UNSPECIFIED |
| C162 | 1491 | Malignant neoplasm of body of stomach | MALIGNANT NEOPLASM OF WALDEYER'S RING |
| C163 | 1498 | Malignant neoplasm of pyloric antrum | MALIGNANT NEOPLASM OF OTHER SITES WITHIN THE LIP |
| | | | AND ORAL CAVITY |
| C164 | 1499 | Malignant neoplasm of pylorus | MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE |
| | | | LIP AND ORAL CAVITY |
| C165 | 150 | Malignant neoplasm of lesser curvature of stomach, unspecified | MALIGNANT NEOPLASM OF ESOPHAGUS |
| C166 | 1500 | Malignant neoplasm of greater curvature of stomach, unspecified | MALIGNANT NEOPLASM OF CERVICAL ESOPHAGUS |
| C168 | 1501 | Malignant neoplasm of overlapping sites of stomach | MALIGNANT NEOPLASM OF THORACIC ESOPHAGUS |
| C169 | 1502 | Malignant neoplasm of stomach, unspecified | MALIGNANT NEOPLASM OF ABDOMINAL ESOPHAGUS |
| C170 | 1503 | Malignant neoplasm of duodenum | MALIGNANT NEOPLASM OF UPPER THIRD OF ESOPHAGUS |
| C171 | 1504 | Malignant neoplasm of jejunum | MALIGNANT NEOPLASM OF MIDDLE THIRD OF ESOPHAGUS |
| C172 | 1505 | Malignant neoplasm of ileum | MALIGNANT NEOPLASM OF LOWER THIRD OF ESOPHAGUS |
| C173 | 1508 | Meckel's diverticulum, malignant | MALIGNANT NEOPLASM OF OTHER SPECIFIED PART OF |
| | | The state of the s | ESOPHAGUS |
| C178 | 1509 | Malignant neoplasm of overlapping sites of small intestine | MALIGNANT NEOPLASM OF ESOPHAGUS UNSPECIFIED SITE |
| C179 | 151 | Malignant neoplasm of small intestine, unspecified | MALIGNANT NEOPLASM OF STOMACH |
| C180 | 1510 | Malignant neoplasm of cecum | MALIGNANT NEOPLASM OF CARDIA |
| C181 | 1511 | Malignant neoplasm of appendix | MALIGNANT NEOPLASM OF PYLORUS |
| C182 | 1512 | Malignant neoplasm of ascending colon | MALIGNANT NEOPLASM OF PYLORIC ANTRUM |
| C183 | 1513 | Malignant neoplasm of hepatic flexure | MALIGNANT NEOPLASM OF FUNDUS OF STOMACH |
| C184 | 1514 | Malignant neoplasm of transverse colon | MALIGNANT NEOPLASM OF BODY OF STOMACH |
| C185 | 1515 | Malignant neoplasm of splenic flexure | MALIGNANT NEOPLASM OF LESSER CURVATURE OF |
| | | | STOMACH UNSPECIFIED |
| C186 | 1516 | Malignant neoplasm of descending colon | MALIGNANT NEOPLASM OF GREATER CURVATURE OF |
| | | J | STOMACH UNSPECIFIED |
| C187 | 1518 | Malignant neoplasm of sigmoid colon | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| - | | | STOMACH |
| C188 | 1519 | Malignant neoplasm of overlapping sites of colon | MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED SITE |
| C189 | 152 | Malignant neoplasm of colon, unspecified | MALIGNANT NEOPLASM OF SMALL INTESTINE INCLUDING |
| | | | DUODENUM |
| C19 | 1520 | Malignant neoplasm of rectosigmoid junction | MALIGNANT NEOPLASM OF DUODENUM |

| C20 | 1521 | Malignant neoplasm of rectum | MALIGNANT NEOPLASM OF JEJUNUM |
|---|---|---|---|
| C210 | 1522 | Malignant neoplasm of anus, unspecified | MALIGNANT NEOPLASM OF ILEUM |
| C211 | 1523 | Malignant neoplasm of anal canal | MALIGNANT NEOPLASM OF MECKEL'S DIVERTICULUM |
| C212 | 1528 | Malignant neoplasm of cloacogenic zone | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| <del></del> | | | SMALL INTESTINE |
| C218 | 1529 | Malignant neoplasm of overlapping sites of rectum, anus | MALIGNANT NEOPLASM OF SMALL INTESTINE UNSPECIFIED |
| | | and anal canal | SITE |
| C220 | 153 | Liver cell carcinoma | MALIGNANT NEOPLASM OF COLON |
| C221 | 1530 | Intrahepatic bile duct carcinoma | MALIGNANT NEOPLASM OF HEPATIC FLEXURE |
| C222 | 1531 | Hepatoblastoma | MALIGNANT NEOPLASM OF TRANSVERSE COLON |
| C223 | 1532 | Angiosarcoma of liver | MALIGNANT NEOPLASM OF DESCENDING COLON |
| C224 | 1533 | Other sarcomas of liver | MALIGNANT NEOPLASM OF SIGMOID COLON |
| C227 | 1534 | Other specified carcinomas of liver | MALIGNANT NEOPLASM OF CECUM |
| C228 | 1535 | Malignant neoplasm of liver, primary, unspecified as to type | MALIGNANT NEOPLASM OF APPENDIX VERMIFORMIS |
| C229 | 1536 | Malignant neoplasm of liver, not specified as primary or secondary | MALIGNANT NEOPLASM OF ASCENDING COLON |
| C23 | 1537 | Malignant neoplasm of gallbladder | MALIGNANT NEOPLASM OF SPLENIC FLEXURE |
| C240 | 1538 | Malignant neoplasm of extrahepatic bile duct | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | LARGE INTESTINE |
| C241 | 1539 | Malignant neoplasm of ampulla of Vater | MALIGNANT NEOPLASM OF COLON UNSPECIFIED SITE |
| C248 | 154 | Malignant neoplasm of overlapping sites of biliary tract | MALIGNANT NEOPLASM OF RECTUM RECTOSIGMOID |
| | | , , , | JUNCTION AND ANUS |
| C249 | 1540 | Malignant neoplasm of biliary tract, unspecified | MALIGNANT NEOPLASM OF RECTOSIGMOID JUNCTION |
| C250 | 1541 | Malignant neoplasm of head of pancreas | MALIGNANT NEOPLASM OF RECTUM |
| C251 | 1542 | Malignant neoplasm of body of pancreas | MALIGNANT NEOPLASM OF ANAL CANAL |
| C252 | 1543 | Malignant neoplasm of tail of pancreas | MALIGNANT NEOPLASM OF ANUS UNSPECIFIED SITE |
| C253 | 1548 | Malignant neoplasm of pancreatic duct | MALIGNANT NEOPLASM OF OTHER SITES OF RECTUM |
| | | | RECTOSIGMOID JUNCTION AND ANUS |
| C254 | 155 | Malignant neoplasm of endocrine pancreas | MALIGNANT NEOPLASM OF LIVER AND INTRAHEPATIC BILE DUCTS |
| C257 | 1550 | Malignant neoplasm of other parts of pancreas | MALIGNANT NEOPLASM OF LIVER PRIMARY |
| C258 | 1551 | Malignant neoplasm of overlapping sites of pancreas | MALIGNANT NEOPLASM OF INTRAHEPATIC BILE DUCTS |
| C259 | 1552 | Malignant neoplasm of pancreas, unspecified | MALIGNANT NEOPLASM OF LIVER NOT SPECIFIED AS PRIMARY OR SECONDARY |
| C260 | 156 | Malignant neoplasm of intestinal tract, part unspecified | MALIGNANT NEOPLASM OF GALLBLADDER AND EXTRAHEPATIC BILE DUCTS |
| C261 | 1560 | Malignant neoplasm of spleen | MALIGNANT NEOPLASM OF GALLBLADDER |
| C269 | 1561 | Malignant neoplasm of ill-defined sites within the digestive | MALIGNANT NEOPLASM OF EXTRAHEPATIC BILE DUCTS |
| | | system | |
| C300 | 1562 | Malignant neoplasm of nasal cavity | MALIGNANT NEOPLASM OF AMPULLA OF VATER |
| C301 | 1568 | Malignant neoplasm of middle ear | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | GALLBLADDER AND EXTRAHEPATIC BILE DUCTS |
| C310 | 1569 | Malignant neoplasm of maxillary sinus | MALIGNANT NEOPLASM OF BILIARY TRACT PART |
| | | | UNSPECIFIED SITE |
| C311 | 157 | Malignant neoplasm of ethmoidal sinus | MALIGNANT NEOPLASM OF PANCREAS |
| C312 | 1570 | Malignant neoplasm of frontal sinus | MALIGNANT NEOPLASM OF HEAD OF PANCREAS |
| C313 | 1571 | Malignant neoplasm of sphenoid sinus | MALIGNANT NEOPLASM OF BODY OF PANCREAS |
| C318 | 1572 | Malignant neoplasm of overlapping sites of accessory | MALIGNANT NEOPLASM OF TAIL OF PANCREAS |
| C319 | 1573 | Sinuses Malignant neoplasm of accessory sinus, unspecified | MALIGNANT NEOPLASM OF PANCREATIC DUCT |
| C319 | 1573 | Malignant neoplasm of accessory sinus, unspectified Malignant neoplasm of glottis | MALIGNANT NEOPLASM OF PANCREATIC DUCT MALIGNANT NEOPLASM OF ISLETS OF LANGERHANS |
| C320 | 1574 | Malignant neoplasm of glottis Malignant neoplasm of supraglottis | MALIGNANT NEOPLASM OF ISLETS OF LANGERHANS MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C321 | 13/8 | Manghant heopiasin of supragiotits | PANCREAS |
| C322 | 1579 | Malignant neoplasm of subglottis | MALIGNANT NEOPLASM OF PANCREAS PART UNSPECIFIED |
| C323 | 158 | Malignant neoplasm of laryngeal cartilage | MALIGNANT NEOPLASM OF RETROPERITONEUM AND |
| 0020 | | | PERITONEUM |
| C328 | 1580 | Malignant neoplasm of overlapping sites of larynx | MALIGNANT NEOPLASM OF RETROPERITONEUM |
| C329 | 1588 | Malignant neoplasm of larynx, unspecified | MALIGNANT NEOPLASM OF SPECIFIED PARTS OF |
| | | · | PERITONEUM |


| C438 | 1722 | Malignant melanoma of overlapping sites of skin | MALIGNANT MELANOMA OF SKIN OF EAR AND EXTERNAL |
|---|---|---|---|
| | | | AUDITORY CANAL |
| C439 | 1723 | Malignant melanoma of skin, unspecified | MALIGNANT MELANOMA OF SKIN OF OTHER AND UNSPECIFIED PARTS OF FACE |
| C450 | 1724 | Mesothelioma of pleura | MALIGNANT MELANOMA OF SKIN OF SCALP AND NECK |
| C451 | 1725 | Mesothelioma of peritoneum | MALIGNANT MELANOMA OF SKIN OF TRUNK EXCEPT SCROTUM |
| C452 | 1726 | Mesothelioma of pericardium | MALIGNANT MELANOMA OF SKIN OF UPPER LIMB INCLUDING SHOULDER |
| C457 | 1727 | Mesothelioma of other sites | MALIGNANT MELANOMA OF SKIN OF LOWER LIMB |
| C459 | 1728 | Mesothelioma, unspecified | MALIGNANT MELANOMA OF OTHER SPECIFIED SITES OF |
| C460 | 1729 | Kaposi's sarcoma of skin | SKIN |
| C460<br>C461 | 1729 | Kaposi's sarcoma of soft tissue | MELANOMA OF SKIN SITE UNSPECIFIED MALIGNANT NEOPLASM OF FEMALE BREAST |
| C461 | 1740 | | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF |
| | | Kaposi's sarcoma of palate | FEMALE BREAST |
| C463 | 1741 | Kaposi's sarcoma of lymph nodes | MALIGNANT NEOPLASM OF CENTRAL PORTION OF FEMALE BREAST |
| C464 | 1742 | Kaposi's sarcoma of gastrointestinal sites | MALIGNANT NEOPLASM OF UPPER-INNER QUADRANT OF FEMALE BREAST |
| C4650 | 1743 | Kaposi's sarcoma of unspecified lung | MALIGNANT NEOPLASM OF LOWER-INNER QUADRANT OF |
| | | | FEMALE BREAST |
| C4651 | 1744 | Kaposi's sarcoma of right lung | MALIGNANT NEOPLASM OF UPPER-OUTER QUADRANT OF |
| | | | FEMALE BREAST |
| C4652 | 1745 | Kaposi's sarcoma of left lung | MALIGNANT NEOPLASM OF LOWER-OUTER QUADRANT OF |
| | | | FEMALE BREAST |
| C467 | 1746 | Kaposi's sarcoma of other sites | MALIGNANT NEOPLASM OF AXILLARY TAIL OF FEMALE |
| C-107 | 1740 | Raposi s surcoma of other sites | BREAST |
| C469 | 1748 | Kaposi's sarcoma, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C 103 | 17 10 | haposi s surcoma, unspecimea | FEMALE BREAST |
| C470 | 1749 | Malignant neoplasm of peripheral nerves of head, face and | MALIGNANT NEOPLASM OF BREAST (FEMALE) UNSPECIFIED |
| C+70 | 1743 | neck | SITE |
| C4710 | 175 | Malignant neoplasm of peripheral nerves of unspecified | MALIGNANT NEOPLASM OF MALE BREAST |
| C4711 | 1750 | upper limb, including shoulder Malignant neoplasm of peripheral nerves of right upper | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF MALE |
| C4/11 | 1/50 | | BREAST |
| C4712 | 1750 | limb, including shoulder Malignant neoplasm of peripheral nerves of left upper limb, | |
| C4712 | 1759 | | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED SITE: |
| 04700 | 476 | including shoulder | OF MALE BREAST |
| C4720 | 176 | Malignant neoplasm of peripheral nerves of unspecified lower limb, including hip | KAPOSI'S SARCOMA |
| C4721 | 1760 | Malignant neoplasm of peripheral nerves of right lower limb, including hip | KAPOSI'S SARCOMA SKIN |
| C4722 | 1761 | Malignant neoplasm of peripheral nerves of left lower limb, including hip | KAPOSI'S SARCOMA SOFT TISSUE |
| | 1762 | | |
| C473 | 1/02 | Malignant neoplasm of peripheral nerves of thorax | KAPOSI'S SARCOMA PALATE |
| C474 | 1763 | Malignant neoplasm of peripheral nerves of abdomen | KAPOSI'S SARCOMA GASTROINTESTINAL SITES |
| | | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, | |
| C474<br>C475 | 1763<br>1764 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG |
| C474<br>C475<br>C476 | 1763<br>1764<br>1765 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768<br>1769 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE |
| C474<br>C475<br>C476<br>C478<br>C479 | 1763<br>1764<br>1765<br>1768<br>1769 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS |
| C474<br>C475<br>C476<br>C478<br>C479<br>C480<br>C481 | 1763<br>1764<br>1765<br>1768<br>1769<br>179<br>180 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum Malignant neoplasm of specified parts of peritoneum Malignant neoplasm of peritoneum, unspecified Malignant neoplasm of overlapping sites of retroperitoneum | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS MALIGNANT NEOPLASM OF CERVIX UTERI MALIGNANT NEOPLASM OF ENDOCERVIX |
| C474<br>C475<br>C476<br>C478<br>C479<br>C480<br>C481<br>C482 | 1763<br>1764<br>1765<br>1768<br>1769<br>179<br>180<br>1800 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum Malignant neoplasm of specified parts of peritoneum Malignant neoplasm of peritoneum, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS MALIGNANT NEOPLASM OF CERVIX UTERI MALIGNANT NEOPLASM OF ENDOCERVIX |


| C50929 | 1909 | Malignant neoplasm of unspecified site of unspecified male breast | MALIGNANT NEOPLASM OF EYE PART UNSPECIFIED |
|---|---|---|---|
| C510 | 191 | Malignant neoplasm of labium majus | MALIGNANT NEOPLASM OF BRAIN |
| C511 | 1910 | Malignant neoplasm of labium minus | MALIGNANT NEOPLASM OF CEREBRUM EXCEPT LOBES AN VENTRICLES |
| C512 | 1911 | Malignant neoplasm of clitoris | MALIGNANT NEOPLASM OF FRONTAL LOBE |
| C518 | 1912 | Malignant neoplasm of overlapping sites of vulva | MALIGNANT NEOPLASM OF TEMPORAL LOBE |
| C519 | 1913 | Malignant neoplasm of vulva, unspecified | MALIGNANT NEOPLASM OF PARIETAL LOBE |
| C52 | 1914 | Malignant neoplasm of vagina | MALIGNANT NEOPLASM OF OCCIPITAL LOBE |
| C530 | 1915 | Malignant neoplasm of endocervix | MALIGNANT NEOPLASM OF VENTRICLES |
| C531 | 1916 | Malignant neoplasm of exocervix | MALIGNANT NEOPLASM OF CEREBELLUM NOT OTHERWIS |
| 0001 | 1510 | mang. and neephasm of electricity | SPECIFIED |
| C538 | 1917 | Malignant neoplasm of overlapping sites of cervix uteri | MALIGNANT NEOPLASM OF BRAIN STEM |
| C539 | 1918 | Malignant neoplasm of cervix uteri, unspecified | MALIGNANT NEOPLASM OF OTHER PARTS OF BRAIN |
| C540 | 1919 | Malignant neoplasm of isthmus uteri | MALIGNANT NEOPLASM OF BRAIN UNSPECIFIED SITE |
| C541 | 192 | Malignant neoplasm of endometrium | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF NERVOUS SYSTEM |
| C542 | 1920 | Malignant neoplasm of myometrium | MALIGNANT NEOPLASM OF CRANIAL NERVES |
| | | Malignant neoplasm of fundus uteri | MALIGNANT NEOPLASM OF CRANIAL NERVES MALIGNANT NEOPLASM OF CEREBRAL MENINGES |
| C543 | 1921 | · | |
| C548 | 1922 | Malignant neoplasm of overlapping sites of corpus uteri | MALIGNANT NEOPLASM OF SPINAL CORD |
| C549 | 1923 | Malignant neoplasm of corpus uteri, unspecified | MALIGNANT NEOPLASM OF SPINAL MENINGES |
| C55 | 1928 | Malignant neoplasm of uterus, part unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF NERVOUS SYSTEM |
| CEC1 | 1020 | Malignant needlasm of right overv | MALIGNANT NEOPLASM OF NERVOUS SYSTEM PART |
| C561 | 1929 | Malignant neoplasm of right ovary | UNSPECIFIED |
| CEGO | 102 | Malignant needless of left every | |
| C562 | 193 | Malignant neoplasm of left ovary | MALIGNANT NEOPLASM OF THYROID GLAND |
| C569 | 194 | Malignant neoplasm of unspecified ovary | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 05700 | 1010 | | AND RELATED STRUCTURES |
| C5700 | 1940 | Malignant neoplasm of unspecified fallopian tube | MALIGNANT NEOPLASM OF ADRENAL GLAND |
| C5701 | 1941 | Malignant neoplasm of right fallopian tube | MALIGNANT NEOPLASM OF PARATHYROID GLAND |
| C5702 | 1943 | Malignant neoplasm of left fallopian tube | MALIGNANT NEOPLASM OF PITUITARY GLAND AND |
| | | | CRANIOPHARYNGEAL DUCT |
| C5710 | 1944 | Malignant neoplasm of unspecified broad ligament | MALIGNANT NEOPLASM OF PINEAL GLAND |
| C5711 | 1945 | Malignant neoplasm of right broad ligament | MALIGNANT NEOPLASM OF CAROTID BODY |
| C5712 | 1946 | Malignant neoplasm of left broad ligament | MALIGNANT NEOPLASM OF AORTIC BODY AND OTHER PARAGANGLIA |
| C5720 | 1948 | Malignant neoplasm of unspecified round ligament | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 03720 | 25 .0 | manghant heopiasin of anopeanies rouns ngament | AND RELATED STRUCTURES |
| C5721 | 1949 | Malignant neoplasm of right round ligament | MALIGNANT NEOPLASM OF ENDOCRINE GLAND SITE |
| C3721 | 1343 | Wanghane neoplasm of right round ngament | UNSPECIFIED |
| C5722 | 195 | Malignant neoplasm of left round ligament | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITE |
| C573 | 1950 | Malignant neoplasm of parametrium | MALIGNANT NEOPLASM OF HEAD FACE AND NECK |
| C574 | 1951 | Malignant neoplasm of uterine adnexa, unspecified | MALIGNANT NEOPLASM OF THORAX |
| C577 | 1952 | Malignant neoplasm of other specified female genital organs | s MALIGNANT NEOPLASM OF ABDOMEN |
| C578 | 1953 | Malignant neoplasm of overlapping sites of female genital | MALIGNANT NEOPLASM OF PELVIS |
| C579 | 1954 | organs Malignant neoplasm of female genital organ, unspecified | MALIGNANT NEOPLASM OF UPPER LIMB |
| C579 | 1954 | Malignant neoplasm of lemale genital organ, unspecified Malignant neoplasm of placenta | MALIGNANT NEOPLASM OF LOWER LIMB |
| C600 | | Malignant neoplasm of prepuce | |
| | 1958 | Malignant neoplasm of prepuce Malignant neoplasm of glans penis | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| C601 | 196 | Mangnant neoplasm of glans penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM LYMPH NODES |
| C602 | 1960 | Malignant neoplasm of body of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 0000 | | | LYMPH NODES OF HEAD FACE AND NECK |
| C608 | 1961 | Malignant neoplasm of overlapping sites of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM INTRATHORACIC LYMPH NODES |
| C609 | 1962 | Malignant neoplasm of penis, unspecified | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 2233 | 1332 | | INTRA-ABDOMINAL LYMPH NODES |
| C61 | 1963 | Malignant neoplasm of prostate | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| COI | 1,000 | manghant neoplasm of prostate | SESSIONIL AND ONSI EGI IED MALIGINAMI MEOFEASIM |


| C7491 | 20071 | Malignant neoplasm of unspecified part of right adrenal | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF |
|---|---|---|---|
| | | gland | HEAD FACE AND NECK |
| C7492 | 20072 | Malignant neoplasm of unspecified part of left adrenal gland | LARGE CELL LYMPHOMA INVOLVING INTRATHORACIC LYMPH<br>NODES |
| C750 | 20073 | Malignant neoplasm of parathyroid gland | LARGE CELL LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| C751 | 20074 | Malignant neoplasm of pituitary gland | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF |
| 6750 | 20075 | | AXILLA AND UPPER LIMB |
| C752 | 20075 | Malignant neoplasm of craniopharyngeal duct | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| C753 | 20076 | Malignant neoplasm of pineal gland | LARGE CELL LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| C754 | 20077 | Malignant neoplasm of carotid body | LARGE CELL LYMPHOMA INVOLVING SPLEEN |
| C755 | 20078 | Malignant neoplasm of aortic body and other paraganglia | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| C758 | 2008 | Malignant neoplasm with pluriglandular involvement, unspecified | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA |
| C759 | 20080 | Malignant neoplasm of endocrine gland, unspecified | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND |
| | | | RETICULOSARCOMA UNSPECIFIED SITE |
| C760 | 20081 | Malignant neoplasm of head, face and neck | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| C761 | 20082 | Malignant neoplasm of thorax | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRATHORACIC LYMPH NODES |
| C762 | 20083 | Malignant neoplasm of abdomen | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| C763 | 20084 | Malignant neoplasm of pelvis | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| C7640 | 20085 | Malignant neoplasm of unspecified upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF INGUINA REGION AND LOWER LIMB |
| C7641 | 20086 | Malignant neoplasm of right upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRAPELVIC LYMPH NODES |
| C7642 | 20087 | Malignant neoplasm of left upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING SPLEEN |
| C7650 | 20088 | Malignant neoplasm of unspecified lower limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| C7651 | 201 | Malignant neoplasm of right lower limb | HODGKIN'S DISEASE |
| | 2010 | 0 1 0 | |
| C7652 | 1 | Malignant neoplasm of left lower limb | HODGKIN'S PARAGRANULOMA |
| C768<br>C770 | 20100<br>20101 | Malignant neoplasm of other specified ill-defined sites Secondary and unspecified malignant neoplasm of lymph | HODGKIN'S PARAGRANULOMA UNSPECIFIED SITE HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES |
| C771 | 20102 | nodes of head, face and neck Secondary and unspecified malignant neoplasm of | OF HEAD FACE AND NECK HODGKIN'S PARAGRANULOMA INVOLVING INTRATHORACIC |
| | | intrathoracic lymph nodes | LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING INTRA- |
| C772 | 20103 | Secondary and unspecified malignant neoplasm of intra- | HODOKIN STANAGIANOLOMA INVOLVING INTIA- |
| | | abdominal lymph nodes | ABDOMINAL LYMPH NODES |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes Secondary and unspecified malignant neoplasm of | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB HODGKIN'S PARAGRANULOMA INVOLVING INTRAPELVIC |
| C773 C774 C775 | 20104<br>20105<br>20106 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes Secondary and unspecified malignant neoplasm of intrapelvic lymph nodes Secondary and unspecified malignant neoplasm of lymph | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB HODGKIN'S PARAGRANULOMA INVOLVING INTRAPELVIC LYMPH NODES |


| D 100 | I November of the state of the land of the land | |
|---|---|---|
| D409 | Neoplasm of uncertain behavior of male genital organ, | |
| D 44.00 | unspecified | |
| D4100 | Neoplasm of uncertain behavior of unspecified kidney | |
| D4101 | Neoplasm of uncertain behavior of right kidney | |
| D4102 | Neoplasm of uncertain behavior of left kidney | |
| D4110 | Neoplasm of uncertain behavior of unspecified renal pelvis | |
| D4111 | Neoplasm of uncertain behavior of right renal pelvis | |
| D4112 | Neoplasm of uncertain behavior of left renal pelvis | |
| D4120 | Neoplasm of uncertain behavior of unspecified ureter | |
| D4121 | Neoplasm of uncertain behavior of right ureter | |
| D4122 | Neoplasm of uncertain behavior of left ureter | |
| D413 | Neoplasm of uncertain behavior of urethra | |
| D414 | Neoplasm of uncertain behavior of bladder | |
| D418 | Neoplasm of uncertain behavior of other specified urinary | |
| | organs | |
| D419 | Neoplasm of uncertain behavior of unspecified urinary organ | |
| D420 | Neoplasm of uncertain behavior of cerebral meninges | |
| D421 | Neoplasm of uncertain behavior of spinal meninges | |
| D429 | Neoplasm of uncertain behavior of meninges, unspecified | |
| D430 | Neoplasm of uncertain behavior of brain, supratentorial | |
| D431 | Neoplasm of uncertain behavior of brain, infratentorial | |
| D432 | Neoplasm of uncertain behavior of brain, unspecified | |
| D433 | Neoplasm of uncertain behavior of cranial nerves | |
| D434 | Neoplasm of uncertain behavior of spinal cord | |
| D438 | Neoplasm of uncertain behavior of other specified parts of | |
| | central nervous system | |
| D439 | Neoplasm of uncertain behavior of central nervous system, | |
| | unspecified | |
| D440 | Neoplasm of uncertain behavior of thyroid gland | |
| D4410 | Neoplasm of uncertain behavior of unspecified adrenal gland | |
| , | | |
| D4411 | Neoplasm of uncertain behavior of right adrenal gland | |
| D4412 | Neoplasm of uncertain behavior of left adrenal gland | |
| D442 | Neoplasm of uncertain behavior of parathyroid gland | |
| D443 | Neoplasm of uncertain behavior of pituitary gland | |
| D444 | Neoplasm of uncertain behavior of greatery grand Neoplasm of uncertain behavior of craniopharyngeal duct | |
| D445 | Neoplasm of uncertain behavior of pineal gland | |
| D446 | Neoplasm of uncertain behavior of carotid body | |
| D447 | Neoplasm of uncertain behavior of aortic body Neoplasm of uncertain behavior of aortic body and other | |
| D447 | paraganglia | |
| D449 | Neoplasm of uncertain behavior of unspecified endocrine | |
| D443 | gland | |
| D45 | Polycythemia vera | |
| D460 | Refractory anemia without ring sideroblasts, so stated | |
| D460<br>D461 | Refractory anemia without ring sideroblasts, so stated | |
| D461<br>D4620 | Refractory anemia with ring sideroblasts Refractory anemia with excess of blasts, unspecified | |
| D4620<br>D4621 | · | |
| | Refractory anemia with excess of blasts 1 | |
| D4622 | Refractory anemia with excess of blasts 2 | |
| D464 | Refractory anemia, unspecified | |
| D469 | Myelodysplastic syndrome, unspecified | |
| D46A | Refractory cytopenia with multilineage dysplasia | |
| D46B | Refractory cytopenia with multilineage dysplasia and ring | |
| D.163 | sideroblasts | |
| D46C | Myelodysplastic syndrome with isolated del(5q) | |
| | chromosomal abnormality | |
| D46Z | Other myelodysplastic syndromes | |
| D470 | Histiocytic and mast cell tumors of uncertain behavior | |
| | | 1 |
| D471 | Chronic myeloproliferative disease | |
| D473 | Essential (hemorrhagic) thrombocythemia | |


Drug abuse or dependence (includes alcohol)


| PRESSANT TYPE ABUSE EPISODIC PRESSANT TYPE ABUSE IN MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
|---|
| PRESSANT TYPE ABUSE IN MIXED OR UNSPECIFIED DRUG CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| PRESSANT TYPE ABUSE IN MIXED OR UNSPECIFIED DRUG CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| CIFIED DRUG ABUSE UNSPECIFIED MIXED OR UNSPECIFIED DRUG MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |
| MIXED OR UNSPECIFIED DRUG |


Venous throm boem bolism


## Appendix A Comorbid conditions
